Data Analysis for Drug Repurposing for Effective Alzheimer's Medicines – PDE5 inhibitors vs endothelin receptor antagonists

NCT05039086

October 27, 2021

### 1. Comparison Details

### a. Intended aim(s)

To evaluate the comparative risk of dementia onset between patients treated with <u>PDE5 inhibitors (sildenafil, tadalafil)</u> versus endothelin receptor antagonists (bosentan, ambrisentan, macitentan) for pulmonary arterial hypertension.

### b. Primary endpoint

Incident dementia (i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere).

### 2. Person responsible for implementation of replication in Aetion

Mufaddal Mahesri

## 3. Data Source(s)

Medicare, 2008-2018

### 4. Study Design Diagrams





#### 5. Cohort Identification

#### a. Cohort Summary

This study will employ a new user, active comparator, observational cohort study design comparing <u>PDE5 inhibitors</u> (sildenafil, tadalafil) versus endothelin receptor antagonists (bosentan, ambrisentan, macitentan). The patients will be required to have continuous enrollment during the baseline period of 365 days before initiation of study drugs (cohort entry/index date). Follow-up for the outcome (dementia) differs between analyses. Follow-up begins the day after drug initiation (analysis 1, 3, 4); 180 days after drug initiation (analysis 2).

#### b. Key details regarding cohort creation

#### Index date:

• Day of initiation of new <u>PDE5 inhibitors (sildenafil, tadalafil) versus endothelin receptor antagonists (bosentan, ambrisentan, macitentan)</u> use

Inclusion criteria for analyses 1, 3, 4:

- Aged > 65 years on the index date
- 365 days enrollment in Medicare Parts A, B, and D with no HMO coverage
- No use of <u>PDE5 inhibitors (sildenafil, tadalafil) versus endothelin receptor antagonists (bosentan, ambrisentan, macitentan)</u>, any time prior to index date (all available lookback approach with a minimum of 365 days)
- No diagnosis of dementia any time prior to and including index date
- No history of nursing home admission recorded in any time prior to and including index date
- At least two claims with pulmonary arterial hypertension diagnosis recorded in 365 days prior to index date (ICD-9 416.0, 416.8, 416.9 or ICD-10 I27.0, I27.2, I27.8, I27.9)<sup>1</sup>

### Inclusion criteria for analysis 2:

- Aged ≥ 65 years on the index date
- 365 days enrollment in Medicare Parts A, B, and D with no HMO coverage or 365 days registration with a practice contributing data to CPRD prior to index date
- No use of <u>PDE5 inhibitors (sildenafil, tadalafil) versus endothelin receptor antagonists (bosentan, ambrisentan, macitentan)</u>, any time prior to index date (all available lookback approach with a minimum of 365 days)
- No diagnosis of dementia any time prior to and including index date

- No history of nursing home admission recorded in any time prior to and including index date
- At least two claims with pulmonary arterial hypertension diagnosis recorded in 365 days prior to index date (ICD-9 416.0, 416.8, 416.9 or ICD-10 I27.0, I27.2, I27.8, I27.9)<sup>1</sup>
- 180-day continuous use of <u>PDE5 inhibitors (sildenafil, tadalafil) versus endothelin receptor antagonists (bosentan, ambrisentan, macitentan)</u> starting on the index date

# c. Flowchart of the study cohort assembly

| | Less Excluded Patients | Remaining Patients |
|---|---|---|
| All patients | | 25,300,359 |
| Did not meet cohort entry criteria | -25,152,975 | 147,384 |
| Excluded due to insufficient enrollment | -75,128 | 72,256 |
| Excluded due to prior use of referent | -5,776 | 66,480 |
| Excluded due to prior use of exposure | -42,086 | 24,394 |
| Excluded because patient qualified in >1 exposure category | -24 | 24,370 |
| Excluded based on Dementia Exclusion | -1,187 | 23,183 |
| Excluded based on PAH Diagnosis | -9,086 | 14,097 |
| Excluded based on Nursing Home Admission | -1,008 | 13,089 |
| Excluded because of use PDE5i OR EndoRecA | -68 | 13,021 |
| Excluded because patient did not begin follow-up | -74 | 12,947 |
| Patients in Endothelin receptor antagonists group | | 3,019 |
| Patients in PDE5 inhibitors group | | 9,928 |
| Final cohort | | 12,947 |

## 6. Variables

## a. Exposure-related variables:

### Study drug:

The study exposure of interest is initiation of PDE5 inhibitors (sildenafil, tadalafil)

### Comparator:

Endothelin receptor antagonists (bosentan, ambrisentan, macitentan)

## b. Covariates:

| Demographics | |
|--------------|-----------------------------|
| Age Region | |
| Gender | Calendar year of index date |
| Race | Low income subsidy |

| Dementia risk factors | |
|-------------------------------|---------------|
| Diabetes Depression | |
| Obesity | Anxiety |
| Hypertension Bipolar disorder | |
| Coronary artery disease | Schizophrenia |

| Markers for healthy behavior, frailty, healthcare use | |
|---|---|
| Smoking | Number of physician office visits |
| Mammography | Number of pulmonologist visits |
| Colonoscopy | Number of cardiologist visits |
| Fecal occult blood test | Number of serum creatinine tests ordered |
| Influenza vaccination | Composite frailty score |
| Pneumococcal vaccination | Number of C-reactive protein tests ordered |
| Herpes zoster vaccination | Osteoporosis |

| Bone mineral density test | Fractures |
|-----------------------------------|----------------------------|
| Number of distinct generic agents | Falls |
| Number of emergency room visits | Use of supplemental oxygen |
| Number of outpatient visits | Combined comorbidity score |
| Number of hospitalizations | |

| Other PAH treatments and PAH severity indicators | |
|---|---|
| Calcium channel blockers Prostanoids (Beraprost, Epoprosteno | |
| | lloprost, Treprostinil) |
| Riociguat | Number of hospitalization with PAH as the |
| | primary discharge diagnosis |

| Comedication use | |
|---|---|
| Lithium Nitrates | |
| Anti-epileptic mood stabilizers | Lipid lowering drugs |
| Anti-epileptics (other than mood stabilizers) | Non-insulin diabetes medications |
| Atypical antipsychotics | Insulin |
| Benzodiazepines | Antidepressants |
| Serotonin-norepinephrine reuptake Inhibitors | Typical antipsychotics |
| Selective serotonin reuptake inhibitors | itors Anticoagulants |
| Tricyclic antidepressants (TCAs) Antiplatelet agents | |
| SAMA/SABA | LAMA/LABA |
| Inhaled corticosteroids | nhaled corticosteroids Any DMARDs |

| Comorbid conditions | |
|---|---|
| Atrial fibrillation | Chronic liver disease |
| Coronary artery disease | Asthma |
| Heart failure | Ischemic heart disease |
| Stroke or transient ischemic attack | Chronic obstructive pulmonary disease |
| Peripheral vascular disease | Malignancy |
| Diabetes | Drug or alcohol abuse or dependence |
| Hyperlipidemia | Venous thromboembolism |

| Renal dysfunction | Hypertension |
|----------------------|------------------------------|
| Erectile dysfunction | Rheumatoid Arthritis |
| Raynaud's syndrome | Systemic lupus erythematosus |

ICD-9, ICD-10, HCPCS, and NDC codes used to define the covariates listed above are available in Appendix A.

- c. Outcome variables and study follow-up:
- <u>Primary outcome</u>: incident dementia, i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere. Outcome will be defined by 1 inpatient claim or 2 outpatient claims in analysis 1, 2, 3. In analysis 4, the outcome will be defined by 1 inpatient or 1 outpatient claims and 1 prescription claim for a symptomatic treatment [donepezil, galantamine, rivastigmine, and memantine] within 6 months of each other with outcome date assigned to second event in the sequence.
- Secondary outcomes: Individual component: Alzheimer's disease

| Condition | ICD-9 and ICD-10 codes |
|---|---|
| Alzheimer's disease | 331.0*, F00*, G30* |
| Vascular dementia | 290.4*, F01* |
| Senile, presenile, or unspecified dementia | 290.0*, 290.1*. 290.3*, 797*, F03* |
| Dementia in other diseases classified elsewhere | 331.1*, 331.2*, 331.7*, 294.1*, F02* |

For analysis 1,3, and 4 the follow-up will start the day after initiation of PDE5 inhibitors and endothelin receptor antagonists and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (PDE5 inhibitors and endothelin receptor antagonists) plus a defined grace period (i.e., 90 days after the end of the last prescription's days' supply in main analyses).

For analysis 2, the follow-up will start 180 days after initiation of PDE5 inhibitors and endothelin receptor antagonists and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Maximum allowed follow-up time (1095 days) reached

### 7. Feasibility counts

| Analysis scheme | Total PDE5<br>inhibitors/Endothelin<br>receptor antagonists | N outcome | Dementia Rate per 1,000<br>person-years (95% CI) | Follow-up time in days;<br>Median [IQR] |
|---|---|---|---|---|
| 1: As treated | 9,968 (76.6%) | 307 | 18.42 (16.36, 20.49) | 242 [64 .660] |
| | 3,053 (23.4%) | 307 | 18.42 (16.56, 20.43) | 242 [61, 669] |
| 2: 6 mo induction period, 'as started' | 5,453 (74.5%) | 286 | 22.20 (19.63, 24.77) | 638 [294, 1,095] |
| 1,871 (25.5%) | 200 | 22.20 (19.63, 24.77) | 030 [234, 1,033] | |
| 3: exclude 6 mo follow-up (symptoms | 5,416 (74.4%) | 238 | 19.79 (17.39, 22.43) | 422 [163, 844] |
| to claims period) | 1,866 (25.6%) | 236 | 13.73 (17.53, 22.43) | 422 [103, 844] |
| 4: Outcome Dx + Rx | 9,968 (76.6%) | 67 | 3.98 (3.02, 4.93) | 244 [61, 678] |
| | 3,053 (23.4%) | 07 | 3.98 (3.02, 4.93) | 244 [01, 078] |

### 8. Propensity score analysis

We will use a propensity-score (PS)²-based approach to account for measured confounding in this study. The PS will be calculated as the predicted probability of initiating the exposure of interest (i.e., the repurposing candidate) versus the reference drug conditional on baseline covariates using multivariable logistic regression constructed separately in each data source. On average, patients with similar PSs have similar distribution of potential confounders used to estimate the PS. Therefore, analyses conditioned on the PS provide effect estimates that are free from measured confounding. For all our analyses, initiators of each exposure of interest will be matched with initiators of the reference exposure based on their PS within each data source.³ Pair matching will be conducted using a nearest-neighbor algorithm, which seeks to minimize the distance between propensity scores in each pair of treated and reference patients,⁴ and a caliper of 0.025 on the natural scale of the PS will be used to ensure similarity between the matched patients.⁵

We report multiple diagnostics for PS analysis in this protocol. First, the PS distributional overlap is provided between two groups before and after matching to ensure comparability of these groups.<sup>6</sup> Next, balance in each individual covariate between two treatment groups is reported using standardized differences.<sup>7</sup>

## a. PS distributions stratified by treatment group

## Pre-matching propensity score overlap:



# Post-matching propensity score overlap:



# b. Table for covariate balance

| | Unmatched | | | PS-Matched | | |
|---|---|---|---|---|---|---|
| Variable | PDE5 inhibitors<br>(N = 9,968) | Endothelin<br>receptor<br>antagonists<br>(N = 3,053) | St.<br>Diff | PDE5 inhibitors<br>(N = 2,888) | Endothelin<br>receptor<br>antagonists<br>(N = 2,888) | St.<br>Diff |
| Demographics | | | | | | |
| Age, mean (SD) | 74.74 (6.78) | 73.79 (6.14) | 0.15 | 73.87 (6.43) | 73.84 (6.15) | 0.00 |
| Gender, n (%) | | | | | | 0.00 |
| Male | 3,899 (39.1%) | 936 (30.7%) | 0.18 | 889 (30.8%) | 898 (31.1%) | -0.01 |
| Female | 6,069 (60.9%) | 2,117 (69.3%) | -0.18 | 1,999 (69.2%) | 1,990 (68.9%) | 0.01 |
| Race, n (%) | | | | | | 0.00 |
| White | 8,031 (80.6%) | 2,435 (79.8%) | 0.02 | 2,293 (79.4%) | 2,311 (80.0%) | -0.01 |
| Black | 1,330 (13.3%) | 441 (14.4%) | -0.03 | 421 (14.6%) | 411 (14.2%) | 0.01 |
| Asian | 192 (1.9%) | 58 (1.9%) | 0.00 | 51 (1.8%) | 53 (1.8%) | 0.00 |
| Hispanic | 204 (2.0%) | 49 (1.6%) | 0.03 | 48 (1.7%) | 46 (1.6%) | 0.01 |
| Native American | 30 (0.3%) | 13 (0.4%) | -0.02 | 11 (0.4%) | 11 (0.4%) | 0.00 |
| Other | 136 (1.4%) | 42 (1.4%) | 0.00 | 49 (1.7%) | 41 (1.4%) | 0.02 |
| Unknown | 45 (0.5%) | 15 (0.5%) | 0.00 | 15 (0.5%) | 15 (0.5%) | 0.00 |
| Region, n (%) | | | | | | 0.00 |
| Northeast; n (%) | 1,737 (17.4%) | 461 (15.1%) | 0.06 | 431 (14.9%) | 439 (15.2%) | -0.01 |
| South; n (%) | 4,237 (42.5%) | 1,391 (45.6%) | -0.06 | 1,301 (45.0%) | 1,314 (45.5%) | -0.01 |
| Midwest; n (%) | 2,151 (21.6%) | 623 (20.4%) | 0.03 | 606 (21.0%) | 602 (20.8%) | 0.00 |
| West; n (%) | 1,822 (18.3%) | 568 (18.6%) | -0.01 | 550 (19.0%) | 533 (18.5%) | 0.01 |
| Missing; n (%) | 21 (0.2%) | 10 (0.3%) | -0.02 | | | 0.00 |
| Calendar year of index date, n (%) | | | | | | 0.00 |
| 2008 | 362 (3.6%) | 282 (9.2%) | -0.23 | 249 (8.6%) | 251 (8.7%) | 0.00 |

| 1 | 104 (4 004) | 076 (0.00() | | 0.00 (0.40() | 0.40 (0.60() | |
|---|---|---|---|---|---|---|
| 2009 | 401 (4.0%) | 276 (9.0%) | -0.20 | 262 (9.1%) | 249 (8.6%) | 0.02 |
| 2010 | 460 (4.6%) | 194 (6.4%) | -0.08 | 189 (6.5%) | 188 (6.5%) | 0.00 |
| 2011 | 444 (4.5%) | 190 (6.2%) | -0.08 | 176 (6.1%) | 185 (6.4%) | -0.01 |
| 2012 | 472 (4.7%) | 166 (5.4%) | -0.03 | 169 (5.9%) | 163 (5.6%) | 0.01 |
| 2013 | 1,676 (16.8%) | 515 (16.9%) | 0.00 | 512 (17.7%) | 513 (17.8%) | 0.00 |
| 2014 | 1,896 (19.0%) | 466 (15.3%) | 0.10 | 431 (14.9%) | 450 (15.6%) | -0.02 |
| 2015 | 1,593 (16.0%) | 396 (13.0%) | 0.09 | 381 (13.2%) | 374 (13.0%) | 0.01 |
| 2016 | 1,212 (12.2%) | 277 (9.1%) | 0.10 | 250 (8.7%) | 260 (9.0%) | -0.01 |
| 2017 | 974 (9.8%) | 172 (5.6%) | 0.16 | 161 (5.6%) | 152 (5.3%) | 0.01 |
| 2018 | 478 (4.8%) | 119 (3.9%) | 0.04 | 108 (3.7%) | 103 (3.6%) | 0.01 |
| Low income subsidy, n (%) | 2,382 (23.9%) | 713 (23.4%) | 0.01 | 706 (24.4%) | 682 (23.6%) | 0.02 |
| Dementia risk factors, n (%) | | | | | | 0.00 |
| Diabetes | 4,486 (45.0%) | 1,204 (39.4%) | 0.11 | 1,180 (40.9%) | 1,145 (39.6%) | 0.03 |
| Obesity | 3,351 (33.6%) | 968 (31.7%) | 0.04 | 911 (31.5%) | 918 (31.8%) | -0.01 |
| Hypertension | 8,877 (89.1%) | 2,729 (89.4%) | -0.01 | 2,587 (89.6%) | 2,595 (89.9%) | -0.01 |
| Coronary artery disease | 7,445 (74.7%) | 2,273 (74.5%) | 0.00 | 2,136 (74.0%) | 2,150 (74.4%) | -0.01 |
| Depression | 1,995 (20.0%) | 571 (18.7%) | 0.03 | 515 (17.8%) | 537 (18.6%) | -0.02 |
| Anxiety | 1,824 (18.3%) | 494 (16.2%) | 0.06 | 466 (16.1%) | 465 (16.1%) | 0.00 |
| Bipolar disorder | 88 (0.9%) | 33 (1.1%) | -0.02 | 28 (1.0%) | 32 (1.1%) | -0.01 |
| Schizophrenia | 26 (0.3%) | 12 (0.4%) | -0.02 | 12 (0.4%) | 12 (0.4%) | 0.00 |
| Markers for healthy behavior, frailty, | | | | | | |
| healthcare use | | | | | | 0.00 |
| Smoking, n (%) | 4,286 (43.0%) | 1,126 (36.9%) | 0.12 | 1,056 (36.6%) | 1,068 (37.0%) | -0.01 |
| Mammography, n (%) | 1,743 (17.5%) | 630 (20.6%) | -0.08 | 593 (20.5%) | 597 (20.7%) | 0.00 |
| Colonoscopy, n (%) | 1,239 (12.4%) | 345 (11.3%) | 0.03 | 327 (11.3%) | 317 (11.0%) | 0.01 |
| Fecal occult blood test, n (%) | 774 (7.8%) | 238 (7.8%) | 0.00 | 232 (8.0%) | 223 (7.7%) | 0.01 |
| Influenza vaccination, n (%) | 6,953 (69.8%) | 2,150 (70.4%) | -0.01 | 2,037 (70.5%) | 2,036 (70.5%) | 0.00 |

| Pneumococcal vaccination, n (%) | 3,134 (31.4%) | 764 (25.0%) | 0.14 | 696 (24.1%) | 713 (24.7%) | -0.01 |
|---|---|---|---|---|---|---|
| Number of distinct prescriptions, mean | | | | | | |
| (SD) | 17.94 (6.76) | 17.54 (6.82) | 0.06 | 17.73 (6.72) | 17.56 (6.83) | 0.03 |
| Number of emergency room visits, mean | | | | | | |
| (SD) | 1.50 (2.02) | 1.25 (1.74) | 0.13 | 1.31 (1.85) | 1.25 (1.75) | 0.03 |
| Number of outpatient visits, mean (SD) | 21.99 (19.80) | 22.66 (19.58) | -0.03 | 22.95 (23.37) | 22.70 (19.84) | 0.01 |
| Number of hospitalizations, mean (SD) | 1.54 (1.77) | 1.14 (1.56) | 0.24 | 1.19 (1.47) | 1.15 (1.58) | 0.03 |
| Number of physician office visits, mean (SD) | 6.31 (10.05) | 6.56 (9.61) | -0.03 | 6.65 (11.64) | 6.60 (9.73) | 0.00 |
| Number of cardiologist visits, mean (SD) | 10.14 (10.08) | 8.24 (7.26) | 0.22 | 8.27 (7.64) | 8.29 (7.30) | 0.00 |
| Number of pulmonologist visits, mean (SD) | 4.38 (5.12) | 4.89 (4.77) | -0.10 | 4.82 (5.53) | 4.83 (4.70) | 0.00 |
| Number of C-reactive protein tests ordered, mean (SD) | 0.35 (1.04) | 0.39 (1.04) | -0.04 | 0.40 (1.13) | 0.38 (1.00) | 0.02 |
| Number of serum creatinine tests ordered, mean (SD) | 6.96 (5.60) | 6.30 (4.54) | 0.13 | 6.31 (4.89) | 6.28 (4.54) | 0.01 |
| Composite frailty score, mean (SD) | 0.26 (0.07) | 0.26 (0.06) | 0.00 | 0.26 (0.07) | 0.26 (0.06) | 0.00 |
| Osteoporosis, n (%) | 1,340 (13.4%) | 488 (16.0%) | -0.07 | 451 (15.6%) | 460 (15.9%) | -0.01 |
| Fractures, n (%) | 803 (8.1%) | 235 (7.7%) | 0.01 | 216 (7.5%) | 220 (7.6%) | 0.00 |
| Falls, n (%) | 512 (5.1%) | 148 (4.8%) | 0.01 | 136 (4.7%) | 142 (4.9%) | -0.01 |
| Use of supplemental oxygen, n (%) | 2,385 (23.9%) | 629 (20.6%) | 0.08 | 611 (21.2%) | 602 (20.8%) | 0.01 |
| Combined comorbidity score, mean (SD) | 8.73 (2.81) | 7.95 (2.64) | 0.29 | 8.00 (2.71) | 7.98 (2.63) | 0.01 |
| Comedication use, n (%) | | | | | | 0.00 |
| Lithium | 7 (0.1%) | 6 (0.2%) | -0.03 | 3 (0.1%) | 4 (0.1%) | 0.00 |
| Anti-epileptic mood stabilizers | 98 (1.0%) | 32 (1.0%) | 0.00 | 24 (0.8%) | 29 (1.0%) | -0.02 |
| Anti-epileptics (other than mood stabilizers) | 1,940 (19.5%) | 590 (19.3%) | 0.01 | 571 (19.8%) | 558 (19.3%) | 0.01 |
| Atypical antipsychotics | 167 (1.7%) | 54 (1.8%) | -0.01 | 43 (1.5%) | 53 (1.8%) | -0.02 |
| Benzodiazepines | 1,868 (18.7%) | 460 (15.1%) | 0.10 | 428 (14.8%) | 433 (15.0%) | -0.01 |

| Serotonin-norepinephrine reuptake | | | | | | |
|---|---|---|---|---|---|---|
| inhibitors | 479 (4.8%) | 196 (6.4%) | -0.07 | 186 (6.4%) | 184 (6.4%) | 0.00 |
| Selective serotonin reuptake inhibitors | 2,132 (21.4%) | 711 (23.3%) | -0.05 | 658 (22.8%) | 667 (23.1%) | -0.01 |
| Tricyclic antidepressants (TCAs) | 447 (4.5%) | 138 (4.5%) | 0.00 | 120 (4.2%) | 127 (4.4%) | -0.01 |
| Typical antipsychotics | 16 (0.2%) | 8 (0.3%) | -0.02 | 6 (0.2%) | 7 (0.2%) | 0.00 |
| Anticoagulants | 4,462 (44.8%) | 1,175 (38.5%) | 0.13 | 1,121 (38.8%) | 1,102 (38.2%) | 0.01 |
| Antiplatelet agents | 1,853 (18.6%) | 610 (20.0%) | -0.04 | 570 (19.7%) | 576 (19.9%) | -0.01 |
| Nitrates | 2,132 (21.4%) | 753 (24.7%) | -0.08 | 716 (24.8%) | 712 (24.7%) | 0.00 |
| Lipid lowering drugs | 7,020 (70.4%) | 2,149 (70.4%) | 0.00 | 2,020 (69.9%) | 2,030 (70.3%) | -0.01 |
| Non-insulin diabetes medications | 4,036 (40.5%) | 1,421 (46.5%) | -0.12 | 1,358 (47.0%) | 1,347 (46.6%) | 0.01 |
| Insulin | 2,250 (22.6%) | 725 (23.7%) | -0.03 | 714 (24.7%) | 696 (24.1%) | 0.01 |
| Antidepressants | 3,244 (32.5%) | 1,067 (34.9%) | -0.05 | 983 (34.0%) | 1,002 (34.7%) | -0.01 |
| SAMA/SABA | 3,624 (36.4%) | 1,070 (35.0%) | 0.03 | 1,083 (37.5%) | 1,016 (35.2%) | 0.05 |
| LAMA/LABA | 152 (1.5%) | 31 (1.0%) | 0.05 | 29 (1.0%) | 28 (1.0%) | 0.00 |
| Inhaled corticosteroids | 469 (4.7%) | 158 (5.2%) | -0.02 | 155 (5.4%) | 151 (5.2%) | 0.01 |
| Any DMARDs | 717 (7.2%) | 285 (9.3%) | -0.08 | 264 (9.1%) | 261 (9.0%) | 0.00 |
| Other PAH treatments and PAH severity indicators, n (%) | | | | | | 0.00 |
| Use of calcium channel blockers | 4,652 (46.7%) | 1,506 (49.3%) | -0.05 | 1,462 (50.6%) | 1,422 (49.2%) | 0.03 |
| Riociguat | 26 (0.3%) | 90 (2.9%) | -0.21 | 26 (0.9%) | 25 (0.9%) | 0.00 |
| Prostanoids | 96 (1.0%) | 55 (1.8%) | -0.07 | 54 (1.9%) | 48 (1.7%) | 0.02 |
| Number of hospitalization with PAH as the primary discharge diagnosis | 0.10 (0.34) | 0.11 (0.35) | -0.03 | 0.12 (0.37) | 0.11 (0.34) | 0.03 |
| Comorbid conditions, n (%) | | | | | | 0.00 |
| Atrial fibrillation | 5,321 (53.4%) | 1,282 (42.0%) | 0.23 | 1,232 (42.7%) | 1,228 (42.5%) | 0.00 |
| Heart failure | 8,064 (80.9%) | 2,197 (72.0%) | 0.21 | 2,088 (72.3%) | 2,088 (72.3%) | 0.00 |
| Stroke or transient ischemic attack | 1,020 (10.2%) | 276 (9.0%) | 0.04 | 254 (8.8%) | 260 (9.0%) | -0.01 |

| Peripheral vascular disease | 2,637 (26.5%) | 748 (24.5%) | 0.05 | 707 (24.5%) | 724 (25.1%) | -0.01 |
|---|---|---|---|---|---|---|
| Hyperlipidemia | 8,503 (85.3%) | 2,606 (85.4%) | 0.00 | 2,463 (85.3%) | 2,461 (85.2%) | 0.00 |
| Renal dysfunction | 5,227 (52.4%) | 1,318 (43.2%) | 0.18 | 1,263 (43.7%) | 1,266 (43.8%) | 0.00 |
| Chronic liver disease | 1,524 (15.3%) | 365 (12.0%) | 0.10 | 330 (11.4%) | 344 (11.9%) | -0.02 |
| Asthma | 3,575 (35.9%) | 1,034 (33.9%) | 0.04 | 981 (34.0%) | 965 (33.4%) | 0.01 |
| Ischemic heart disease | 7,148 (71.7%) | 2,204 (72.2%) | -0.01 | 2,060 (71.3%) | 2,084 (72.2%) | -0.02 |
| Chronic obstructive pulmonary disease | 6,521 (65.4%) | 2,020 (66.2%) | -0.02 | 1,941 (67.2%) | 1,915 (66.3%) | 0.02 |
| Malignancy | 3,064 (30.7%) | 847 (27.7%) | 0.07 | 806 (27.9%) | 799 (27.7%) | 0.00 |
| Drug or alcohol abuse or dependence | 1,172 (11.8%) | 277 (9.1%) | 0.09 | 249 (8.6%) | 262 (9.1%) | -0.02 |
| Venous thromboembolism | 1,725 (17.3%) | 583 (19.1%) | -0.05 | 526 (18.2%) | 522 (18.1%) | 0.00 |
| Erectile dysfunction | 343 (3.4%) | 49 (1.6%) | 0.12 | 41 (1.4%) | 49 (1.7%) | -0.02 |
| Rheumatoid Arthritis | 788 (7.9%) | 267 (8.7%) | -0.03 | 279 (9.7%) | 249 (8.6%) | 0.04 |
| Raynaud's syndrome | 359 (3.6%) | 162 (5.3%) | -0.08 | 161 (5.6%) | 151 (5.2%) | 0.02 |
| Systemic lupus erythematosus | 185 (1.9%) | 106 (3.5%) | -0.10 | 88 (3.0%) | 90 (3.1%) | -0.01 |

#### 9. Statistical analysis plans

Incidence rates for the outcome will be estimated for the treatment and reference groups before and after PS matching. The competing risk of death could be of concern for the current set of analyses if mortality is frequent among patients included in the cohort and if differences in the risk of mortality between treatment and reference groups are substantial. In the PS-matched sample, we will use cause-specific hazard models<sup>8</sup> to provide hazard ratios averaged over the entire follow-up period as well as interval specific hazard ratios (1, 2, and 3 years) for the association between the treatment of interest and risk of ADRD after considering all-cause mortality as a competing event. Pre-specified subgroup analyses will be conducted based on age, sex, and baseline cardiovascular disease.

#### 10. References

- 1. Sprecher VP, Didden E-M, Swerdel JN, Muller A. Evaluation of code-based algorithms to identify pulmonary arterial hypertension and chronic thromboembolic pulmonary hypertension patients in large administrative databases. *Pulmonary circulation*. 2020;10(4):2045894020961713.
- **2.** Rosenbaum PR, Rubin DB. The central role of the propensity score in observational studies for causal effects. *Biometrika*. 1983;70(1):41-55.
- 3. Rassen JA, Avorn J, Schneeweiss S. Multivariate-adjusted pharmacoepidemiologic analyses of confidential information pooled from multiple health care utilization databases. *Pharmacoepidemiology and drug safety.* 2010;19(8):848-857.
- **4.** Rassen JA, Shelat AA, Myers J, Glynn RJ, Rothman KJ, Schneeweiss S. One-to-many propensity score matching in cohort studies. *Pharmacoepidemiol Drug Saf.* May 2012;21 Suppl 2:69-80.
- **5.** Austin PC. Some Methods of Propensity-Score Matching had Superior Performance to Others: Results of an Empirical Investigation and Monte Carlo simulations. *Biometrical Journal*. 2009;51(1):171-184.
- **6.** AM Walker AM, Patrick A, Lauer M, et al. Tool for Assessing the Feasibility of Comparative Effectiveness Research. *Comp Effect Res* 2013;3:11-20.
- 7. Franklin JM, Rassen JA, Ackermann D, Bartels DB, Schneeweiss S. Metrics for covariate balance in cohort studies of causal effects. *Statistics in medicine*. May 10 2014;33(10):1685-1699.
- **8.** Austin PC, Lee DS, Fine JP. Introduction to the analysis of survival data in the presence of competing risks. *Circulation.* 2016;133(6):601-609.

| # | Implementation in routine care | |
|---|---|---|
| | | EXPOSURE vs. COMPARISON |
| | PDE5 inhibitors vs Endothelin recepto | rantagonists |
| | | INCLUSION CRITERIA |
| 1 | Age | Aged > 65 years on the index date |
| 2 | No prior use of study drugs Depending on the comparison group, we will require new-use (defined as no an anytime prior to index date) of PDE5 inhibitors (sildenafil, tadalafil) and endot receptor antagonists (bosentan, ambrisentan, macitentan) | |
| 3 | Sufficient enrollment Medicare Part A, B, and D enrollment with no HMO coverage for 365 days pri and on the cohort entry date | |
| | | EXCLUSION CRITERIA |
| | Prior history of dementia | Measured any time prior to drug initiation in any diagnosis position and inpatient or outpatient setting – |
| | | ICD9 diagnosis – 046.1x, 290.xx (excluding 290.8), 291.2, 292.82, 294.1x, 294.2x, 331.0-331.2, 331.7, 331.82, 331.83, 333.4, 780.93, 797 ICD10 diagnosis – F01.xx-F03.xx, G30.xx-G31.85, R41.xx |
| 1 | | NDC brand name – ""ARICEPT", "ARICEPT ODT", "EXELON", "NAMENDA", "NAMENDA XR", "NAMZARIC", "RAZADYNE", "RAZADYNE ER", or "REMINYL" |
| | | NDC generic name — "DONEPEZIL HCL", "GALANTAMINE HBR", "MEMANTINE HCL", "MEMANTINE HCL/DONEPEZIL HCL", "RIVASTIGMINE", or "RIVASTIGMINE TARTRATE" |
| | No prior history of pulmonary arterial hypertension | Measured 365 days prior to drug initiation in any diagnosis position and inpatient or outpatient setting – |
| 2 | | ICD9 diagnosis – 416.0, 416.8, 416.9<br>ICD10 diagnosis – I27.0, I27.2, I27.8, I27.9 |
| | Nursing home admission | Measured 365 days prior to drug initiation – |
| 3 | | MEDPAR - Short Stay/Long Stay/SNF Indicator Code — N = SNF Stay (Prvdr3 = 5, 6, U W, Y, or Z) |

## **Covariate list Potential confounders** Category ICD-9 Age Gender Race **Demographics** Region Calendar year of index date Low income subsidy Diabetes Obesity Hypertension Coronary artery disease **Dementia risk factors** Depression Anxiety Bipolar disorder Schizophrenia **Smoking** Mammography Colonoscopy Fecal occult blood test Lifestyle factors and markers for healthy behavior Influenza vaccination Pneumococcal vaccination Herpes zoster vaccination BMD test Number of distinct generic agents Number of emergency room visits Number of outpatient visits Number of hospitalizations Healthcare utilization measures Number of physician office visits Number of cardiologist visits Number of pulmonologist visits Number of CRP tests ordered Number of serum creatinine tests ordered Composite frailty score Osteoporosis Fractures Frailty markers Falls Use of supplemental oxygen A combined comorbidity score

| | Lithium |
|---|---|
| | Anti-epileptic mood stabilizers |
| | Anti-epileptics (other than mood stabilizers) |
| | Atypical antipsychotics |
| | Benzodiazepines |
| | SNRIs |
| | SSRIs |
| | TCAs |
| | Typical antipsychotics |
| | Anticoagulants |
| Comedications | Antiplatelet agents |
| | Nitrates |
| | Lipid lowering drugs |
| | Non-insulin diabetes medications |
| | Insulin |
| | Antidepressants |
| | SAMA/SABA |
| | LAMA/LABA Inhaled corticosteroids |
| | Any DMARDs |
| | Calcium channel blockers |
| | Riociguat |
| Other PAH treatments and PAH severity indicators | Prostanoids (Beraprost, Epoprostenol, Iloprost, |
| · | (reprostinii) |
| | Number of hospitalization with PAH as the primary |
| | discharge diagnosis |
| | Atrial fibrillation |
| | Coronary artery disease |
| | Heart failure |
| | Stroke or TIA |
| | Peripheral vascular disease |
| | Hypertension |
| | Diabetes |
| | Hyperlipidemia |
| | Renal dysfunction |
| Comorbid conditions | Chronic liver disease |
| Comorbia Conditions | Asthma |
| | Ischemic heart disease |
| | isometric real carsease |
| | COPD |
| | COPD |
| | COPD<br>Malignancy |
| | COPD Malignancy Drug or alcohol abuse or dependence |
| | COPD Malignancy Drug or alcohol abuse or dependence VTE |
| | COPD Malignancy Drug or alcohol abuse or dependence VTE Erectile dysfunction |

## Demographics

| Calendar year of index date |
|-----------------------------|
| Year |
| 2007 |
| 2008 |
| 2009 |
| 2010 |
| 2011 |
| 2012 |
| 2013 |
| 2014 |
| 2015 |
| 2016 |
| 2017 |

#### Low income subsidy

https://www.cms.gov/Medicare/Eligibility-and-

Enrollment/LowIncSubMedicarePresCov/Downloads/StateLISGuidance021009.pd

£

#### Diabetes


### Dementia risk factors


#### Obesity


#### Dementia risk factors


Hypertension

Sibutramine
Phentermine
Benzphetamine
Phendimetrazine
Diethylpropion

| Hypertension | | | |
|---|---|---|---|
| ICD10 Dx | ICD9 Dx | LongDeslCD10 | LongDeslCD9 |
| I10 | 4010 | Essential (primary) hypertension | Malignant essential hypertension |
| I10 | 4011 | Essential (primary) hypertension | Benign essential hypertension |
| I10 | 4019 | Essential (primary) hypertension | Unspecified essential hypertension |
| I160 | 4019 | Hypertensive urgency | Unspecified essential hypertension |
| l161 | 4019 | Hypertensive emergency | Unspecified essential hypertension |
| I169 | 4019 | Hypertensive crisis, unspecified | Unspecified essential hypertension |
| l119 | 40200 | Hypertensive heart disease without heart failure | Malignant hypertensive heart disease without heart failure |
| l110 | 40201 | Hypertensive heart disease with heart failure | Malignant hypertensive heart disease with heart failure |
| l119 | 40210 | Hypertensive heart disease without heart failure | Benign hypertensive heart disease without heart failure |
| l110 | 40211 | Hypertensive heart disease with heart failure | Benign hypertensive heart disease with heart failure |
| l119 | 40290 | Hypertensive heart disease without heart failure | Unspecified hypertensive heart disease without heart failure |
| l110 | 40291 | Hypertensive heart disease with heart failure | Unspecified hypertensive heart disease with heart failure |
| 1129 | 40300 | Hypertensive chronic kidney disease with stage 1 through stage 4 chronic kidney disease, or unspecified chronic kidney disease | Hypertensive chronic kidney disease, malignant, with chronic kidney disease stage I through stage IV, or unspecified |
| l120 | 40301 | Hypertensive chronic kidney disease with stage 5 chronic kidney disease or end stage renal disease | Hypertensive chronic kidney disease, malignant, with chronic kidney disease stage V or end stage renal disease |
| l129 | 40310 | Hypertensive chronic kidney disease with stage 1 through | Hypertensive chronic kidney disease, benign, with chronic |
| | | stage 4 chronic kidney disease, or unspecified chronic kidney disease | , |
| l120 | 40311 | Hypertensive chronic kidney disease with stage 5 chronic | Hypertensive chronic kidney disease, benign, with chronic |
| | | kidney disease or end stage renal disease | kidney disease stage V or end stage renal disease |
| l129 | 40390 | Hypertensive chronic kidney disease with stage 1 through stage 4 chronic kidney disease, or unspecified chronic kidney disease | Hypertensive chronic kidney disease, unspecified, with chronic kidney disease stage I through stage IV, or unspecified |
| l120 | 40391 | Hypertensive chronic kidney disease with stage 5 chronic kidney disease or end stage renal disease | Hypertensive chronic kidney disease, unspecified, with chronic kidney disease stage V or end stage renal disease |
| I1310 | 40400 | Hypertensive heart and chronic kidney disease without heart failure, with stage 1 through stage 4 chronic kidney disease, or unspecified chronic kidney disease | Hypertensive heart and chronic kidney disease, malignant, without heart failure and with chronic kidney disease stage I through stage IV, or unspecified |
| l130 | 40401 | Hypertensive heart and chronic kidney disease with heart failure and stage 1 through stage 4 chronic kidney disease, or unspecified chronic kidney disease | Hypertensive heart and chronic kidney disease, malignant, with heart failure and with chronic kidney disease stage I through stage IV, or unspecified |

#### Dementia risk factors

| l1311 | 40402 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, malignant, |
|---|---|---|---|
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| l132 | 40403 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, malignant, |
| | | failure and with stage 5 chronic kidney disease, or end | with heart failure and with chronic kidney disease stage V |
| | | stage renal disease | or end stage renal disease |
| I1310 | 40410 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, benign, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | I through stage IV, or unspecified |
| I130 | 40411 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, benign, with |
| | | failure and stage 1 through stage 4 chronic kidney disease, | heart failure and with chronic kidney disease stage I |
| | | or unspecified chronic kidney disease | through stage IV, or unspecified |
| l1311 | 40412 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, benign, |
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| l132 | 40413 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, benign, with |
| | | failure and with stage 5 chronic kidney disease, or end | heart failure and chronic kidney disease stage V or end |
| | | stage renal disease | stage renal disease |
| I1310 | 40490 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, unspecified, |
| | | heart failure, with stage 1 through stage 4 chronic kidney | without heart failure and with chronic kidney disease stage |
| | | disease, or unspecified chronic kidney disease | I through stage IV, or unspecified |
| I130 | 40491 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, unspecified, |
| | | failure and stage 1 through stage 4 chronic kidney disease, | with heart failure and with chronic kidney disease stage I |
| | | or unspecified chronic kidney disease | through stage IV, or unspecified |
| 11311 | 40492 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, unspecified, |
| | | heart failure, with stage 5 chronic kidney disease, or end | without heart failure and with chronic kidney disease stage |
| | | stage renal disease | V or end stage renal disease |
| 1132 | 40493 | Hypertensive heart and chronic kidney disease with heart | Hypertensive heart and chronic kidney disease, unspecified, |
| | | failure and with stage 5 chronic kidney disease, or end | with heart failure and chronic kidney disease stage V or end |
| | | stage renal disease | stage renal disease |
| I150 | 40501 | Renovascular hypertension | Malignant renovascular hypertension |
| I158 | 40509 | Other secondary hypertension | Other malignant secondary hypertension |
| I150 | 40511 | Renovascular hypertension | Benign renovascular hypertension |
| I158 | 40519 | Other secondary hypertension | Other benign secondary hypertension |
| I150 | 40591 | Renovascular hypertension | Unspecified renovascular hypertension |
| l151 | 40591 | Hypertension secondary to other renal disorders | Unspecified renovascular hypertension |
| N262 | 40591 | Page kidney | Unspecified renovascular hypertension |
| I152 | 40599 | Hypertension secondary to endocrine disorders | Other unspecified secondary hypertension |
| I158 | 40599 | Other secondary hypertension | Other unspecified secondary hypertension |
| I159 | 40599 | Secondary hypertension, unspecified | Other unspecified secondary hypertension |

#### onary artery disease


#### Dementia risk factors


| Dementia risl | k factors | |
|---------------|-----------|----------------|
| 33519 | | |
| 33520 | | |
| 33521 | | |
| 33522 | | |
| 33523 | | |
| 33524 | | |
| 33525 | | |
| 33526 | | |
| 33527 | | |
| 33528 | | |
| 33529 | | |
| 33530 | | |
| 33531 | | |
| 33532 | | |
| 33533 | | |
| 33534 | | |
| 33535 | | |
| 33536 | | |
| 33545 | | |
| 33572 | | |
| CPT | | |
| 92973 | | |
| 92982 | | |
| 92984 | | |
| 92995 | | |
| 92996 | | |
| 92920 | | |
| 92921 | | |
| 92924 | | |
| 92925 | | |
| 92937 | | |
| 92938 | | |
| 92941 | | |
| 92943 | | |
| 92944 | | I |
| ICD10 Dx | ICD9 Dx | LongDeslCD |
| 1208 | 4130 | Other forms of |
| 1201 | 4131 | Angina pector |
| 1201 | 4131 | Tugina pecior |
| 1208 | 4139 | Other forms of |
| 1209 | 4139 | Angina pector |
| | | Atheroscleroti |
| | 1 | |


| | | Dilation of Coronary Artery, Four or More | Insertion of |
|---|---|---|---|
| | | Arteries, Bifurcation, with Two Drug-eluting | drug-eluting |
| | | Intraluminal Devices, Percutaneous | coronary artery |
| 0273456 | 3607 | Endoscopic Approach | stent(s) |
| | | Dilation of Coronary Artery, Four or More | Insertion of |
| | | Arteries with Two Drug-eluting Intraluminal | drug-eluting |
| | | Devices, Percutaneous Endoscopic | coronary artery |
| 027345Z | 3607 | Approach | stent(s) |
| | | Dilation of Coronary Artery, Four or More | Insertion of |
| | | Arteries, Bifurcation, with Three Drug-eluting | drug-eluting |
| | | Intraluminal Devices, Percutaneous | coronary artery |
| 0273466 | 3607 | Endoscopic Approach | stent(s) |
| | | Dilation of Coronary Artery, Four or More | Insertion of |
| | | Arteries with Three Drug-eluting Intraluminal | drug-eluting |
| | | Devices, Percutaneous Endoscopic | coronary artery |
| 027346Z | 3607 | Approach | stent(s) |
| | | Dilation of Coronary Artery, Four or More | Insertion of |
| | | Arteries, Bifurcation, with Four or More | drug-eluting |
| | | Drug-eluting Intraluminal Devices, | coronary artery |
| 0273476 | 3607 | Percutaneous Endoscopic Approach | stent(s) |
| | | Dilation of Coronary Artery, Four or More | Insertion of |
| | | Arteries with Four or More Drug-eluting | drug-eluting |
| | | Intraluminal Devices, Percutaneous | coronary artery |
| 027347Z | 3607 | Endoscopic Approach | stent(s) |
| | | | Insertion of |
| | | | drug-eluting |
| | | | coronary artery |
| NoPCS | 3607 | | stent(s) |
| СРТ | | | |
| | 4 | | |
| 92980 | _ | | |
| 92980<br>92981 | ] | | |
| | - | | |
| 92981<br>92928 | - | | |
| 92981<br>92928<br>92929 | - | | |
| 92981<br>92928<br>92929<br>92933 | | | |
| 92981<br>92928<br>92929 | | | |
| 92981<br>92928<br>92929<br>92933 | ICD9 Dx | LongDeslCD10 | LongDesICD9 |
| 92981<br>92928<br>92929<br>92933<br>92934 | ICD9 Dx | Long DeslCD10 | LongDesICD9 Postmyocardial |
| 92981<br>92928<br>92929<br>92933<br>92934 | ICD9 Dx<br>4110 | LongDesICD10 Dressler's syndrome | |
| 92981<br>92928<br>92929<br>92933<br>92934<br>ICD10 Dx | | | Postmyocardial |
| 92981<br>92928<br>92929<br>92933<br>92934<br>ICD10 Dx | | Dressler's syndrome Unstable angina | Postmyocardial infarction syndrome |
| 92981 92928 92929 92933 92934 ICD10 Dx | 4110 | Dressler's syndrome | Postmyocardial infarction syndrome Intermediate |
| 92981 92928 92929 92933 92934 ICD10 Dx | 4110 | Dressler's syndrome Unstable angina | Postmyocardial infarction syndrome Intermediate |
| 92981 92928 92929 92933 92934 ICD10 Dx | 4110 | Dressler's syndrome Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris | Postmyocardial infarction syndrome Intermediate coronary syndrome |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 | 4110 | Dressler's syndrome Unstable angina Atherosclerotic heart disease of native coronary artery with | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 | 4110 | Dressler's syndrome Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 | 4110 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 | 4110<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 | 4110<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 | 4110<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 125110 | 4110<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 125110 | 4110<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 125110 | 4110<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 125110 | 4110<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 125710 | 4110<br>4111<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate Intermediate Intermediate Intermediate Intermediate |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 125710 | 4110<br>4111<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina pectoris | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate Intermediate Intermediate Intermediate Intermediate |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 125710 | 4110<br>4111<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of nonautologous | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate coronary syndrome Intermediate Intermediate Intermediate Intermediate Intermediate |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 125710 | 4110<br>4111<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of nonautologous biological coronary artery bypass | Postmyocardial infarction syndrome Intermediate coronary syndrome |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 125710 | 4110<br>4111<br>4111<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of nonautologous biological coronary artery bypass graft(s) with unstable angina | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate Intermediate Intermediate Intermediate Intermediate |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 125710 | 4110<br>4111<br>4111<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of nonautologous biological coronary artery bypass graft(s) with unstable angina pectoris | Postmyocardial infarction syndrome Intermediate coronary syndrome Intermediate Intermediate Intermediate Intermediate Intermediate |
| 92981 92928 92929 92933 92934 ICD10 Dx 1241 1200 125710 | 4110<br>4111<br>4111<br>4111<br>4111<br>4111 | Unstable angina Atherosclerotic heart disease of native coronary artery with unstable angina pectoris Atherosclerosis of coronary artery bypass graft(s), unspecified, with unstable angina pectoris Atherosclerosis of autologous vein coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of autologous artery coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of nonautologous biological coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of nonautologous biological coronary artery bypass graft(s) with unstable angina pectoris Atherosclerosis of native coronary | Postmyocardial infarction syndrome Intermediate coronary syndrome |

#### Dementia risk factors


Depression


### Dementia risk factors


Anxiety

#### Dementia risk factors


#### Bipolar disorder


#### Dementia risk factors


Schizophrenia


#### Dementia risk factors


Lifestyle factors and markers for healthy behavior

#### **Smoking**


CPT codes
99406
99407
G0436
G0437
G9016
S9453
S4995
G9276
G9458
1034F
4001F
4004F

OR dispensing of: At least one nicotine or varenicline prescription

#### Mammography


Colonoscopy


**CPT**45378
45379

111

Lifestyle factors and markers for healthy behavior

| 45380 | |
|-------|---|
| 45381 | |
| 45382 | |
| 45383 | |
| 45384 | |
| 45385 | |
| 45386 | |
| 45387 | |
| 45388 | |
| 45389 | |
| 45390 | |
| 45391 | |
| 45392 | |
| HCPCS | • |
| G0105 | |
| G0121 | |

#### Fecal occult blood test


#### Influenza vaccination


#### **Pneumococcal vaccination**


Lifestyle factors and markers for healthy behavior

| 90670 |
|-------|
| 90732 |

#### Herpes zoster vaccination


#### BMD test

| CPT |
|-------|
| 76070 |
| 76075 |
| 76076 |
| 76977 |
| 77080 |
| 77085 |

#### Healthcare utilization

#### Number of generic medications

NDC generic drug name has any value

If multiple events on a single day, the value is measured as combined values.

#### Number of ED visits

| HCPCS | | | | | |
|-------|-------|-------|-------|-------|-------|
| 99281 | 99282 | 99283 | 99284 | 99285 | 99288 |

#### Number of outpatient visits

| HCPCS | | | | | |
|-------|-------|-------|-------|-------|-------|
| 99201 | 99214 | 99272 | 99381 | 99392 | 99403 |
| 99202 | 99215 | 99273 | 99382 | 99393 | 99404 |
| 99203 | 99241 | 99274 | 99383 | 99394 | 99420 |
| 99204 | 99242 | 99275 | 99384 | 99395 | 99450 |
| 99205 | 99243 | 99354 | 99385 | 99396 | 99455 |
| 99211 | 99244 | 99355 | 99386 | 99397 | 99456 |
| 99212 | 99245 | 99356 | 99387 | 99401 | 99499 |
| 99213 | 99271 | 99357 | 99391 | 99402 | |

#### Number of hospitalizations

The occurrence of MEDPAR with the following attributes:

Inpatient admission type code exists

The occurrence of carrier claims with the following attributes:

20 = Non swing bed SNF claim

30 = Swing bed SNF claim

50 = Hospice claim

60 = Inpatient claim

61 = Inpatient 'full-encounter' claim

#### Number of PCP visits

The occurrence of carrier claims line with the following attributes:

Line HCFA provider specialty code is any of:

01 = General practice

08 = Family practice

11 = Internal medicine

84 = Preventive medicine (eff 5/92)

| HCPCS | | | | | |
|-------|-------|-------|-------|-------|-------|
| 99201 | 99214 | 99272 | 99381 | 99392 | 99403 |
| 99202 | 99215 | 99273 | 99382 | 99393 | 99404 |
| 99203 | 99241 | 99274 | 99383 | 99394 | 99420 |
| 99204 | 99242 | 99275 | 99384 | 99395 | 99429 |
| 99205 | 99243 | 99354 | 99385 | 99396 | 99450 |
| 99211 | 99244 | 99355 | 99386 | 99397 | 99455 |
| 99212 | 99245 | 99356 | 99387 | 99401 | 99456 |
| 99213 | 99271 | 99357 | 99391 | 99402 | 99499 |

#### **Number of Cardiologist visits**

The occurrence of carrier claims line with the following attributes:

Line HCFA provider specialty code is any of:

06 = Cardiology

#### Number of Pulmonologist visits

The occurrence of carrier claims line with the following attributes:

Line HCFA provider specialty code is any of:

29 = Pulmonary disease

#### Number of CRP tests


#### Number of serum creatinine tests

| CPT | |
|-------|-------|
| 80048 | 80054 |
| 80049 | 80069 |
| 80053 | 82565 |

#### Frailty markers

#### Frailty Score for Claims Data

Kim DH. Schneeweiss S. Glynn RJ. Lipsitz LA. Rockwood K. Avorn J. Measuring frailty in Medicare data: Development and validation of a claims-based frailty index. Journals of Gerontology: Medical Sciences 2018;73(7):980-87.

Codes used for each component of the frailty score

| Codes used for each component of the fra<br>Condition | ICD9 Dx | ICD10 Dx | Coefficient |
|---|---|---|---|
| Intercept | | | 0.10288 |
| Intestinal infectious diseases | 001-009 | A00-A09 (exclude A02.1) | 0.00582 |
| Other and unspecified effects of external causes | 990-995 | A02.1, A22.7, A26.7, A32.7, A40, A41, A42.7, A45.8, B37.7, R65, T33, T34, T36-T50, T66-T78, T88 | 0.0085 |
| Other bacterial diseases | 030-041 | A30-A39; A42-A49 (exclude A32.7,A42.7,A45) | 0.01188 |
| Mycoses | 110-118 | B35-B49 (exclude B37.7) | 0.00831 |
| Malignant neoplasm of other and unspecified sites | 190-199 | C69-C80 | 0.00797 |
| Organic psychotic conditions | 290-294 | D01, D03, F02, F04, F05, F06, F10.159, F10.180, F10.181, F10.182, F10.188, F10.231, F10.239, F10.259, F10.27, F10.280, F10.281, F10.282, F10.288, F10.929, F10.950, F10.951, F10.959, F10.96, F10.980, F10.982, F10.99, F11.182, F11.282, F11.159, F11.181, F11.188, F11.222, F11.259, F11.281, F11.288, F11.922, F11.959, F11.981, F11.982, F11.988, F12.122, F12.159, F12.180, F12.188, F12.222, F12.259, F12.280, F12.288, F12.922, F12.959, F12.980, F12.988, F13.159, F13.180, F13.181, F13.182, F13.188, F13.259, F13.280, F13.281, F13.282, F13.288, F13.959, F13.980, F13.982, F13.988, F14.122, F14.159, F14.180, F14.181, F14.182, F14.188, F14.222, F14.259, F14.280, F14.281, F14.282, F14.288, F14.922, F14.959, F14.980, F14.981, F15.222, F15.259, F15.280, F15.281, F15.282, F15.288, F15.122, F15.188, F15.222, F15.259, F15.280, F15.281, F15.282, F15.288, F16.122, F16.159, F16.180, F16.183, F16.188, F16.259, F16.280, F16.283, F16.288, F16.959, F16.980, F16.983, F16.988, F16.988, F17.208, F17.218, F17.228, F17.298, F18.159, F18.180, F18.188, F18.259, F18.280, F18.288, F19.122, F19.159, F19.180, F19.181, F19.182, F19.188, F19.222, F19.259, F19.280, F19.281, F19.282, F19.991, F19.982, F19.999, F19.94, F19.950, F19.951, F19.96, F19.97, F19.99 | 0.04745 |
| Benign neoplasms | 210-229 | D10-D36 | -0.00513 |
| Neoplasms of uncertain behavior | 235-238 | D37-D48 | -0.00061 |
| Other and unspecified anemias | 285 | D62, D64 | 0.0085 |
| Purpura and other hemorrhagic conditions | 287 | D69 | -0.00804 |
| Diseases of white blood cells | 288 | D70, D71, D72, D76 | -0.0068 |
| Other metabolic and immunity disorders | 270-279 | D80-D84, D89, E65-E68, E70-E88, M10 (exclude E75.02, E75.19, E75.23, E75.25, E75.29, E75.4) | -0.00564 |
| Disorders of thyroid gland | 240-246 | E00-E07 | 0.00439 |
| Diseases of other endocrine glands | 250-259 | E08-E16,E20-E35 | 0.01078 |
| Hereditary and degenerative diseases of the central nervous system | 330-337 | E75.02, E75.19, E75.23, E75.25, E75.29, E75.4, F84.2, G10, G11, G12, G20, G21.0, G23, G24, G25, G30.9, G31, G80.3, G90, G91, G93.7, G93.89, G93.9, G94, G95, G99.2 | 0.01078 |

| Neurotic Disorders, Personality<br>Disorders, And Other Nonpsychotic<br>Mental Disorders | 300-316 | F07, F09, F32.9, F40-F44, F48, F54, F60, F64-F66, F68, F10-F19, F45.8, F45.9, F50, F51, F63.3, F80-F82, F88-F91, F93-F95, F98, R45.1, R48.0 (exclude F10.159, F10.180, F10.181, F10.182, F10.188, F10.231, F10.239, F10.259, F10.27, F10.280, F10.281, F10.282, F10.288, F10.929, F10.950, F10.951, F10.959, F10.96, F10.980, F10.982, F10.99, F11.182, F11.282, F11.159, F11.181, F11.188, F11.222, F11.259, F11.281, F11.288, F11.922, F11.959, F11.981, F11.982, F11.988, F12.122, F12.159, F12.180, F12.188, F12.222, F12.259, F12.280, F12.288, F12.922, F12.959, F12.980, F12.988, F13.159, F13.180, F13.181, F13.182, F13.188, F13.259, F13.280, F13.281, F13.282, F13.288, F13.959, F13.980, F13.982, F13.988, F14.122, F14.159, F14.180, F14.181, F14.182, F14.188, F14.222, F14.259, F14.280, F14.281, F14.282, F14.288, F14.922, F14.959, F14.981, F14.982, F14.988, F15.122, F15.159, F15.180, F15.181, F15.182, F15.188, F15.222, F15.259, F15.280, F15.281, F15.282, F15.288, F15.920, F15.922, F15.959, F15.980, F15.981, F15.982, F15.988, F16.122, F16.159, F16.180, F16.183, F16.188, F16.259, F16.280, F16.283, F16.288, F16.959, F16.80, F16.983, F16.988, F16.988, F17.208, F17.218, F17.228, F17.298, F18.159, F18.180, F18.188, F18.259, F18.280, F18.288, F18.289, F18.989, F18.988, F19.122, F19.159, F19.180, F19.181, F19.182, F19.188, F19.222, F19.259, F19.280, F19.281, F19.282, F19.991, F19.982, F19.939, F19.94, F19.950, F19.951, F19.96, | 0.01353 |
|---|---|---|---|
| Other psychoses | 295-299 | F20, F22-F25, F28-F34, F39, F44.89, F84 (exclude F84.2, F32.9) | 0.02112 |
| Other disorders of the central nervous system | 340-349 | G35, G37, G40, G43, G47.4, G80-G83, G92, G93.0-G93.2, G93.4-G93.6, G96-G97, G98.8 (exclusion G80.3 ) | 0.04031 |
| Disorders of the peripheral nervous system | 350-359 | G60-G65 | 0.00338 |
| Disorders of the eye and adnexa | 360-379 | H00-H59 (exclude H54.7) | -0.00061 |
| Hypertensive disease | 401-405 | 110-116 | 0.0174 |
| Ischemic heart disease | 410-414 | 120-125 | 0.0192 |
| Other forms of heart disease | 420-429 | 130-152 | 0.01989 |
| Cerebrovascular disease | 430-438 | 160-169 | -0.00046 |
| Diseases of arteries, arterioles, and capillaries | 440-448 | 170-179 | 0.00106 |
| Diseases of veins and lymphatics, and other diseases of circulatory system | 451-459 | 180-189;195-199 | 0.01234 |
| Pneumonia and influenza | 480-487 | J09-J18 | 0.01185 |
| Other diseases of the upper respiratory tract | 470-478 | J30-J39 | -0.0052 |
| Chronic obstructive pulmonary disease and allied conditions | 490-496 | J40-J45,J47,J67 | 0.01295 |
| Diseases of oral cavity, salivary glands, and jaws | 520-529 | K00-K14 | 0.00261 |
| Diseases of esophagus, stomach, and duodenum | 530-537 | K20-K31 | 0.0005 |
| Hernia of abdominal cavity | 550-553 | K40-K46 | 0.00388 |
| Infections of skin and subcutaneous tissue | 680-686 | L00-L08 | 0.00561 |
| Other inflammatory conditions | 690-698 | L10-L49, L51-L59 | -0.00053 |
| Arthropathies and related disorders | 710-719 | M00-M02, M04, M05-M09 M11-M14, M15-M19, M20-M25, M30-M36 (excluded M35.3) | 0.01408 |
| Rheumatism, excluding the back | 725-729 | M35.3, M60-M79,R25.2,R29.8x | 0.00021 |
| Dorsopathies | 720-724 | M40-M54 | 0.00984 |

| Osteopathies, chondropathies, and acquired musculoskeletal deformities | 730-739 | M80-M85, M86-M90, M91-M95, M99 | 0.00389 |
|---|---|---|---|
| Nephritis, nephrotic syndrome, and nephrosis | 580-589 | N00-N05, N08,N17,N18, N25, N26,N27 | 0.01047 |
| Other diseases of urinary system | 590-599 | N30-N39 | 0.01062 |
| Diseases of male genital organs | 600-608 | N40-N53 | -0.02131 |
| Congenital anomalies in urinary system | 753 | Q60-Q64 | -0.00836 |
| Congenital anomalies in musculoskeletal system | 754-756 | Q65-Q79 | 0.00073 |
| Symptoms | 780-789 | R00-R39, R50-R63 (exclude R09.1, R09.2,R13,R25.2,R29.8,R51, R52) | 0.00593 |
| III-defined and unknown causes of morbidity and mortality | 797-799 | R09.1, R09.2,R41.8x,R68.13,R68.82, R64,R69,R99 | 0.01119 |
| Nonspecific abnormal findings | 790-796 | R70-R97 | -0.00231 |
| Contusion with intact skin surface | 920-924 | \$00.93, \$10.93, \$00.10-\$00.12, \$05.10-\$05.12, \$05.90-\$05.92, \$20.00-\$20.02, \$20.20-\$20.22, \$30.0-\$30.3, T14.8-T14.9, \$40.01-\$40.02, \$50.0-\$50.1, \$60.0-\$60.2, \$70.0-\$70.1, \$80.0-\$80.1, \$90.0-\$90.3 | 0.01074 |
| Open wound of lower limb | 890-897 | \$81 | 0.02042 |
| Persons with a condition influencing their health status | V40-V49 | F48.9, F52.9, F69, F81.9, H54.7, H93.9x, J95.850, M96.0, R13.10, R43.9, R46.8x, R47.89, R68.89, Z48.22-Z48.298, Z66, Z73.82, Z74.0x, Z76.82, Z78.x, Z86.59, Z87.898, Z89.0x (excluding 789.52x), 790.x (excluding (Z90.41x. Z90.71x), 791.15, 791.83, 792.82, 793.x-795.x, 796.3x-Z96.9, 797.x-799.x (excluding 798.5x, 795.87x) | 0.00191 |
| Persons without reported diagnosis encountered during examination and investigation of individuals and populations | V70-V82 | Z00-Z13 | -0.01208 |
| Persons with potential health hazards related to communicable diseases | V01-V09 | Z20-Z29 | -0.00189 |
| Persons encountering health services for specific procedures and aftercare | V50-V59 | Z40-Z53, Z79 (exclude Z48.280, Z48.23, Z48.24, Z48.288, Z48.298 , Z48.22, Z48.290) | 0.00118 |

| Condition | CPT Code | Coefficient |
|---|---|---|
| Office/other outpatient visit – established patient | 99214 | 0.00149 |
| Hospital care – initial | 99222 | 0.0017 |
| Office consultation | 99242 | -0.00094 |
| Office consultation | 99245 | 0.00169 |
| Nursing facility care – subsequent | 99308 | 0.01389 |
| Preventive medicine services | 99381-99429 | -0.00712 |
| Anesthesia – head | 00100-00222 | -0.00049 |
| Anesthesia – neck | 00300-00352 | 0.00614 |
| Anesthesia – intrathoracic | 00500-00580 | -0.01568 |
| Anesthesia – lower abdomen | 00800-00882 | -0.01053 |
| Anesthesia – knee and popliteal area | 01320-01444 | -0.01215 |
| Surgery – respiratory system | 30000-32999 | -0.00129 |
| Surgery – female genital system | 56405-58999 | 0.00327 |
| Surgery – nervous system | 61000-64999 | 0.00843 |
| Radiology – nuclear medicine | 78000-79999 | -0.00301 |
| Therapeutic drug assays | 80150-80299 | 0.00789 |
| Cytopathology | 88104-88199 | -0.01082 |
| Surgical pathology | 88300-88399 | -0.00427 |

| Medicine – Ophthalmology | 92002-92499 | -0.00295 |
|----------------------------------------------------|-------------|----------|
| Medicine – Cardiovascular | 92950-93799 | -0.00046 |
| Medicine – Noninvasive vascular diagnostic studies | 93875-93990 | -0.00828 |
| Allergy and clinical immunology | 95004-95199 | -0.0084 |
| Physical medicine and rehabilitation | 97001-97799 | -0.00012 |
| Chiropractic manipulative treatment | 98940-98943 | -0.01426 |
| Special services, procedures and reports | 99000-99091 | 0.00127 |

| Condition | HCPCS Code | Coefficient |
|---|---|---|
| Transportation services including ambulance | A0021-A0999 | 0.01022 |
| Other supplies including diabetes supplies and contraceptives | A4244-A4290 | 0.0236 |
| Diabetic footwear | A5500-A5513 | 0.02375 |
| Breathing aids | A7000-A7046 | 0.00947 |
| Administrative, miscellaneous and experimental | A9150-A9999 | -0.00167 |
| Walking aids and attachments | E0100-E0159 | 0.02821 |
| Hospital beds and associated supplies | E0250-E0373 | 0.08649 |
| Oxygen delivery systems and related supplies | E0424-E0486 | 0.00665 |
| Humidifiers and nebulizers with related equipment | E0550-E0601 | 0.00385 |
| Wheelchair or transport chair and related accessories | E0950-E1298,<br>E2201-E2294,<br>E2300-E2399,<br>E2601-E2621 | 0.00805 |
| Accessories for oxygen delivery devices | E1353-E1406 | 0.02702 |
| Vaccine administration | G0008-G0010 | -0.00158 |
| Screening examinations and disease management training | G0101-G0124 | -0.01136 |
| Drugs, administered by injection | J0120-J7130 | 0.00664 |
| Inhalation solutions | J7608-J7684 | 0.00412 |
| Wheelchairs, components, and accessories | K0001-K0462,<br>K0669 | 0.07802 |

### Frailty markers

Osteoporosis

| OSCCOPOI OSIS | | | |
|---|---|---|---|
| ICD10 Dx | ICD9 Dx | LongDeslCD10 | LongDeslCD9 |
| M810 | 73300 | Age-related osteoporosis without current pathological | Osteoporosis, unspecified |
| | | fracture | |
| M810 | 73301 | Age-related osteoporosis without current pathological | Senile osteoporosis |
| | | fracture | |
| M818 | 73302 | Other osteoporosis without current pathological fracture | Idiopathic osteoporosis |
| M818 | 73303 | Other osteoporosis without current pathological fracture | Disuse osteoporosis |
| M816 | 73309 | Localized osteoporosis [Lequesne] | Other osteoporosis |
| M818 | 73309 | Other osteoporosis without current pathological fracture | Other osteoporosis |


| rachnoid, subdural, less than one hour] |
|---|
| rachnoid, subdural, less than one hour] rachnoid, subdural, less than one hour] rachnoid, subdural, less than one hour] rachnoid, subdural, less than one hour] |
| rachnoid, subdural, less than one hour] rachnoid, subdural, less than one hour] rachnoid, subdural, less than one hour] rachnoid, subdural, less than one hour] |
| rachnoid, subdural, less than one hour] rachnoid, subdural, less than one hour] rachnoid, subdural, less than one hour] rachnoid, subdural, less than one hour] |
| rachnoid, subdural, less than one hour] rachnoid, subdural, less than one hour] rachnoid, subdural, less than one hour] rachnoid, subdural, rachnoid, subdural, |
| rachnoid, subdural,<br>less than one hour]<br>rachnoid, subdural,<br>less than one hour]<br>rachnoid, subdural, |
| rachnoid, subdural,<br>less than one hour]<br>rachnoid, subdural,<br>less than one hour]<br>rachnoid, subdural, |
| rachnoid, subdural,<br>less than one hour]<br>rachnoid, subdural,<br>less than one hour] |
| rachnoid, subdural,<br>less than one hour] |
| rachnoid, subdural,<br>less than one hour] |
| rachnoid, subdural,<br>less than one hour]<br>rachnoid, subdural, |
| rachnoid, subdural, |
| rachnoid, subdural, |
| rachnoid, subdural, |
| less than one hour |
| rachnoid, subdural, |
| ate [1-24 hours] loss |
| rachnoid, subdural, |
| ged [more than 24 |
| o pre-existing |
| ) pre existing |
| rachnoid, subdural, |
| nged [more than 24 |
| o pre-existing |
| rachnoid, subdural, |
| nged [more than 24 |
| nged [more than 24<br>o pre-existing |
| nged [more than 24 to pre-existing rachnoid, subdural, |
| nged [more than 24<br>o pre-existing |
| nged [more than 24 to pre-existing rachnoid, subdural, |
| nged [more than 24<br>to pre-existing<br>rachnoid, subdural,<br>nged [more than 24 |
| nged [more than 24<br>to pre-existing<br>rachnoid, subdural,<br>nged [more than 24 |
| nged [more than 24<br>to pre-existing<br>rachnoid, subdural,<br>nged [more than 24<br>to pre-existing |
| nged [more than 24 to pre-existing rachnoid, subdural, nged [more than 24 to pre-existing rachnoid, subdural, rachnoid, subdural, |


| 8065 | Unspecified injury to L3 level of lumbar spinal cord, initial encounter | Open fracture of lumbar spine with spinal cord injury |
|---|---|---|
| 8065 | Unspecified injury to L4 level of lumbar spinal cord, initial encounter | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Unspecified injury to L5 level of lumbar spinal cord, initial encounter | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Unspecified injury to unspecified level of lumbar spinal cord, | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Complete lesion of L1 level of lumbar spinal cord, initial | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Complete lesion of L2 level of lumbar spinal cord, initial | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Complete lesion of L3 level of lumbar spinal cord, initial | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Complete lesion of L4 level of lumbar spinal cord, initial | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Complete lesion of L5 level of lumbar spinal cord, initial encounter | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Complete lesion of unspecified level of lumbar spinal cord, | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Incomplete lesion of L1 level of lumbar spinal cord, initial | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Incomplete lesion of L2 level of lumbar spinal cord, initial | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Incomplete lesion of L3 level of lumbar spinal cord, initial | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Incomplete lesion of L4 level of lumbar spinal cord, initial | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Incomplete lesion of L5 level of lumbar spinal cord, initial | Open fracture of lumbar spine with spinal cord injury |
| 8065 | Incomplete lesion of unspecified level of lumbar spinal cord, | Open fracture of lumbar spine with spinal cord injury |
| 80660 | Unspecified fracture of sacrum, initial encounter for closed fracture | Closed fracture of sacrum and coccyx with unspecified spinal cord injury |
| 80660 | Fracture of coccyx, initial encounter for closed fracture | Closed fracture of sacrum and coccyx with unspecified spinal cord injury |
| 80660 | Unspecified injury to sacral spinal cord, initial encounter | Closed fracture of sacrum and coccyx with unspecified spinal cord injury |
| 80661 | Unspecified fracture of sacrum, initial encounter for closed fracture | Closed fracture of sacrum and coccyx with complete cauda equina lesion |
| 80661 | Fracture of coccyx, initial encounter for closed fracture | Closed fracture of sacrum and coccyx with complete cauda equina lesion |
| 80661 | Injury of cauda equina, initial encounter | Closed fracture of sacrum and coccyx with complete cauda equina lesion |
| 80662 | Unspecified fracture of sacrum, initial encounter for closed fracture | Closed fracture of sacrum and coccyx with other cauda equina injury |
| 80662 | Fracture of coccyx, initial encounter for closed fracture | Closed fracture of sacrum and coccyx with other cauda equina injury |
| 80662 | Injury of cauda equina, initial encounter | Closed fracture of sacrum and coccyx with other cauda equina injury |
| 80669 | Unspecified fracture of sacrum, initial encounter for closed fracture | Closed fracture of sacrum and coccyx with other spinal cord injury |
| 80669 | Fracture of coccyx, initial encounter for closed fracture | Closed fracture of sacrum and coccyx with other spinal cord injury |
| 80669 | Complete lesion of sacral spinal cord, initial encounter | Closed fracture of sacrum and coccyx with other spinal cord injury |
| 80669 | Incomplete lesion of sacral spinal cord, initial encounter | Closed fracture of sacrum and coccyx with other spinal cord injury |
| 80670 | Unspecified fracture of sacrum, initial encounter for open | Open fracture of sacrum and coccyx with unspecified spinal |
| | fracture | cord injury |
| | 8065 | encounter 8065 Unspecified injury to L4 level of lumbar spinal cord, initial encounter 8065 Unspecified injury to unspecified level of lumbar spinal cord, initial encounter 8065 Complete lesion of L1 level of lumbar spinal cord, initial encounter 8065 Complete lesion of L2 level of lumbar spinal cord, initial encounter 8065 Complete lesion of L3 level of lumbar spinal cord, initial encounter 8065 Complete lesion of L4 level of lumbar spinal cord, initial encounter 8065 Complete lesion of L5 level of lumbar spinal cord, initial encounter 8065 Complete lesion of L5 level of lumbar spinal cord, initial encounter 8065 Complete lesion of L6 level of lumbar spinal cord, initial encounter 8065 Complete lesion of L7 level of lumbar spinal cord, initial encounter 8065 Incomplete lesion of L7 level of lumbar spinal cord, initial encounter 8065 Incomplete lesion of L8 level of lumbar spinal cord, initial encounter 8065 Incomplete lesion of L8 level of lumbar spinal cord, initial encounter 8065 Incomplete lesion of L9 level of lumbar spinal cord, initial encounter 8065 Incomplete lesion of L9 level of lumbar spinal cord, initial encounter 8065 Incomplete lesion of L9 level of lumbar spinal cord, initial encounter 8066 Incomplete lesion of L9 level of lumbar spinal cord, initial encounter 8066 Incomplete lesion of unspecified level of lumbar spinal cord, initial encounter 8066 Unspecified fracture of sacrum, initial encounter for closed fracture 80660 Unspecified fracture of sacrum, initial encounter for closed fracture 80661 Unspecified fracture of sacrum, initial encounter for closed fracture 80662 Injury of cauda equina, initial encounter 80663 Unspecified fracture of sacrum, initial encounter for closed fracture 80669 Unspecified fracture of sacrum, initial encounter for closed fracture 80669 Unspecified fracture of sacrum, initial encounter for closed fracture |


## Frailty markers


## Frailty markers


## Frailty markers


Falls


## Frailty markers


## Frailty markers


### Frailty markers

#### Combined Comorbidity Score for Claims Data

Gagne JJ, Glynn RJ, Avorn J, Levin R, Schneeweiss S. A combined comorbidity score predicted mortality in elderly patients better than existing scores. Journal of Clinical Epidemiology 2011:64(7):749-59.

Sun JW. Rogers JR. Her O. Welch EC. Panozzo CA. Toh S. Gagne JJ. Adaptation and Validation of the Combined Comorbidity Score for ICD-10-CM. Medical Care. 2017 Dec 1:55(12):1046-51.

Codes used for each ICD-10-CM and ICD-9-CM version of the combined comorbidity score


## Appendix A Frailty markers


BM, backward mapping; GEMs, General Equivalence Mappings; FBM, forward-backward mapping; ICD-9-CM, International Classification of Diseases, 9<sup>th</sup> Revision, Clinical Modification; ICD-10-CM, International Classification of Diseases, 10<sup>th</sup> Revision, Clinical Modification

### Comedications

#### Lithium

| NDC Generic Name | |
|-------------------|------------------------------|
| LITHIUM ASPARTATE | LITHIUM CITRATE |
| LITHIUM CARBONATE | LITHIUM CITRATE TETRAHYDRATE |

#### Anti-epileptic mood stabilizers

| NDC Generic Name | |
|-------------------|---------------------------------------------------|
| CARBAMAZEPINE | OXCARBAZEPINE |
| DIVALPROEX SODIUM | VALPROIC ACID |
| LAMOTRIGINE | VALPROIC ACID (AS SODIUM SALT) (VALPROATE SODIUM) |

#### Anti-epileptic non-mood stabilizers

| And epileptic non mood stabilizers | |
|------------------------------------|---------------|
| NDC Generic Name | |
| RUFINAMIDE | LACOSAMIDE |
| VIGABATRIN | ETHOSUXIMIDE |
| EZOGABINE | FELBAMATE |
| TIAGABINE HCL | LEVETIRACETAM |
| PHENYTOIN | TOPIRAMATE |
| ZONISAMIDE | PHENOBARBITAL |
| PRIMIDONE | GABAPENTIN |
| PREGABALIN | |

#### Atypical antipsychotics

| NDC Generic Name | |
|----------------------|---------------------|
| ZIPRASIDONE MESYLATE | ARIPIPRAZOLE |
| PALIPERIDONE | OLANZAPINE |
| ZIPRASIDONE HCL | RISPERIDONE |
| CLOZAPINE | QUETIAPINE FUMARATE |

#### Benzodiazepines

| 201120414120 | |
|-------------------------|----------------|
| NDC Generic Name | |
| ALPRAZOLAM | FLURAZEPAM HCL |
| CHLORDIAZEPOXIDE | LORAZEPAM |
| CLOBAZAM | MIDAZOLAM |
| CLONAZEPAM | OXAZEPAM |
| CLORAZEPATE DIPOTASSIUM | QUAZEPAM |
| DIAZEPAM | TEMAZEPAM |
| ESTAZOLAM | TRIAZOLAM |

#### Serotonin-norepinephrine reuptake inhibitor

| NDC Generic Name | |
|--------------------------|---------------------|
| DESVENLAFAXINE | DULOXETINE HCL |
| DESVENLAFAXINE FUMARATE | VENLAFAXINE HCL |
| DESVENLAFAXINE SUCCINATE | LEVOMILNACIPRAN HCL |

#### Selective serotonin reuptake inhibitor

| NDC Generic Name | |
|---------------------------|-----------------------------------------|
| PAROXETINE MESYLATE | CITALOPRAM HYDROBROMIDE |
| FLUOXETINE | FLUOXETINE HCL |
| OLANZAPINE/FLUOXETINE HCL | SERTRALINE HCL |
| FLUVOXAMINE MALEATE | FLUOXETINE HCL/DIETARY SUPPLEMENT NO.17 |
| ESCITALOPRAM OXALATE | FLUOXETINE HCL/DIETARY SUPPLEMENT NO.8 |
| PAROXETINE HCL | VILAZODONE HCL |

#### Tricyclic antidepressants

| NDC Generic Name | | |
|------------------------------------|--------------------------------|---|
| PROTRIPTYLINE HCL | DESIPRAMINE HCL | • |
| IMIPRAMINE PAMOATE | PERPHENAZINE/AMITRIPTYLINE HCL | |
| TRIMIPRAMINE MALEATE | NORTRIPTYLINE HCL | |
| AMITRIPTYLINE HCL/CHLORDIAZEPOXIDE | IMIPRAMINE HCL | |
| AMOXAPINE | DOXEPIN HCL | |
| CLOMIPRAMINE HCL | AMITRIPTYLINE HCL | • |

#### Typical antipsychotics

| NDC Generic Name | |
|------------------------|--------------------------------|
| FLUPHENAZINE ENANTHATE | THIOTHIXENE |
| LOXAPINE | FLUPHENAZINE HCL |
| PIMOZIDE | PERPHENAZINE/AMITRIPTYLINE HCL |

331

## Comedications

| MESORIDAZINE BESYLATE | TRIFLUOPERAZINE HCL |
|------------------------|---------------------|
| MOLINDONE HCL | CHLORPROMAZINE HCL |
| THIOTHIXENE HCL | HALOPERIDOL |
| FLUPHENAZINE DECANOATE | THIORIDAZINE HCL |
| PERPHENAZINE | |

## Anticoagulants

| NDC Generic Name | |
|---|---|
| APIXABAN | HEPARIN SODIUM, PORCINE IN 0.9 % SODIUM CHLORIDE |
| DABIGATRAN ETEXILATE MESYLATE | HEPARIN SODIUM, PORCINE IN 0.9 % SODIUM CHLORIDE/PF |
| DALTEPARIN SODIUM,PORCINE | HEPARIN SODIUM, PORCINE/DEXTROSE 5 % IN WATER |
| EDOXABAN TOSYLATE | HEPARIN SODIUM, PORCINE/DEXTROSE 5 % IN WATER/PF |
| ENOXAPARIN SODIUM | HEPARIN SODIUM, PORCINE/PF |
| FONDAPARINUX SODIUM | RIVAROXABAN |
| HEPARIN SODIUM,BEEF | TINZAPARIN SODIUM,PORCINE |
| HEPARIN SODIUM, PORCINE | WARFARIN SODIUM |
| HEPARIN SODIUM, PORCINE IN 0.45 % SODIUM CHLORIDE | |

#### Antiplatelet agents

| Antiplatelet agents | |
|---|---|
| NDC Generic Name | |
| ABCIXIMAB | CILOSTAZOL |
| ASPIRIN | CINNAMEDRINE HCL/ASPIRIN/CAFFEINE |
| ASPIRIN (CALCIUM CARB & MAGNESIUM BUFFERS)/PRAVASTATIN | CLOPIDOGREL BISULFATE |
| ASPIRIN/ACETAMINOPHEN | CODEINE PHOSPHATE/BUTALBITAL/ASPIRIN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/CAFFEINE | CODEINE PHOSPHATE/CARISOPRODOL/ASPIRIN |
| ASPIRIN/ACETAMINOPHEN/CAFFEINE/CALCIUM | CODEINE/ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/CAFFEINE/POTASSIUM | DIHYDROCODEINE BITARTRATE/ASPIRIN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/CALCIUM CARBONATE | DIHYDROCODEINE/ASPIRIN/CAFFEINE |
| ASPIRIN/ACETAMINOPHEN/MAGNESIUM/ALUMINUM HYDROXIDE/CAFFEIN | DIPYRIDAMOLE |
| ASPIRIN/CAFFEINE | EPHEDRINE/ASPIRIN/ACETANILIDE/CAFFEINE |
| ASPIRIN/CALCIUM CARBONATE | HYDROCODONE BITARTRATE/ASPIRIN |
| ASPIRIN/CALCIUM CARBONATE/MAGNESIUM | METHOCARBAMOL/ASPIRIN |
| ASPIRIN/CALCIUM CARBONATE/MAGNESIUM/ALUMINUM HYDROXIDE | ORPHENADRINE CITRATE/ASPIRIN/CAFFEINE |
| ASPIRIN/CODEINE PHOSPHATE | OXYCODONE HCL/ASPIRIN |
| ASPIRIN/DIPHENHYDRAMINE CITRATE | OXYCODONE HCL/OXYCODONE TEREPHTHALATE/ASPIRIN |
| ASPIRIN/DIPHENHYDRAMINE HCL | OXYCODONE/ASPIRIN |
| ASPIRIN/DIPHENHYDRAMINE/SODIUM BICARBONATE/CITRIC ACID | PENTAZOCINE HCL/ASPIRIN |
| ASPIRIN/DIPYRIDAMOLE | PHENYLEPHRINE HCL/ASPIRIN |
| ASPIRIN/MAGNESIUM CARBONATE/DIHYDROXYALUMINUM AMINOACETAT | PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN |
| ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE | PHENYLPROPANOLAMINE BITARTRATE/ASPIRIN/CHLORPHENIRAMINE |
| ASPIRIN/MAGNESIUM HYDROXIDE/ALUMINUM HYDROXIDE/CAFFEINE | PHENYLPROPANOLAMINE HCL/ASPIRIN |
| ASPIRIN/MEPROBAMATE | PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE |
| ASPIRIN/SALICYLAMIDE/ACETAMINOPHEN/CAFFEINE | PHENYLPROPANOLAMINE HCL/ASPIRIN/CHLORPHENIRAMINE/CAFFEINE |
| ASPIRIN/SALICYLAMIDE/CAFFEINE | PHENYLPROPANOLAMINE HCL/ASPIRIN/DIPHENHYDRAMINE |
| ASPIRIN/SODIUM BICARBONATE/CITRIC ACID | PRASUGREL HCL |
| BUTALBITAL/ASPIRIN/CAFFEINE | PROPOXYPHENE HCL/ASPIRIN/CAFFEINE |
| CARISOPRODOL/ASPIRIN | PSEUDOEPHEDRINE HCL/ASPIRIN/CHLORPHENIRAMINE |
| CHLORPHENIRAMINE MAL/PHENYLEPHRINE/D-METHORPHAN HB/ASPIRIN | TICAGRELOR |
| CHLORPHENIRAMINE MALEATE/PHENYLEPHRINE BITARTRATE/ASPIRIN | VORAPAXAR SULFATE |
| NDC Brand Name | |
| ARTHRITIS PAIN | BAYER ASPIRIN |
| ARTHRITIS PAIN FORMULA | BAYER ASPIRIN MAXIMUM |
| ARTHRITIS PAIN FORMULA A-F | ECOTRIN |
| ARTHRITIS PAIN RELIEF | ECOTRIN MAXIMUM STRENGTH |
| ARTHRITIS PAIN RELIEVER | MAPAP ARTHRITIS PAIN |
| BAYER ARTHRITIS PAIN REGIMEN | PLAVIX |

#### Nitrates

| NDC Generic Name | |
|---|---|
| ISOSORBIDE DINITRATE | NITROGLYCERIN |
| ISOSORBIDE DINITRATE/HYDRALAZINE HCL | NITROGLYCERIN/DEXTROSE 5 % IN WATER |
| ISOSORBIDE MONONITRATE | RANOLAZINE |
| NDC Brand Name | |
| ANG-O-SPAN | NITRO-TRANS SYSTEM |
| ANGINABID | NITRO-TRANSDERMAL |
| BIDIL | NITRO-TRANSDERMAL SYSTEM |
| CARDABID | NITROBART |
| DEPONIT | NITROCAP |

332

## Comedications

| DILATRATE-SR | NITROCINE |
|---------------------------|----------------------|
| IMDUR | NITROCOT |
| ISD | NITRODISC |
| ISMO | NITROGARD |
| ISO-BID | NITROGLYCERIN |
| ISO-D | NITROGLYCERIN IN D5W |
| ISOCHRON | NITROGLYCERIN PATCH |
| ISODITRATE | NITROGLYCERIN T/R |
| ISONATE | NITROGLYN |
| ISONATE TR | NITROGYLCERIN |
| ISOR-BID | NITROL |
| ISORDIL | NITROLINGUAL |
| ISORDIL TITRADOSE | NITROMED |
| ISOREX-10 | NITROMIST |
| ISOREX-2.5 | NITRONAL |
| ISOREX-5 | NITRONG |
| ISOSORBIDE DINITRATE | NITROQUICK |
| ISOSORBIDE MONONITRATE | NITROREX |
| ISOSORBIDE MONONITRATE ER | NITROSPAN |
| ISOTRATE | NITROSTAT |
| ISOTRATE ER | NITROSTAT IV |
| KENSORBIDE | NITROSTAT SR |
| LEMOTRATE | NITROTAB |
| MI-TRATES 2.5 | NITROTYM |
| MI-TRATES 6.5 | NTG |
| MINITRAN | NTS |
| MONOKET | ONSET-10 |
| N-G-C | ONSET-5 |
| N.T.S. | RANEXA |
| NITREK | RECTIV |
| NITRO | SORATE-2.5 |
| NITRO MAST TIMED RELEASE | SORATE-40 |
| NITRO S.A. | SORATE-5 |
| NITRO T.D. | SORBATE-10 |
| NITRO TRANSDERM | SORBATE-5 |
| NITRO TRANSDERMAL | SORBIDE |
| NITRO-BID | SORBITRATE |
| NITRO-BID IV | SORBITRATE SA |
| NITRO-CAPS TIME DOSE | TRANSDERM-NITRO |
| NITRO-DUR | TRATES |
| NITRO-PAR | TRIDIL |
| NITRO-TD-ACA | WF-NITRO |
| NITRO-TIME | |

Lipid lowering drugs

| IPRIC &ZN OX |
|--------------|
| NA /0.4 TS |
| *** (O * TS |
| 114 /OATS |
| NA/OATS |
| , |
| , |
| , |
| ALS |
| ACID |
| , |
| , |
| , |
| PROTEASE |
| RIDOXINE |
| B12/C/FA |
| T C/FA |
| / F |

### Comedications

| IRON FUMARATE & POLYSAC COMP/FOLIC ACID/VITAMIN C/NIACIN | THIAMINE/RIBOFLAVIN/NIACIN/CA PANTOTHENATE/VIT B6/B12/IRON |
|---|---|
| IRON FUMARATE & POLYSAC COMP/VITAMIN C/NIACIN | THIAMINE/RIBOFLAVIN/NIACIN/PANT ACID/B6/IRON/METHION/CHOLINE |
| IRON PYROPHOSPHATE/CYANOCOBALAMIN/FA/NIACIN/PYRIDOXINE HCL | VIT B2/NIACINAMIDE/PYRIDOXINE HCL/CYANOCOBALAMIN/D-PANTHENOL |
| LECITHIN/SITOSTEROLS/NIACIN/BETAINE/CHITOSAN | VIT C/PYRIDOXINE HCL/NIACIN/FA/VIT B12/HERBAL COMPLEX NO.192 |
| LOVASTATIN | VITAMIN B COMPLEX NO.12/NIACINAMIDE |
| LYSINE HCL/NIACINAMIDE/THIAMINE | VITAMIN B COMPLEX/NIACINAMIDE/PANTOTHENIC ACID/HERBAL DRUGS |
| MELATONIN/TRYPTOPHAN/VALERIAN/CHAMOMILE/NIACIN/INOSITOL/B6 | |

#### Non-insulin diabetes medications

| Non-insulin diabetes medications | |
|---|---|
| NDC Generic Name | |
| ACARBOSE | MIGLITOL |
| ACETOHEXAMIDE | NATEGLINIDE |
| ALOGLIPTIN BENZOATE | PIOGLITAZONE HCL |
| ALOGLIPTIN BENZOATE/METFORMIN HCL | PIOGLITAZONE HCL/GLIMEPIRIDE |
| ALOGLIPTIN BENZOATE/PIOGLITAZONE HCL | PIOGLITAZONE HCL/METFORMIN HCL |
| CANAGLIFLOZIN/METFORMIN HCL | REPAGLINIDE |
| CHLORPROPAMIDE | REPAGLINIDE/METFORMIN HCL |
| GLIMEPIRIDE | ROSIGLITAZONE MALEATE |
| GLIPIZIDE | ROSIGLITAZONE MALEATE/GLIMEPIRIDE |
| GLIPIZIDE/METFORMIN HCL | ROSIGLITAZONE MALEATE/METFORMIN HCL |
| GLYBURIDE | SAXAGLIPTIN HCL |
| GLYBURIDE/METFORMIN HCL | SAXAGLIPTIN HCL/METFORMIN HCL |
| LINAGLIPTIN | SITAGLIPTIN PHOSPHATE |
| LINAGLIPTIN/METFORMIN HCL | SITAGLIPTIN PHOSPHATE/METFORMIN HCL |
| METFORMIN HCL | SITAGLIPTIN PHOSPHATE/SIMVASTATIN |
| METFORMIN/AMINO ACIDS COMB. #7/HERBAL COMB.#125/CHOLINE | |
| | TOLAZAMIDE |
| METFORMIN/CAFFEINE/AMINO ACIDS#7/HERBAL COMB#125/CHOLINE BIT | TOLBUTAMIDE |
| NDC Brand Name | light TOLANA |
| ACARBOSE | ICN-TOLAM |
| ACETOHEXAMIDE | INSULASE |
| ACTOPLUS MET | INVOKAMET |
| ACTOPLUS MET XR | JANUMET |
| ACTOS | JANUMET XR |
| AMARYL | JANUVIA |
| APPFORMIN | JENTADUETO |
| APPFORMIN-D | JUVISYNC |
| AVANDAMET | KAZANO |
| AVANDARYL | KOMBIGLYZE XR |
| AVANDIA | METAGLIP |
| CHLORABETIC 250 | METFORMIN HCL |
| CHLORPROPAMIDE | METFORMIN HCL ER |
| DIABETA | MICRONASE |
| DIABINESE | NATEGLINIDE |
| DIBATROL | NESINA |
| DUETACT | ONGLYZA |
| DYMELOR | ORIBETIC |
| FORTAMET | ORINASE |
| GLIMEPIRIDE | |
| | OSENI<br>DIOCUTA ZONE LICI |
| GLIPIZIDE | PIOGLITAZONE HCL |
| GLIPIZIDE ER | PIOGLITAZONE-GLIMEPIRIDE |
| GLIPIZIDE XL | PIOGLITAZONE-METFORMIN |
| GLIPIZIDE-METFORMIN | PRANDIMET |
| GLUCAMIDE | PRANDIN |
| GLUCOPHAGE | PRECOSE |
| GLUCOPHAGE XR | REPAGLINIDE |
| GLUCOTROL | RIOMET |
| GLUCOTROL XL | RONASE |
| GLUCOVANCE | SK-TOLBUTAMIDE |
| GLUMETZA | STARLIX |
| GLYBURIDE | TOLAMIDE |
| GLYBURIDE MICRONIZED | TOLAZAMIDE |
| GLYBURIDE-METFORMIN HCL | TOLBUTAMIDE |
| GLYCRON | TOLINASE |
| GLYNASE | TRADJENTA |
| GLYSET | |
| GEIGET | |

Insulin HCPCS

## Comedications

| T | In |
|---|---|
| A4230 | \$5553 |
| A4231 | S5560 |
| A4232 | S5561 |
| A9274 | S5566 |
| E0784 | S5570 |
| J1815 | S5571 |
| J1817 | S8490 |
| S5550 | S9145 |
| \$5551 | S9353 |
| \$5552 | |
| NDC Generic Name | |
| INSULIN ASPART | INSULIN NPH HUMAN SEMI-SYN |
| INSULIN ASPART PROTAMINE HUMAN/INSULIN ASPART | INSULIN REG HUMAN SEMI-SYN |
| INSULIN DETEMIR | INSULIN ZINC BEEF |
| INSULIN GLULISINE | INSULIN ZINC EXTEND HUMAN REC |
| INSULIN LISPRO | INSULIN ZINC HUMAN REC |
| INSULIN LISPRO PROTAMINE & INSULIN LISPRO | INSULIN ZINC HUMAN SEMI-SYN |
| NDC Brand Name | |
| APIDRA | INSULIN LENTE PURIFIED PORK |
| APIDRA SOLOSTAR | INSULIN N PURIFIED PORK |
| EXUBERA COMBINATION PACK 12 | INSULIN NPH BEEF |
| EXUBERA COMBINATION PACK 15 | INSULIN NPH PURIFIED PORK |
| EXUBERA KIT | INSULIN R PORK PURIFIED |
| EXUBERA PATIENT PACK | INSULIN R PURIFIED PORK |
| HUMALOG | INSULIN REGULAR PORK |
| HUMALOG MIX 50-50 | INSULIN REGULAR PURIFIED PORK |
| | ISOPHANE INSULIN BEEF |
| HUMALOG MIX 50/50 | |
| HUMALOG MIX 75-25 | ISOPHANE PURIFIED BEEF INSULIN |
| HUMULIN 50-50 | LANTUS |
| HUMULIN 70-30 | LANTUS SOLOSTAR |
| HUMULIN 70/30 | LENTE INSULIN BEEF |
| HUMULIN 70/30 KWIKPEN | LEVEMIR |
| HUMULIN BR | LEVEMIR FLEXPEN |
| HUMULIN L | LEVEMIR FLEXTOUCH |
| HUMULIN N | MONOTARD HUMAN LENTE |
| HUMULIN N KWIKPEN | NOVOLIN 70-30 |
| HUMULIN R | NOVOLIN 70-30 INNOLET |
| HUMULIN U | NOVOLIN 70/30 |
| ILETIN I LENTE | NOVOLIN L |
| ILETIN I NPH | NOVOLIN N |
| ILETIN I REGULAR | NOVOLIN N INNOLET |
| ILETIN I SEMILENTE | NOVOLIN R |
| ILETIN I ULTRALENTE | NOVOLOG |
| ILETIN II LENTE(BEEF) | NOVOLOG FLEXPEN |
| ILETIN II LENTE(PORK) | NOVOLOG MIX 70-30 |
| ILETIN II NPH(BEEF) | NOVOLOG MIX 70-30 FLEXPEN |
| ILETIN II NPH(PORK) | PROTAMINE ZINC INSULIN BEEF |
| ILETIN II REGULAR(BEEF) | PURIFIED BEEF INSULIN ZINC |
| ILETIN II REGULAR(PORK) | PURIFIED PORK INSULIN |
| ILETIN II REGULAR(PORK)CONC | VELOSULIN HUMAN |
| INSULATARD HUMAN N | VELOSULIN HUMAN BR |
| INSULATARD N | VELOSULIN HUMAN R |
| INSULATARD NPH HUMAN | VELOSULIN R |
| INSULIN L PURIFIED PORK | ZINC |
| INSULIN LENTE BEEF | - |
| | <u> </u> |

#### Antidepressants

| , | |
|---|---|
| HCPCS | |
| J1320 | |
| NDC Generic Name | |
| AMITRIPTYLINE HCL | IMIPRAMINE HCL |
| AMITRIPTYLINE HCL/CHLORDIAZEPOXIDE | IMIPRAMINE PAMOATE |
| AMOXAPINE | ISOCARBOXAZID |
| BUPROPION HBR | LEVOMILNACIPRAN HYDROCHLORIDE |
| BUPROPION HCL | MAPROTILINE HCL |
| BUPROPION HCL/DIETARY SUPPLEMENT, MISC COMB15 | MIRTAZAPINE |
| BUPROPION HCL/DIETARY SUPPLEMENT, MISC COMB16 | NEFAZODONE HCL |
| CITALOPRAM HYDROBROMIDE | NORTRIPTYLINE HCL |

## Comedications

| | Tax |
|---|---|
| CLOMIPRAMINE HCL | OLANZAPINE/FLUOXETINE HCL |
| DESIPRAMINE HCL | PAROXETINE HCL |
| DESVENLAFAXINE | PAROXETINE MESYLATE |
| DESVENLAFAXINE FUMARATE | PERPHENAZINE/AMITRIPTYLINE HCL |
| DESVENLAFAXINE SUCCINATE | PHENELZINE SULFATE |
| DOXEPIN HCL | PROTRIPTYLINE HCL |
| DULOXETINE HCL | SERTRALINE HCL |
| ESCITALOPRAM OXALATE | TRAZODONE HCL |
| FLUOXETINE | TRAZODONE HCL/DIETARY SUPPLEMENT,MISC.COMBO8 |
| FLUOXETINE HCL | TRIMIPRAMINE MALEATE |
| FLUOXETINE HCL/DIETARY SUPPLEMENT,MISC COMB17 | VENLAFAXINE HCL |
| FLUOXETINE HCL/DIETARY SUPPLEMENT,MISC.COMBO8 | VILAZODONE HYDROCHLORIDE |
| FLUVOXAMINE MALEATE | VORTIOXETINE HYDROBROMIDE |
| NDC Brand Name | |
| ADAPIN | LIMBITROL DS |
| AMITID | LUDIOMIL |
| AMITRIPTYLINE HCL | LUVOX |
| AMITRIPTYLINE W/PERPHENAZINE | LUVOX CR |
| AMITRIPTYLINE-CHLORDIAZEPOXIDE | MAPROTILINE HCL |
| AMITRIPTYLINE-PERPHENAZINE | MARPLAN |
| AMITRIPTYLINE/CHLORDIAZEPOXIDE | MIRTAZAPINE |
| AMOXAPINE | MIRTAZAPINE ANHYDROUS |
| ANAFRANIL | NARDIL |
| APLENZIN | NEFAZODONE HCL |
| APPBUTAMONE | NORFRANIL |
| APPBUTAMONE-D | NORPRAMIN |
| ASENDIN | NORTRIPTYLINE HCL |
| AVENTYL HCL | OLANZAPINE-FLUOXETINE HCL |
| BRINTELLIX | OLEPTRO ER |
| BRISDELLE | PAMELOR |
| BUDEPRION SR | PAROXETINE HCL |
| BUDEPRION XL | PAXIL |
| BUPROBAN | PAXIL CR |
| BUPROPION HCL | PER-TRIP |
| BUPROPION HCL ER | PERPHENAZINE-AMITRIPTYLINE |
| BUPROPION HCL SR | PEXEVA |
| BUPROPION XL | PHENELZINE SULFATE |
| CELEXA | PRISTIQ ER |
| CHLORDIAZEPOXIDE-AMITRIPTYLINE | PROTRIPTYLINE HCL |
| CITALOPPAMALUP | PROZAC WEEKLY |
| CITALOPRAM HBR | PROZAC WEEKLY |
| CLOMIPRAMINE HCL | PRUDOXIN |
| CYMBALTA | Q.E.L |
| DECONIL | RAPIFLUX |
| DESIPRAMINE HCL | RE-LIVE |
| DESVENLAFAXINE ER | REMERON |
| DESVENLAFAXINE FUMARATE ER | SARAFEM |
| DESYREL | SELFEMRA |
| DOXEPIN HCL | SENTROXATINE |
| DULOXETINE HCL | SERTRALINE HCL |
| E-VILL 10 | SERZONE |
| E-VILL 100 | SILENOR |
| E-VILL 25 | SINEQUAN |
| E-VILL 50 | SK-AMITRIPTYLINE |
| E-VILL 75 | SK-PRAMINE |
| EFFEXOR | STABANIL |
| EFFEXOR XR | SURMONTIL |
| ELAVIL | SYMBYAX |
| EMITRIP | TOFRANIL |
| ENDEP | TOFRANIL-PM |
| ENOVIL | TRAZAMINE |
| ESCITALOPRAM OXALATE | TRAZODONE HCL |
| ETNOFRIL | TRIAVIL 10-2 |
| ETRAFON 2-10 | TRIAVIL 2-10 |
| ETRAFON 2-25 | TRIAVIL 2-25 |
| ETRAFON A 4-10 | TRIAVIL 25-2 |
| ETRAFON FORTE 4-25 | TRIAVIL 25-4 |
| FETZIMA | TRIAVIL 4-10 |
| | • |

## Comedications

| FLUOXETINE DR | TRIAVIL 4-25 |
|------------------------|----------------------|
| FLUOXETINE HCL | TRIAVIL 4-50 |
| FLUVOXAMINE MALEATE | TRIMIPRAMINE MALEATE |
| FLUVOXAMINE MALEATE ER | VANATRIP |
| FORFIVO XL | VENLAFAXINE HCL |
| GABOXETINE | VENLAFAXINE HCL ER |
| IMAVATE | VIIBRYD |
| IMIPRAMINE HCL | VIVACTIL |
| IMIPRAMINE PAMOATE | WELLBUTRIN |
| JANIMINE | WELLBUTRIN SR |
| KENVIL | WELLBUTRIN XL |
| KHEDEZLA | ZOLOFT |
| LEXAPRO | ZONALON |
| LIMBITROL | ZYBAN |

### SAMA/SABA

| NDC Generic Name | |
|---------------------------------------|---------------------|
| LEVALBUTEROL TARTRATE | LEVALBUTEROL HCL |
| IPRATROPIUM BROMIDE/ALBUTEROL SULFATE | IPRATROPIUM BROMIDE |
| ALBUTEROL | ALBUTEROL SULFATE |
| TERBUTALINE SULFATE | |

#### LAMA/LABA

| NDC Generic Name | |
|---|---|
| INDACATEROL MALEATE/GLYCOPYRROLATE | GLYCOPYRROLATE/FORMOTEROL FUMARATE |
| TIOTROPIUM BROMIDE/OLODATEROL HCL | UMECLIDINIUM BROMIDE/VILANTEROL TRIFENATATE |

#### Inhaled corticosteroids

| illiarea coi treoster olas | |
|----------------------------|----------------|
| NDC Generic Name | |
| BUDESONIDE, MICRONIZED | BUDESONIDE |
| NDC Brand Name | |
| FLOVENT ROTADISK | PULMICORT |
| ARMONAIR RESPICLICK | FLOVENT DISKUS |
| ASMANEX HFA | QVAR |
| PULMICORT FLEXHALER | ASMANEX |
| AEROSPAN | ALVESCO |
| ARNUITY ELLIPTA | FLOVENT |
| QVAR REDIHALER | FLOVENT HFA |

#### **DMARDs**


## Comedications

| FOLEX PFS | CYCLOPHOSPHAMIDE MONOHYDRATE |
|--------------------------------|------------------------------|
| FOLEX-PFS | NEOSAR |
| RHEUMATREX | NEOSAR FOR INJECTION |
| TREXALL | CYTOXAN LYOPHILIZED |
| METHOTREXATE SODIUM PARENTERAL | CYTOXAN |
| OTREXUP | CYCLOPHOSPHAMIDE |
| METHOTREXATE LPF | SANGCYA |
| RASUVO | NEORAL |
| METHOTREXATE SODIUM | GENGRAF |
| METHOTREXATE | RESTASIS |
| QUINEPROX | SANDIMMUNE |
| PLAQUENIL | CYCLOSPORINE MODIFIED |
| HYDROXYCHLOROQUINE SULFATE | CYCLOSPORINE |
| S.A.S500 | AUROLATE |
| SULFA DYNE | GOLD SODIUM THIOMALATE |
| SULFASALAZINE DR | MYOCHRYSINE |
| SULFAZINE | HUMIRA |
| AZULFIDINE | CIMZIA |
| SULFASALAZINE | ENBREL |
| ARAVA | SIMPONI ARIA |
| LEFLUNOMIDE | SIMPONI |
| XELJANZ XR | REMICADE |
| XELIANZ | ORENCIA |
| RIDAURA | ACTEMRA |
| AZASAN | KINERET |

#### Calcium channel blockers

| Calcium channel blockers | |
|-----------------------------------------------|------------------------|
| NDC Brand Name | |
| ADALAT | ISOPTIN |
| ADALAT CC | ISOPTIN SR |
| AFEDITAB CR | ISRADIPINE |
| AMLODIPINE BESILATE | LEXXEL |
| AMLODIPINE BESYLATE | LOTREL |
| AMLODIPINE BESYLATE-BENAZEPRIL | MATZIM LA |
| AMLODIPINE-ATORVASTATIN | NICARDIPINE HCL |
| AMLODIPINE-VALSARTAN | NICARDIPINE HCL-D5W |
| AMTURNIDE | NIFEDIAC CC |
| AZOR | NIFEDICAL XL |
| CADUET | NIFEDIPINE |
| CALAN | NIFEDIPINE ER |
| CALAN SR | NIFEDIPINE XL |
| CARDENE | NIMODIPINE |
| CARDENE I.V. | NIMOTOP |
| CARDENE SR | NISOLDIPINE |
| CARDIZEM | NORVASC |
| CARDIZEM CD | NYMALIZE |
| CARDIZEM LA | PLENDIL |
| CARDIZEM SR | POSICOR |
| CARTIA XT | PROCARDIA |
| CLEVIPREX | PROCARDIA XL |
| COVERA-HS | SULAR |
| DILACOR XR | TARKA |
| DILT-CD | TAZTIA XT |
| DILT-XR | TEKAMLO |
| DILTIA XT | TELMISARTAN-AMLODIPINE |
| DILTIAZEM 24HR CD | TIAMATE |
| DILTIAZEM 24HR ER | TIAZAC |
| DILTIAZEM ER | TRANDOLAPRIL-VERAPAMIL |
| DILTIAZEM HCL | TRIBENZOR |
| DILTIAZEM HCL-NS | TWYNSTA |
| DILTIAZEM XR | VASCOR |
| DILTIAZEM-D5W | VERAPAMIL ER |
| DILTZAC ER | VERAPAMIL ER PM |
| DYNACIRC | VERAPAMIL HCL |
| DYNACIRC CR | VERAPAMIL SR |
| EXFORGE | VERELAN |
| EXFORGE HCT | VERELAN PM |
| FELODIPINE ER | |
| NDC Generic Name | · |
| ALISKIREN HEMIFUMARATE/AMLODIPINE<br>BESYLATE | DILTIAZEM MALATE |

## Other PAH treatments and PAH severity indicators

| NDC Generic Name | |
|---|---|
| ALISKIREN HEMIFUMARATE/AMLODIPINE/HYDROCHLORO THIAZIDE | ENALAPRIL MALEATE/FELODIPINE |
| AMLODIPINE BESYLATE | FELODIPINE |
| AMLODIPINE BESYLATE/ATORVASTATIN CALCIUM | ISRADIPINE |
| AMLODIPINE BESYLATE/BENAZEPRIL HCL | MIBEFRADIL DI-HCL |
| AMLODIPINE BESYLATE/OLMESARTAN MEDOXOMIL | NICARDIPINE HCL |
| AMLODIPINE BESYLATE/VALSARTAN | NIFEDIPINE |
| AMLODIPINE<br>BESYLATE/VALSARTAN/HYDROCHLOROTHIAZI | NIMODIPINE |
| BEPRIDIL HCL | NISOLDIPINE |
| CLEVIDIPINE BUTYRATE | OLMESARTAN MEDOXOMIL/AMLODIPINE BESYLATE/HYDROCHLOROTHIAZIDE |
| DILTIAZEM HCL | TELMISARTAN/AMLODIPINE BESYLATE |
| DILTIAZEM HCL IN 0.9 % SODIUM CHLORIDE | TRANDOLAPRIL/VERAPAMIL HCL |
| DILTIAZEM HCL/DEXTROSE 5 % IN WATER | VERAPAMIL HCL |

#### Riociguat

| NDC Brand Name |
|------------------|
| ADEMPAS |
| NDC Generic Name |
| RIOCIGUAT |

#### Prostanoids

| ICPCS Procedure Code | |
|---|---|
| J1325 | Q4074 |
| J3285 | |
| NDC Generic Name | |
| TREPROSTINIL | TREPROSTINIL DIOLAMINE |
| DILUENT FOR EPOPROSTENOL SODIUM<br>(GLYCINE) | TREPROSTINIL SODIUM |
| EPOPROSTENOL SODIUM (ARGININE) | TREPROSTINIL/NEBULIZER ACCESSORIES |
| EPOPROSTENOL SODIUM (GLYCINE) | TREPROSTINIL/NEBULIZER AND ACCESSORIES |
| ILOPROST TROMETHAMINE | |

### Number of hospitalization with PAH as the primary discharge diagnosis


Other PAH treatments and PAH severity indicators


### Atrial Fibrillation


## Comorbid conditions


**Heart Failure** 


|--|


| ICD10 Dx | ICD9 Dx | LongDeslCD10 | LongDeslCD9 |
|---|---|---|---|
| G450 | 435 | Vertebro-basilar artery syndrome | TRANSIENT CEREBRAL ISCHEMIA |
| G451 | 4350 | Carotid artery syndrome (hemispheric) | BASILAR ARTERY SYNDROME |
| G452 | 4351 | Multiple and bilateral precerebral artery syndromes | VERTEBRAL ARTERY SYNDROME |
| G458 | 4352 | Other transient cerebral ischemic attacks and related | SUBCLAVIAN STEAL SYNDROME |
| | | syndromes | |
| G459 | 4353 | Transient cerebral ischemic attack, unspecified | VERTEBROBASILAR ARTERY SYNDROME |
| G460 | 4358 | Middle cerebral artery syndrome | OTHER SPECIFIED TRANSIENT CEREBRAL ISCHEMIAS |
| G461 | 4359 | Anterior cerebral artery syndrome | UNSPECIFIED TRANSIENT CEREBRAL ISCHEMIA |
| G462 | | Posterior cerebral artery syndrome | |
| 167841 | | Reversible cerebrovascular vasoconstriction syndrome | |
| 167848 | | Other cerebrovascular vasospasm and vasoconstriction | |


| intraluminal Devices, Percutaneous Approach-eluting intraluminal Devices, Percutaneous Approach Diatron of left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach— Diatron of left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach— Diatron of left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach— Diatron of left Thyroid Artery, Siffication, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach— Diatron of left Thyroid Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach— Diatron of left Thyroid Artery with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach— Diatron of left Thyroid Artery, Siffication, with Intraluminal Devices, Percutaneous Approach— Diatron of left Thyroid Artery, Siffication, with Intraluminal Devices, Percutaneous Approach— Diatron of left Thyroid Artery, Siffication, with Intraluminal Devices, Percutaneous Approach— Diatron of left Thyroid Artery, Siffication, with Two Intraluminal Devices, Percutaneous Approach— Diatron of left Thyroid Artery, Siffication, with Two Intraluminal Devices, Percutaneous Approach— Diatron of left Thyroid Artery, Siffication, with Two Intraluminal Devices, Percutaneous Approach— Diatron of left Thyroid Artery, Siffication, with Two Intraluminal Devices, Percutaneous Approach— Diatron of left Thyroid Artery, Siffication, with Tree Intraluminal Devices, Percutaneous Approach— Diatron of left Thyroid Artery, Siffication, with Tree Intraluminal Devices, Percutaneous Approach— Diatron of left Thyroid Artery, Siffication, with Tree Intraluminal Devices, Percutaneous Approach— Diatron of left Thyroid Artery, Siffication, with Prog-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Diatron of left Thyroid Artery, Siffication, with Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Diatron of left Thyroid Artery, Siffication, with Tree Diatron of left Thyroid Artery, Sifficati | Comorbia com | | _ |
|---|---|---|---|
| intraluminal Devices, Percutaneous Approach Direjecting Intraluminal Devices, Percutaneous Approach eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach-eluting Approach eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Four or Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Four or Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Four or Intralumi | | Dilation of Left Thyroid Artery with Two Drug-eluting | |
| Orugeluting intraluminal Devices, Percutaneous Approach Approach Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery, Rifurcation, with Four or More Drug-eluting intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery, Rifurcation, with Four or More Drug-eluting intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery, Rifurcation, with Four or More Drug-eluting intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery with Four or More Drug- eluting intraluminal Devices, Percutaneous Approach- eluting intraluminal Devices, Percutaneous Approach- eluting intraluminal Devices, Percutaneous Approach- eluting intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Rifurcation, with Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Rifurcation, with Two Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Rifurcation, with Tree Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Rifurcation, with Three Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Rifurcation, with Tree Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Rifurcation, with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Rifurcation, with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Rifurcation, with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Rifurcation, Percutaneous Approach- Dilation of Left Thyroid Artery, Rifurcation, Percutaneous Approach- Dilation of Left Thyroid Artery, Rifurcation, Percutaneous Approach- Dilation of Left Thyroid Artery, Rifurcation, Dilation of Left Thyroid Artery, Rifurcation, Dilation of Left Thyroid Artery, Rifurcation, Dilation of Left Thyroid Artery, Rifurcation, with Troe Ung-eluting Intralumin | | | |
| Approach Dilation of Left Thyroid Artery with Three Drug-eluting intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery, with Three Drug-eluting intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery, Bifurcation, with Four or More Drug-eluting intraluminal Devices, Percutaneous Approach—Dilation of Left Thyroid Artery, With Four or More Drug-eluting intraluminal Devices, Percutaneous Approach—Dilation of Left Thyroid Artery with Four or More Drug-eluting intraluminal Devices, Percutaneous Approach—Dilation of Left Thyroid Artery, Bifurcation, with Intraluminal Devices, Percutaneous Approach—Dilation of Left Thyroid Artery, Bifurcation, with Intraluminal Devices, Percutaneous Approach—Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach—Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach—Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach—Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach—Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach—Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach—Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach—Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach—Dilation of Left Thyroid Artery, Bifurcation, with Drug-eluting Intraluminal Devices, Percutaneous Approach—Dilation of Left Thyroid Artery, Bifurcation, with Drug-eluting Intraluminal Devices, Percutaneous Approach—Dilation of Left Thyroid Artery, Bifurcation, with Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—Ulting Intraluminal Devices, Percutaneous Endoscopic Approach—Ulting Intraluminal Devices, Percutaneous Endoscopic Approach—Ulting Intraluminal Devices, Percut | 037V35Z | Intraluminal Devices, Percutaneous Approach | |
| Dilation of Left Thyroid Artery, with Three Drug-eluting intraluminal Devices, Percutaneous Approach-eluting intraluminal Devices, Percutaneous Endoscopic Approach-eluting | | Drug-eluting Intraluminal Devices, Percutaneous | |
| Dilation of Left Thyroid Artery with Three Drug-eluting intraluminal Devices, Percutaneous Approacheluting intraluminal Devices, Percutaneous Approacheluting intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approacheluting Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intraluminal Devices, Percuta | | Approach-eluting Intraluminal Devices, Percutaneous | |
| intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery, Bifurcation, with Four or More Drug-eluting intraluminal Devices, Percutaneous Approach-butting intraluminal Devices, Percutaneous Approach-butting intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery, with Four or More Drug- eluting intraluminal Devices, Percutaneous Approach- eluting intraluminal Devices, Percutaneous Approach- eluting intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, Dilation of Left Th | 037V366 | Approach | |
| Intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approacheluting Intraluminal Device, Percutaneous Approacheluting Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intraluminal Device | | Dilation of Left Thyroid Artery with Three Drug-eluting | |
| Dilation of Left Thyroid Artery, Bifurcation, with Four or More Drug-eluting Intraluminal Devices, Percutaneous Approach-eluting Intraluminal Device, Percutaneous Approach-eluting Intraluminal Device, Percutaneous Approach-Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Device, Percutaneous Approach-Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Device, Percutaneous Approach-Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach-Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach-Dilation of Left Thyroid Artery, Bifurcation, with Four Office Percutaneous Approach-Dilation of Left Thyroid Artery, Bifurcation, with Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-Unity Intraluminal Devices, Percutaneous Endoscopic Approach-Eluting Intraluminal Devices, Percutaneous Endoscopic Approach-Eluting Intraluminal Devices, Percutaneous Endoscopic Approach-Eluting Intraluminal Devices, Percutaneous Endoscopic Approach-Eluting Intraluminal Devices, Percutaneous Endoscopic Approach-Eluting Intraluminal Devices, Percutaneous Endoscopic A | | Intraluminal Devices, Percutaneous Approach-eluting | |
| More Drug-eluting intraluminal Devices, Percutaneous Approach eluting intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery with Four or More Drug- eluting intraluminal Devices, Percutaneous Approach- eluting intraluminal Devices, Percutaneous Approach- eluting intraluminal Devices, Percutaneous Approach- eluting intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with intraluminal Device, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Tree intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Four or intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, Dilation of Left Thyroid | 037V36Z | Intraluminal Devices, Percutaneous Approach | |
| Approach-eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery with Four or More Drug- eluting Intraluminal Devices, Percutaneous Approach- eluting Intraluminal Devices, Percutaneous Approach- eluting Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with intraluminal Device, Percutaneous Approach- Dilation of Left Thyroid Artery with Intraluminal Device, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Tree intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Tree intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach- Dilation of Left Thyroid Artery, Percutaneous Approach- Dilation of Left Thyroid Artery, Percutaneous Approach- Dilation of Left Thyroid Artery, Percutaneous Approach- Dilation of Left Thyroid Artery, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approa | | Dilation of Left Thyroid Artery, Bifurcation, with Four or | |
| Dilation of Left Thyroid Artery, with Four or More Drug- eluting intraluminal Devices, Percutaneous Approach- eluting intraluminal Devices, Percutaneous Approach- eluting intraluminal Devices, Percutaneous Approach- eluting intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with intraluminal Device, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Three intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Four or More intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, with Two Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Four or More intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Four or More intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Percutaneous Approach- Dilation of Left Thyroid Artery, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach- Dilation of Left Thyroid Artery, Percutaneous Approach- Dilation of Left Thyroid Artery, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, With Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, With Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, With Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, With Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneou | | More Drug-eluting Intraluminal Devices, Percutaneous | |
| Dilation of Left Thyroid Artery with Four or More Drug- eluting Intraluminal Devices, Percutaneous Approach- eluting Intraluminal Devices, Percutaneous Supproach Dilation of Left Thyroid Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Two Dilation of Left Thyroid Artery, Bifurcation, with Two Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intra | | Approach-eluting Intraluminal Devices, Percutaneous | |
| Dilation of Left Thyroid Artery, with Four or More Drug- eluting Intraluminal Devices, Percutaneous Approach- eluting Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Dilation of Left Thyroid Artery, Bifurcation, with Two Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Thyroid Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approac | 037V376 | Approach | |
| eluting Intraluminal Devices, Percutaneous Approach eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Device, Percutaneous Approach Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, With Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, With Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, With Three Drug-eluting Intralumi | | Dilation of Left Thyroid Artery with Four or More Drug- | |
| eluting Intraluminal Devices, Percutaneous Approach Dilation of Left Thyroid Artery, Bifurcation, with Intralumianal Device, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Two Intralumianal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Two Intralumianal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Three Intralumianal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Three Intralumianal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Three Intralumianal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intralumianal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intralumianal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Dilation of Left Thyroid Artery, Bifurcation, Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Drug- eluting Intralumianal Devices, Percutaneous Endoscopic Approach-eluting Intralumianal Device, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, With Drug-eluting Intralumianal Device, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery with Drug-eluting Intralumianal Device, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery with Drug-eluting Intralumianal Device, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery with Prop- eluting Intralumianal Device, Percutaneous Endoscopic Approach- eluting Intralumianal Device, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intralumianal Devices, Percutaneous Endoscopic Approach- Dilation of Left Thyroid | | | |
| Dilation of Left Thyroid Artery, Bifurcation, with intraluminal Device, Percutaneous Approach— Dilation of Left Thyroid Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Two intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Two intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Three intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Three intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Drug-eluting Intraluminal Device, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal De | 037V377 | | |
| Intraluminal Device, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Device, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, With Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery, Bifurcation, With Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery, With Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery, With Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery, With Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery with Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery with Thre | 0077072 | | |
| Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Percutaneous Endoscopic Approach- eluting Intral | 037V3D6 | | |
| Dilation of Left Thyroid Artery, Bifurcation, with Two Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Three Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery, With Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneo | 037 4 3 5 0 | | |
| Dilation of Left Thyroid Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Dilation of Left Thyroid Artery, Bifurcation, Dilation of Left Thyroid Artery, Bifurcation, Dilation of Left Thyroid Artery, Bifurcation, Dilation of Left Thyroid Artery, Bifurcation, Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intralum | 027//207 | · | |
| Intraluminal Devices, Percutaneous Approach— | 03/ V 3DL | · | |
| Dilation of Left Thyroid Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, With Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous End | 0271/256 | | |
| Devices, Percutaneous Approach Dilation of Left Thyroid Artery, Bifurcation, with Three intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach—Endoscopic Approach— Dilation of Left Thyroid Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach—Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—Luting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—Luting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach—Luting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery | 037V3E6 | • | |
| Dilation of Left Thyroid Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, With Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery, Bifurcation, with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— United Intraluminal Device, Percutaneous Endoscopic Approach— Endoscopic Approach— Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery, With Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endoscopic Approach— eluting Intraluminal Devices, Percutaneous Endosc | | , , | |
| Intraluminal Devices, Percutaneous Approach- | 037V3EZ | | |
| Dilation of Left Thyroid Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Pe | | * | |
| Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery, Bifurcation, with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intra | 037V3F6 | | |
| Dilation of Left Thyroid Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Dilation of Left Thyroid Artery, Bifurcation, Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery, Bifurcation, with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Thyroid Artery, Bifurcation, with Two Drugeluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous | | · | |
| More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Dilation of Left Thyroid Artery, Bifurcation, Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach—luting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach—eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic | 037V3FZ | Devices, Percutaneous Approach | |
| Dilation of Left Thyroid Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach eluting Intraluminal Devices, Percutaneous Endoscopic Approach eluting Intraluminal Devices, Percutaneous Endoscopic Approach | | Dilation of Left Thyroid Artery, Bifurcation, with Four or | |
| Intraluminal Devices, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach—eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneo | 037V3G6 | More Intraluminal Devices, Percutaneous Approach | |
| Dilation of Left Thyroid Artery, Bifurcation, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percuta | | Dilation of Left Thyroid Artery with Four or More | |
| Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic | 037V3GZ | Intraluminal Devices, Percutaneous Approach | |
| Dilation of Left Thyroid Artery, Percutaneous Approach— Dilation of Left Thyroid Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic | | Dilation of Left Thyroid Artery, Bifurcation, | |
| Dilation of Left Thyroid Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic | 037V3Z6 | Percutaneous Approach- | |
| Dilation of Left Thyroid Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic | 037V3ZZ | Dilation of Left Thyroid Artery, Percutaneous Approach- | |
| eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic | | 1 | |
| Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic | | | |
| Dilation of Left Thyroid Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic | | _ · | |
| Dilation of Left Thyroid Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic | 037V446 | 1 | |
| Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic | 037 7 1 10 | | |
| eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic eluting Intraluminal Devices, Percutaneous Endoscopic | | | |
| Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic | | | |
| Dilation of Left Thyroid Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Bilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Bilation Intraluminal Devices, Percutaneous Endoscopic | 027\/447 | | |
| Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Bilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Bilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic | 037 V 442 | | |
| Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic | | | |
| Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intraluminal Devices, Percutaneous Endoscopic | | | |
| Dilation of Left Thyroid Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intraluminal Devices, Percutaneous Endoscopic | 027)/456 | - | |
| Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- eluting Intraluminal Devices, Percutaneous Endoscopic | U3/V430 | 1 11 | <u> </u> |
| eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic | | | |
| Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic | | · | ] |
| Dilation of Left Thyroid Artery, Bifurcation, with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic | 0271/457 | | |
| Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic | U3/V45Z | | |
| Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic | [ | | |
| Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intraluminal Devices, Percutaneous Endoscopic | | | |
| Dilation of Left Thyroid Artery with Three Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intraluminal Devices, Percutaneous Endoscopic | | - | |
| Intraluminal Devices, Percutaneous Endoscopic Approacheluting Intraluminal Devices, Percutaneous Endoscopic | 037V466 | 1 11 | |
| eluting Intraluminal Devices, Percutaneous Endoscopic | | | |
| | | | 1 |
| O37V46Z Approach | | · · | |
| | 037V46Z | Approach | |


| · |
|---------------------------------------|


| Dilation of Left Peroneal Artery with Four or More Drug eluting Intraluminal Devices, Percutaneous Approach- eluting Intraluminal Devices, Percutaneous Approach- outly Dilation of Left Peroneal Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach- Dilation of Left Peroneal Artery with Intraluminal Device, Percutaneous Approach- Dilation of Left Peroneal Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach- Dilation of Left Peroneal Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach- Dilation of Left Peroneal Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach- Dilation of Left Peroneal Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach- Dilation of Left Peroneal Artery with Three Intraluminal Devices, Percutaneous Approach- Dilation of Left Peroneal Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Peroneal Artery with Four or More Intraluminal Devices, Percutaneous Approach- Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach- Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach- Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach- Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach- Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Peroneal Artery with Two Drug-elu |
|---|
| Deluting Intraluminal Devices, Percutaneous Approach |
| Dilation of Left Peroneal Artery, Bifurcation, with Intraluminal Device, Percutaneous Approach— Dilation of Left Peroneal Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, With Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, Bifurcation, with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Drugeluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery with Two Drugeluting Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Intraluminal Device, Percutaneous Approach- Dilation of Left Peroneal Artery with Intraluminal |
| Dilation of Left Peroneal Artery with Intraluminal Device, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, With Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach—Butting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach—Butting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach—Butting Intraluminal Devices, Percutaneous Endoscopic Approach—Butting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, With Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, With Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, With Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Device, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, With Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, With Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, With Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Drugeluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, Bifurcation, With Two Drugeluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, With Two Drugeluting Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Dilation of Left Peroneal Artery, Bifurcation, with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Drugeluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Drugeluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Drugeluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery with Two Drugeluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery with Two Drugeluting Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Intraluminal Devices, Percutaneous Approach— |
| Dilation of Left Peroneal Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach |
| Dilation of Left Peroneal Artery with Two Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscop |
| Dilation of Left Peroneal Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Dilation of Left Peroneal Artery, Bifurcation, with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, With Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Drugeluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Drugeluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, With Two Drugeluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery with Two Drugeluting Intraluminal Devices, Percutaneous Endoscopic Approach— |
| 047U3F6 Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Dilation of Left Peroneal Artery with Three Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, Bifurcation, with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Drugeluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery, Bifurcation, with Two Drugeluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery with Two Drugeluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery with Two Drugeluting Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Dilation of Left Peroneal Artery, Bifurcation, with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach— eluting Intraluminal Device, Percutaneous Endoscopic Approach—eluting Intraluminal Device, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous E |
| 047U3G6 or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— 047U3Z2 - Dilation of Left Peroneal Artery, Bifurcation, with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach—eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach—eluting Intraluminal Device, Percutaneous Endoscopic Approach—eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach—eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach— |
| Dilation of Left Peroneal Artery with Four or More Intraluminal Devices, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— O47U3ZZ Dilation of Left Peroneal Artery, Bifurcation, with Drugeluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Intraluminal Devices, Percutaneous Approach— |
| Dilation of Left Peroneal Artery, Bifurcation, Percutaneous Approach— Dilation of Left Peroneal Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| 047U3ZZ - Dilation of Left Peroneal Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Dilation of Left Peroneal Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Dilation of Left Peroneal Artery, Bifurcation, with Drug- eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous-eluting Intraluminal Devices, Percutaneous-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous-eluting Intraluminal Devices, Percutaneous-eluting Intraluminal Devices, Percutaneous-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approach-eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous-eluting Intraluminal Devices, Percutaneous-eluting Intraluminal Devices, Percutaneous-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| 047U446 Endoscopic Approach Dilation of Left Peroneal Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approacheluting Intraluminal Device, Percutaneous Endoscopic 047U44Z Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Dilation of Left Peroneal Artery with Drug-eluting Intraluminal Device, Percutaneous Endoscopic Approacheluting Intraluminal Device, Percutaneous Endoscopic 047U44Z Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Intraluminal Device, Percutaneous Endoscopic Approach- eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| eluting Intraluminal Device, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| 047U44Z Approach Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Dilation of Left Peroneal Artery, Bifurcation, with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach-eluting Intraluminal Devices, Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Endoscopic Approach-eluting Intraluminal Devices, 047U456 Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| 047U456 Percutaneous Endoscopic Approach Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Dilation of Left Peroneal Artery with Two Drug-eluting Intraluminal Devices, Percutaneous Endoscopic Approach- |
| Intraluminal Devices, Percutaneous Endoscopic Approach- |
| eluting Intraluminal Devices, Percutaneous Endoscopic |
| 047U45Z Approach |
| Dilation of Left Peroneal Artery, Bifurcation, with Three |
| Drug-eluting Intraluminal Devices, Percutaneous |
| Endoscopic Approach-eluting Intraluminal Devices, |
| 047U466 Percutaneous Endoscopic Approach |
| Dilation of Left Peroneal Artery with Three Drug-eluting |
| Intraluminal Devices, Percutaneous Endoscopic Approach- |
| eluting Intraluminal Devices, Percutaneous Endoscopic |
| 047U46Z Approach |
| Dilation of Left Peroneal Artery, Bifurcation, with Four |
| or More Drug-eluting Intraluminal Devices, |
| Percutaneous Endoscopic Approach-eluting Intraluminal |
| 047U476 Devices, Percutaneous Endoscopic Approach |
| Dilation of Left Peroneal Artery with Four or More Drug |
| eluting Intraluminal Devices, Percutaneous Endoscopic |
| Approach-eluting Intraluminal Devices, Percutaneous |
| 047U47Z Endoscopic Approach Dilation of Loft Paragonal Actors, Diffusertion, with |
| Dilation of Left Peroneal Artery, Bifurcation, with |
| 047U4D6 Intraluminal Device, Percutaneous Endoscopic Approach— |
| Dilation of Left Peroneal Artery with Intraluminal |
| 047U4DZ Device, Percutaneous Endoscopic Approach— |


| Supplement Left Popilized Artery with Nonautologous Tissus Substitute, Open Approach— Supplement Left Popilized Artery with Nonautologous Tissus Substitute, Open Approach— Supplement Left Popilized Artery with Nonautologous Tissus Substitute, Percutaneous Approach— Supplement Left Popilized Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Popilized Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Popilized Artery with Nonautologous Tissus Substitute, Percutaneous Approach— Supplement Left Popilized Artery with Autologous Tissus Substitute, Percutaneous Approach— Supplement Left Popilized Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Popilized Artery with Nonautologous Tissus Substitute, Percutaneous Endoscopic Approach— Supplement Left Popilized Artery with Nonautologous Tissus Substitute, Percutaneous Endoscopic Approach— Supplement Left Popilized Artery with Nonautologous Tissus Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Appr | O4UNO7Z Supplement Left Popliteal Artery with Synthetic Substitute, Open Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Popliteal Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic O4UP37Z Approach— Autologous Tissue Substitute, Percutaneous Endoscopic O4UP47Z Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left |
|---|---|
| Supplement Left Popilized Artery with Nonautologous Tissus Substitute, Open Approach— Supplement Left Popilized Artery with Nonautologous Tissus Substitute, Open Approach— Supplement Left Popilized Artery with Nonautologous Tissus Substitute, Percutaneous Approach— Supplement Left Popilized Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Popilized Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Popilized Artery with Nonautologous Tissus Substitute, Percutaneous Approach— Supplement Left Popilized Artery with Autologous Tissus Substitute, Percutaneous Approach— Supplement Left Popilized Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Popilized Artery with Nonautologous Tissus Substitute, Percutaneous Endoscopic Approach— Supplement Left Popilized Artery with Nonautologous Tissus Substitute, Percutaneous Endoscopic Approach— Supplement Left Popilized Artery with Nonautologous Tissus Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Appr | Supplement Left Popliteal Artery with Synthetic Substitute, Open Approach O4UNOKZ Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Open Approach Supplement Left Popliteal Artery with Mutologous O4UN37Z Tissue Substitute, Percutaneous Approach Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Approach Supplement Left Popliteal Artery with Nonautologous O4UN31Z Substitute, Percutaneous Approach Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Approach Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Approach Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Endoscopic Approach Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach Supplement Right Anterior Tibial Artery |
| Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Open Approach Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Popen Approach Supplement Left Popiliteal Artery with Autologous Tissue Substitute, Popen Approach Supplement Left Popiliteal Artery with Synthetic Substitute, Percutaneous Approach Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Percutaneous Approach Supplement Left Popiliteal Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach Supplement Left Popiliteal Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach Supplement Left Popiliteal Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach Supplement Left Popiliteal Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach Supplement Left Popiliteal Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach Supplement Right Arterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach Supplement L | O4UNOJZ Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Popliteal Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Nonautologous O4UN4KZ Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Appr |
| Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Depen Approach Supplement Left Popiliteal Artery with Autologous Tissue Substitute, Percutaneous Approach Supplement Left Popiliteal Artery with Synthetic Substitute, Percutaneous Approach Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Percutaneous Approach Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Percutaneous Deproach Supplement Left Popiliteal Artery with Autologous O4UNATZ Tissue Substitute, Percutaneous Endoscopic Approach Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Fodoscopic Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach Supplement Left Anterior Tibial Artery with S | Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Popiliteal Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Popiliteal Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Popiliteal Artery with Autologous O4UNAYZ Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popiliteal Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Rig |
| OAUNOICZ Tissue Substitute, Open Approach— Supplement Left Poplitical Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Poplitical Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Poplitical Artery with Nonautologous Tissue Substitute, Percutaneous Approach— OAUNAIZ Supplement Left Poplitical Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Poplitical Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Poplitical Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Poplitical Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Poplitical Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— S | O4UNOKZ Tissue Substitute, Open Approach— Supplement Left Popliteal Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Synthetic O4UN47Z Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic O4UPO7Z Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic O4UP37Z Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic O4UP31Z O4UP37Z Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic O4UP47Z Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic O4UP47Z Supplement Right Anterior Tibial Artery with Synthet |
| Supplement Left Popiliteal Artery with Autologous O4UN372 Supplement Left Popiliteal Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popiliteal Artery with Autologous O4UN472 Supplement Left Popiliteal Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Approach— Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Percutaneous Polyulation Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Nutologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Art | Supplement Left Popliteal Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Supproach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Supproach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Supplement Left Anterior Tibial Artery with Autologous Supplement Left An |
| Tissue Substitute, Percutaneous Approach— Supplement Left Popiliteal Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Popiliteal Artery with Monautologous Tissue Substitute, Percutaneous Approach— Supplement Left Popiliteal Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Popiliteal Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popiliteal Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Popiliteal Artery with Monautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popiliteal Artery with Monautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Mutologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibia | DAUNATZ Tissue Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery With Autologous |
| Supplement telt Popitieal Artery with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement telt Popitieal Artery with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement telt Popitieal Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement telt Popitieal Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement telt Popitieal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement telt Popitieal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Sendoscopic Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— S | Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic |
| Supplement Left Popilteal Artery with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Popilteal Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Popilteal Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popilteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popilteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute. Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Autologous Tissue Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous | O4UN3IZ Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Nonautologous O4UN4IZ Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous |
| Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Percutaneous Approach Supplement Left Popiliteal Artery with Autologous PalunATZ Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endos | Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with O4UPOX Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous |
| Supplement Left Popiliteal Artery with Autologous OAUNAIZ Supplement Left Popiliteal Artery with Synthetic Supplement Left Popiliteal Artery with Synthetic Substitute, Percurateous Endoscopic Approach— Supplement Left Popiliteal Artery with Synthetic Substitute, Percurateous Endoscopic Approach— Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Percurateous Endoscopic Approach— Supplement Right Anterior Tibial Artery with OAUPO7Z Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percurateous Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percurateous Approach— Autologous Tissue Substitute, Percurateous Approach— Nonautologous Tissue Substitute, Percurateous Approach— Nonautologous Tissue Substitute, Percurateous Approach— Autologous Tissue Substitute, Percurateous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percurateous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percurateous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percurateous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percurateous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Nonautologous Tissue Substitute, Percuraneous Approach— Nonautologous Tissue Substitute, Percuraneous Approach— Nonautologous Tissue Substitute, Percuraneous Endoscopic Approach— Nonautologous Tissue Substitute, Percuraneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percuraneous Endoscopic Approach— Suppl | O4UN3KZ Tissue Substitute, Percutaneous Approach— Supplement Left Popliteal Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Nonautologous O4UN4KZ Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with O4UPO7Z Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic O4UP47Z Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Autologous Supplement Left Anterior Tibial Artery with Autologous |
| Supplement Left Popliteal Artery with Autologous 04UN47Z Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Supplement Right Anterior Tibial Artery with Synthetic Supplement Right Anterior Tibial Artery with Synthetic Supplement Right Anterior Tibial Artery with Synthetic Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute | Supplement Left Popliteal Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Nonautologous O4UN4KZ Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with O4UPO7Z Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic O4UPO1Z Substitute, Open Approach— Supplement Right Anterior Tibial Artery with O4UPOKZ Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with O4UP37Z Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic O4UP37Z Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic O4UP31Z Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous O4UP3KZ Approach— Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic O4UP47Z Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic O4UP47Z Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous |
| Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous O4UN4K2 Supplement Right Anterior Tibial Artery with Nonautologous Supplement Right Anterior Tibial Artery with Nonautologous Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutane | O4UN47Z Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Nonautologous O4UN4KZ Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with O4UPO7Z Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic O4UP47Z Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous |
| Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with O4UPO7Z Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Mutologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior T | Supplement Left Popliteal Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with O4UPO7Z Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Supplement Left Anterior Tibial Artery with Autologous |
| Substitute, Percutaneous Endoscopic Approach— Supplement Left Popiliteal Artery with Nonautologous Hissus Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Autologous Tissus Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissus Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissus Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissus Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissus Substitute, Percutaneous Approach— Autologous Tissus Substitute, Percutaneous Approach— Autologous Tissus Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissus Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Autologous Tissus Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute | O4UN4IZ Substitute, Percutaneous Endoscopic Approach— Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic O4UPOIZ Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with O4UP37Z Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic O4UP47Z Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Supplement Left Anterior Tibial Artery with Autologous |
| Supplement Left Popiliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with OAUPOXZ Supplement Right Anterior Tibial Artery with OAUPOXZ Supplement Right Anterior Tibial Artery with OAUPOXZ Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with OAUP37Z Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic App | Supplement Left Popliteal Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous |
| O4UPAKZ Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with O4UPOKZ Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with O4UP37Z Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Syn | O4UNAKZ Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous |
| Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Monautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Budupatz Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery wi | Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with O4UPOKZ Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with O4UP37Z Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic O4UP47Z Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Autologous Supplement Left Anterior Tibial Artery with Autologous |
| Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with O4UP37Z Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery wit | 04UP07Z Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic O4UP47Z Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous O4UP4KZ Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Supplement Left Anterior Tibial Artery with Autologous |
| Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement L | Supplement Right Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Right Anterior Tibial Artery with 04UP0KZ Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous |
| Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endosc | O4UPOIZ Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Autologous Tissue Substitute, Percutaneous Endoscopic O4UP47Z Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous O4UP4KZ Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous |
| Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percu | Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous O4UP4KZ Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous |
| 04UPOKZ Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous End | O4UPOKZ Nonautologous Tissue Substitute, Open Approach— Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic O4UP3JZ Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic O4UP47Z Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous |
| Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach Nonautologous Tissue Substitute, Percutaneous Approach Autologous Tissue Substitute, Percutaneous Approach Autologous Tissue Substitute, Percutaneous Endoscopic O4UP47Z Approach Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic O4UP4IZ Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ07Z Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ01Z Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ37Z Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ31Z Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ41Z Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ41Z Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Ar | Supplement Right Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic O4UP3JZ Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Autologous Tissue Substitute, Percutaneous Endoscopic O4UP47Z Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Supplement Left Anterior Tibial Artery with Autologous |
| Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ01Z Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ01Z Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ31Z Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ31Z Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ31Z Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ41Z Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ41Z Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ41Z Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ41Z Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Sy | Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Supplement Left Anterior Tibial Artery with Autologous |
| Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ01Z Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ01Z Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ31Z Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ31Z Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ31Z Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ41Z Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ41Z Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ41Z Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ41Z Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Sy | Autologous Tissue Substitute, Percutaneous Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Supplement Left Anterior Tibial Artery with Autologous |
| Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with | O4UP3JZ Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic O4UP47Z Approach— Supplement Right Anterior Tibial Artery with Synthetic O4UP4JZ Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous |
| Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with | Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Supplement Left Anterior Tibial Artery with Autologous |
| Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with | Nonautologous Tissue Substitute, Percutaneous Approach— Autologous Tissue Substitute, Percutaneous Endoscopic O4UP47Z Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Supplement Left Anterior Tibial Artery with Autologous |
| Approach— Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with | 04UP3KZ Approach— Autologous Tissue Substitute, Percutaneous Endoscopic 04UP47Z Approach— Supplement Right Anterior Tibial Artery with Synthetic 04UP4JZ Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous |
| 04UP47Z Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with OduQOIZ Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with | 04UP47Z Approach— Supplement Right Anterior Tibial Artery with Synthetic O4UP4JZ Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous |
| 04UP47Z Approach— Supplement Right Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with OduQOIZ Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with | 04UP47Z Approach— Supplement Right Anterior Tibial Artery with Synthetic O4UP4JZ Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous |
| Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous O4UQ07Z Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ01Z Substitute, Open Approach— Supplement Left Anterior Tibial Artery with O4UQ0KZ Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ31Z Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous O4UQ3KZ Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Autologous O4UQ47Z Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ41Z Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ41Z Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with Supplement Right Posterior Tibial Artery with | O4UP4JZ Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous |
| Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous O4UQ07Z Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ01Z Substitute, Open Approach— Supplement Left Anterior Tibial Artery with O4UQ0KZ Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ31Z Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous O4UQ3KZ Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Autologous O4UQ47Z Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ41Z Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic O4UQ41Z Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with Supplement Right Posterior Tibial Artery with | O4UP4JZ Substitute, Percutaneous Endoscopic Approach— Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous |
| Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous O4UQ3/Z Approach— Supplement Left Anterior Tibial Artery with Autologous O4UQ4/Z Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with Supplement Right Posterior Tibial Artery with | Supplement Right Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous |
| DAUQAYZ Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with O4UQOXZ Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with | 04UP4KZ Endoscopic Approach— Supplement Left Anterior Tibial Artery with Autologous |
| Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with O4UQ0KZ Supplement Left Anterior Tibial Artery with O4UQ0KZ Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous O4UQ3IZ Supplement Left Anterior Tibial Artery with Autologous O4UQ3KZ Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with | Supplement Left Anterior Tibial Artery with Autologous |
| Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with O4UQ0KZ Supplement Left Anterior Tibial Artery with O4UQ0KZ Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous O4UQ3IZ Supplement Left Anterior Tibial Artery with Autologous O4UQ3KZ Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with | Supplement Left Anterior Tibial Artery with Autologous |
| Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with 04UQ0KZ Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous 4 Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous 6 Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with Supplement Right Posterior Tibial Artery with | · |
| Supplement Left Anterior Tibial Artery with Synthetic Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Autologous O4UQ3KZ Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous O4UQ4KZ Endoscopic Approach— Supplement Right Posterior Tibial Artery with Supplement Right Posterior Tibial Artery with | |
| Substitute, Open Approach— Supplement Left Anterior Tibial Artery with 04UQ0KZ Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with | Supplement Left Anterior Tibial Artery with Synthetic |
| Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with | |
| Nonautologous Tissue Substitute, Open Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous 04UQ3KZ Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with Supplement Right Posterior Tibial Artery with | |
| Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous O4UQ3KZ Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with | |
| Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Autologous O4UQ47Z Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with Supplement Right Posterior Tibial Artery with | |
| Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Autologous O4UQ47Z Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with Supplement Right Posterior Tibial Artery with | |
| Substitute, Percutaneous Approach— Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Autologous O4UQ47Z Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous O4UQ4KZ Endoscopic Approach— Supplement Right Posterior Tibial Artery with | 11 |
| Nonautologous Tissue Substitute, Percutaneous Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with Supplement Right Posterior Tibial Artery with | |
| Approach— Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous O4UQ4KZ Endoscopic Approach— Supplement Right Posterior Tibial Artery with | |
| Supplement Left Anterior Tibial Artery with Autologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with | |
| Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with | |
| Supplement Left Anterior Tibial Artery with Synthetic Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with | |
| Substitute, Percutaneous Endoscopic Approach— Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with | |
| Supplement Left Anterior Tibial Artery with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach— Supplement Right Posterior Tibial Artery with | |
| Nonautologous Tissue Substitute, Percutaneous O4UQ4KZ Endoscopic Approach— Supplement Right Posterior Tibial Artery with | |
| 04UQ4KZ Endoscopic Approach— Supplement Right Posterior Tibial Artery with | |
| Supplement Right Posterior Tibial Artery with | |
| 04UR07Z Autologous Tissue Substitute, Open Approach— | 04UR07Z Autologous Tissue Substitute, Open Approach- |


| Dilation of Right Foot Vein, Open Approach— | |
|---|---|
| Percutaneous Approach— | |
| Dilation of Right Foot Vein, Percutaneous Approach- | |
| Dilation of Right Foot Vein with Intraluminal Device, | |
| Percutaneous Endoscopic Approach— | |
| Dilation of Right Foot Vein, Percutaneous Endoscopic | |
| Approach- | |
| Dilation of Left Foot Vein with Intraluminal Device, | |
| Open Approach- | |
| Dilation of Left Foot Vein, Open Approach- | |
| Dilation of Left Foot Vein with Intraluminal Device, | |
| Percutaneous Approach- | |
| Dilation of Left Foot Vein, Percutaneous Approach— | |
| Dilation of Left Foot Vein with Intraluminal Device, | |
| Percutaneous Endoscopic Approach— | |
| Dilation of Left Foot Vein, Percutaneous Endoscopic | |
| Approach | |
| · ' | |
| Approach- | |
| Dilation of Lower Vein, Open Approach | |
| Percutaneous Approach- | |
| Dilation of Lower Vein, Percutaneous Approach- | |
| · · | |
| Percutaneous Endoscopic Approach- | |
| Approach | |
| Extirpation of Matter from Right Femoral Vein, Open | |
| _ · · · _ | |
| _ · | |
| · | |
| Extirpation of Matter from Right Greater Saphenous | |
| Vein, Percutaneous Endoscopic Approach- | |
| Extirpation of Matter from Left Greater Saphenous | |
| Vein, Open Approach | |
| Extirpation of Matter from Left Greater Saphenous | |
| Vein, Percutaneous Endoscopic Approach- | |
| Extirpation of Matter from Right Lesser Saphenous Vein, | |
| 1 11 | |
| · ·· | |
| Approach Extirpation of Matter from Right Foot Vein, | |
| Approach- | |
| | Dilation of Right Foot Vein, Percutaneous Approach— Dilation of Right Foot Vein with Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Right Foot Vein, Percutaneous Endoscopic Approach— Dilation of Left Foot Vein with Intraluminal Device, Open Approach— Dilation of Left Foot Vein, Open Approach— Dilation of Left Foot Vein with Intraluminal Device, Percutaneous Approach— Dilation of Left Foot Vein Percutaneous Approach— Dilation of Left Foot Vein with Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Left Foot Vein with Intraluminal Device, Percutaneous Endoscopic Approach— Dilation of Lower Vein with Intraluminal Device, Open Approach— Dilation of Lower Vein, Open Approach— Dilation of Lower Vein, Open Approach— Dilation of Lower Vein, Percutaneous Approach— Dilation of Lower Vein, Percutaneous Approach— Dilation of Lower Vein with Intraluminal Device, Percutaneous Endoscopic Approach— Extirpation of Matter from Right Femoral Vein, Open Approach— Extirpation of Matter from Right Femoral Vein, Percutaneous Endoscopic Approach— Extirpation of Matter from Left Femoral Vein, Percutaneous Endoscopic Approach— Extirpation of Matter from Right Greater Saphenous Vein, Open Approach— Extirpation of Matter from Right Greater Saphenous Vein, Open Approach— Extirpation of Matter from Left Greater Saphenous Vein, Open Approach— Extirpation of Matter from Left Greater Saphenous Vein, Open Approach— Extirpation of Matter from Left Greater Saphenous Vein, Open Approach— Extirpation of Matter from Left Greater Saphenous Vein, Open Approach— Extirpation of Matter from Left Greater Saphenous Vein, Open Approach— |


| Replacement of Lower Vein with Autologous Tissue | |
|---|---|
| Substitute, Percutaneous Endoscopic Approach | |
| 1 ' | |
| Replacement of Lower Vein with Nonautologous Tissue | |
| Substitute, Percutaneous Endoscopic Approach— | |
| Reposition Inferior Vena Cava, Open Approach- | |
| Reposition Inferior Vena Cava, Percutaneous Approach- | |
| Reposition Inferior Vena Cava, Percutaneous Endoscopic | _ |
| Approach | |
| Reposition Splenic Vein, Open Approach | |
| Reposition Splenic Vein, Percutaneous Approach- | |
| Reposition Splenic Vein, Percutaneous Endoscopic | |
| Approach | |
| Reposition Gastric Vein, Open Approach | |
| Reposition Gastric Vein, Percutaneous Approach- | |
| Reposition Gastric Vein, Percutaneous Endoscopic | |
| Approach | |
| Reposition Esophageal Vein, Open Approach— | |
| Reposition Esophageal Vein, Percutaneous Approach— | |
| Reposition Esophageal Vein, Percutaneous Endoscopic | |
| Approach | |
| Reposition Hepatic Vein, Open Approach- | |
| Reposition Hepatic Vein, Percutaneous Approach— | |
| Reposition Hepatic Vein, Percutaneous Endoscopic | |
| Approach | |
| Reposition Superior Mesenteric Vein, Open Approach- | |
| Reposition Superior Mesenteric Vein, Percutaneous | |
| ' | |
| Endoscopic Approach- | |
| Reposition Colic Vein, Open Approach | |
| Reposition Colic Vein, Percutaneous Approach- | |
| Approach | |
| • | |
| 7 1 11 | |
| 7 | |
| 1 | |
| 1 | |
| 1 ' 1 | |
| 1 ' | |
| | Substitute, Percutaneous Endoscopic Approach— Reposition Inferior Vena Cava, Open Approach— Reposition Inferior Vena Cava, Percutaneous Approach— Reposition Inferior Vena Cava, Percutaneous Endoscopic Approach— Reposition Splenic Vein, Open Approach— Reposition Splenic Vein, Percutaneous Approach— Reposition Splenic Vein, Percutaneous Endoscopic Approach— Reposition Gastric Vein, Open Approach— Reposition Gastric Vein, Percutaneous Approach— Reposition Gastric Vein, Percutaneous Approach— Reposition Esophageal Vein, Percutaneous Endoscopic Approach— Reposition Esophageal Vein, Percutaneous Approach— Reposition Esophageal Vein, Percutaneous Endoscopic Approach— Reposition Hepatic Vein, Open Approach— Reposition Hepatic Vein, Percutaneous Approach— Reposition Hepatic Vein, Percutaneous Endoscopic Approach— Reposition Superior Mesenteric Vein, Open Approach— Reposition Superior Mesenteric Vein, Percutaneous Endoscopic Approach— Reposition Superior Mesenteric Vein, Percutaneous Endoscopic Approach— Reposition Inferior Mesenteric Vein, Percutaneous Endoscopic Approach— Reposition Inferior Mesenteric Vein, Percutaneous Endoscopic Approach— Reposition Inferior Mesenteric Vein, Percutaneous Approach— Reposition Inferior Mesenteric Vein, Percutaneous Approach— Reposition Inferior Mesenteric Vein, Percutaneous Approach— Reposition Inferior Mesenteric Vein, Percutaneous Approach— Reposition Inferior Mesenteric Vein, Percutaneous Endoscopic Approach— Reposition Inferior Mesenteric Vein, Percutaneous Endoscopic Approach— Reposition Colic Vein, Open Approach— |


35372


#### Comorbid conditions

| Comorbia | C |
|----------|---|
| 35381 | 1 |
| 35454 | 1 |
| 35456 | 1 |
| 35459 | 1 |
| 35470 | 1 |
| 35473 | 1 |
| 35474 | 1 |
| 35482 | 1 |
| 35483 | 1 |
| 35485 | 1 |
| 35492 | 1 |
| 35493 | 1 |
| 35495 | 1 |
| 35521 | 1 |
| 35533 | |
| 35556 | |
| 35558 | |
| 35563 | |
| 35565 | |
| 35566 | |
| 35571 | |
| 35621 | |
| 35623 | |
| 35641 | |
| 35646 | |
| 35647 | |
| 35650 | |
| 35651 | |
| 35654 | |
| 35656 | |
| 35661 | |
| 35663 | |
| 35666 | |
| 35671 | |

Hypertension

| ICD10 Dx | ICD9 Dx | LongDeslCD10 | LongDeslCD9 |
|---|---|---|---|
| 110 | 4010 | Essential (primary) hypertension | Malignant essential hypertension |
| I10 | 4011 | Essential (primary) hypertension | Benign essential hypertension |
| 110 | 4019 | Essential (primary) hypertension | Unspecified essential hypertension |
| 1160 | 4019 | Hypertensive urgency | Unspecified essential hypertension |
| l161 | 4019 | Hypertensive emergency | Unspecified essential hypertension |
| I169 | 4019 | Hypertensive crisis, unspecified | Unspecified essential hypertension |
| l119 | 40200 | Hypertensive heart disease without heart failure | Malignant hypertensive heart disease without heart |
| l110 | 40201 | Hypertensive heart disease with heart failure | Malignant hypertensive heart disease with heart |
| l119 | 40210 | Hypertensive heart disease without heart failure | Benign hypertensive heart disease without heart |
| l110 | 40211 | Hypertensive heart disease with heart failure | Benign hypertensive heart disease with heart failure |
| 1119 | 40290 | Hypertensive heart disease without heart failure | Unspecified hypertensive heart disease without heart |
| | | | failure |
| I110 | 40291 | Hypertensive heart disease with heart failure | Unspecified hypertensive heart disease with heart |
| 1129 | 40300 | Hypertensive chronic kidney disease with stage 1 | Hypertensive chronic kidney disease, malignant, with |
| | | through stage 4 chronic kidney disease, or unspecified | chronic kidney disease stage I through stage IV, or |
| | | chronic kidney disease | unspecified |

585

#### Comorbid conditions

| 1120 | 40301 | Hypertensive chronic kidney disease with stage 5 | Hypertensive chronic kidney disease, malignant, with |
|---|---|---|---|
| | | chronic kidney disease or end stage renal disease | chronic kidney disease stage V or end stage renal |
| 1129 | 40310 | Hypertensive chronic kidney disease with stage 1 | Hypertensive chronic kidney disease, benign, with |
| | | through stage 4 chronic kidney disease, or unspecified | chronic kidney disease stage I through stage IV, or |
| | | chronic kidney disease | unspecified |
| 1120 | 40311 | Hypertensive chronic kidney disease with stage 5 | Hypertensive chronic kidney disease, benign, with |
| | | chronic kidney disease or end stage renal disease | chronic kidney disease stage V or end stage renal |
| 1129 | 40390 | Hypertensive chronic kidney disease with stage 1 | Hypertensive chronic kidney disease, unspecified, with |
| | | through stage 4 chronic kidney disease, or unspecified | chronic kidney disease stage I through stage IV, or |
| | | chronic kidney disease | unspecified |
| I120 | 40391 | Hypertensive chronic kidney disease with stage 5 | Hypertensive chronic kidney disease, unspecified, with |
| | | chronic kidney disease or end stage renal disease | chronic kidney disease stage V or end stage renal |
| I1310 | 40400 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, |
| | | heart failure, with stage 1 through stage 4 chronic | malignant, without heart failure and with chronic |
| | | kidney disease, or unspecified chronic kidney disease | kidney disease stage I through stage IV, or unspecified |
| I130 | 40401 | Hypertensive heart and chronic kidney disease with | Hypertensive heart and chronic kidney disease, |
| | | heart failure and stage 1 through stage 4 chronic kidney | malignant, with heart failure and with chronic kidney |
| | | disease, or unspecified chronic kidney disease | disease stage I through stage IV, or unspecified |
| l1311 | 40402 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, |
| | | heart failure, with stage 5 chronic kidney disease, or end | malignant, without heart failure and with chronic |
| | | stage renal disease | kidney disease stage V or end stage renal disease |
| l132 | 40403 | Hypertensive heart and chronic kidney disease with | Hypertensive heart and chronic kidney disease, |
| | | heart failure and with stage 5 chronic kidney disease, or | malignant, with heart failure and with chronic kidney |
| | | end stage renal disease | disease stage V or end stage renal disease |
| I1310 | 40410 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, benign, |
| | | heart failure, with stage 1 through stage 4 chronic | without heart failure and with chronic kidney disease |
| | | kidney disease, or unspecified chronic kidney disease | stage I through stage IV, or unspecified |
| I130 | 40411 | Hypertensive heart and chronic kidney disease with | Hypertensive heart and chronic kidney disease, benign, |
| | | heart failure and stage 1 through stage 4 chronic kidney | |
| | | disease, or unspecified chronic kidney disease | stage I through stage IV, or unspecified |
| l1311 | 40412 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, benign, |
| | | heart failure, with stage 5 chronic kidney disease, or end | |
| | | stage renal disease | stage V or end stage renal disease |
| l132 | 40413 | Hypertensive heart and chronic kidney disease with | Hypertensive heart and chronic kidney disease, benign, |
| | 10.120 | heart failure and with stage 5 chronic kidney disease, or | with heart failure and chronic kidney disease stage V |
| | | end stage renal disease | or end stage renal disease |
| l1310 | 40490 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, |
| .2020 | 10.50 | heart failure, with stage 1 through stage 4 chronic | unspecified, without heart failure and with chronic |
| | | kidney disease, or unspecified chronic kidney disease | kidney disease stage I through stage IV, or unspecified |
| l130 | 40491 | Hypertensive heart and chronic kidney disease with | Hypertensive heart and chronic kidney disease, |
| 1130 | 40431 | heart failure and stage 1 through stage 4 chronic kidney | unspecified, with heart failure and with chronic kidney |
| | | disease, or unspecified chronic kidney disease | disease stage I through stage IV, or unspecified |
| l1311 | 40492 | Hypertensive heart and chronic kidney disease without | Hypertensive heart and chronic kidney disease, |
| 11311 | 40432 | heart failure, with stage 5 chronic kidney disease, or end | |
| | | stage renal disease | kidney disease stage V or end stage renal disease |
| l132 | 40493 | Hypertensive heart and chronic kidney disease with | Hypertensive heart and chronic kidney disease, |
| 1132 | 40493 | heart failure and with stage 5 chronic kidney disease, or | unspecified, with heart failure and chronic kidney |
| | | | disease stage V or end stage renal disease |
| 1150 | 40501 | end stage renal disease Renovascular hypertension | |
| 1150<br> 1158 | 40501 | Other secondary hypertension | Malignant renovascular hypertension Other malignant secondary hypertension |
| 1150 | 40503 | Renovascular hypertension | Benign renovascular hypertension |
| I158 | 40519 | Other secondary hypertension | Other benign secondary hypertension |
| 1150 | 40591 | Renovascular hypertension | Unspecified renovascular hypertension |
| l151 | 40591 | Hypertension secondary to other renal disorders | Unspecified renovascular hypertension |
| N262 | 40591 | Page kidney | Unspecified renovascular hypertension |
| l152 | 40599 | Hypertension secondary to endocrine disorders | Other unspecified secondary hypertension |
| I158 | 40599 | Other secondary hypertension | Other unspecified secondary hypertension |
| l159 | 40599 | Secondary hypertension, unspecified | Other unspecified secondary hypertension |

#### Diabetes


#### Comorbid conditions


Hyperlipidem ia

| | турстиристи | | |
|---|---|---|---|
| ICD10 Dx | ICD9 Dx | LongDeslCD10 | LongDeslCD9 |
| E780 | 2720 | Pure hypercholesterolemia | PURE HYPERCHOLESTEROLEMIA |
| E7800 | 2722 | | MIXED HYPERLIPIDEMIA |
| E781 | 2724 | Pure hyperglyceridemia | OTHER AND UNSPECIFIED HYPERLIPIDEMIA |
| E782 | | Mixed hyperlipidemia | |
| E784 | | Other hyperlipidemia | |
| E785 | | Hyperlipidemia, unspecified | |

Renal dysfunction


| 5011101.D.G | 00 | • | |
|---|---|---|---|
| N008 | 5810 | Acute nephritic syndrome with other morphologic | NEPHROTIC SYNDROME WITH LESION OF |
| | | changes | PROLIFERATIVE GLOMERULONEPHRITIS |
| N009 | 5811 | Acute nephritic syndrome with unspecified morphologic | NEPHROTIC SYNDROME WITH LESION OF |
| | | changes | MEMBRANOUS GLOMERULONEPHRITIS |
| N010 | 5812 | Rapidly progressive nephritic syndrome with minor | NEPHROTIC SYNDROME WITH LESION OF |
| | | glomerular abnormality | MEMBRANOPROLIFERATIVE GLOMERULONEPHRITIS |
| N011 | 5813 | Rapidly progressive nephritic syndrome with focal and | NEPHROTIC SYNDROME WITH LESION OF MINIMAL |
| | | segmental glomerular lesions | CHANGE GLOMERULONEPHRITIS |
| N012 | 5818 | Rapidly progressive nephritic syndrome with diffuse | NEPHROTIC SYNDROME WITH OTHER SPECIFIED |
| | | membranous glomerulonephritis | PATHOLOGICAL LESION IN KIDNEY |
| N013 | 58181 | Rapidly progressive nephritic syndrome with diffuse | NEPHROTIC SYNDROME IN DISEASES CLASSIFIED |
| | | mesangial proliferative glomerulonephritis | ELSEWHERE |
| N014 | 58189 | Rapidly progressive nephritic syndrome with diffuse | OTHER NEPHROTIC SYNDROME WITH SPECIFIED |
| | | endocapillary proliferative glomerulonephritis | PATHOLOGICAL LESION IN KIDNEY |
| N015 | 5819 | Rapidly progressive nephritic syndrome with diffuse | NEPHROTIC SYNDROME WITH UNSPECIFIED |
| | | mesangiocapillary glomerulonephritis | PATHOLOGICAL LESION IN KIDNEY |
| N016 | 5820 | Rapidly progressive nephritic syndrome with dense | CHRONIC GLOMERULONEPHRITIS WITH LESION OF |
| | | deposit disease | PROLIFERATIVE GLOMERULONEPHRITIS |
| N017 | 5821 | Rapidly progressive nephritic syndrome with diffuse | CHRONIC GLOMERULONEPHRITIS WITH LESION OF |
| | | crescentic glomerulonephritis | MEMBRANOUS GLOMERULONEPHRITIS |
| N018 | 5822 | Rapidly progressive nephritic syndrome with other | CHRONIC GLOMERULONEPHRITIS WITH LESION OF |
| | 3022 | morphologic changes | MEMBRANOPROLIFERATIVE GLOMERULONEPHRITIS |
| N019 | 5824 | Rapidly progressive nephritic syndrome with unspecified | |
| NOIS | 3024 | morphologic changes | RAPIDLY PROGRESSIVE GLOMERULONEPHRITIS |
| N020 | 5828 | Recurrent and persistent hematuria with minor | CHRONIC GLOMERULONEPHRITIS WITH OTHER |
| 11020 | 3020 | glomerular abnormality | SPECIFIED PATHOLOGICAL LESION IN KIDNEY |
| N021 | 5829 | , | CHRONIC GLOMERULONEPHRITIS WITH UNSPECIFIED |
| NUZI | 5829 | Recurrent and persistent hematuria with focal and segmental glomerular lesions | |
| NOSS | 5830 | | PATHOLOGICAL LESION IN KIDNEY |
| N022 | 5830 | Recurrent and persistent hematuria with diffuse | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS |
| | | membranous glomerulonephritis | ACUTE OR CHRONIC WITH LESION OF PROLIFERATIVE |
| 11000 | 5004 | D | GLOMERULONEPHRITIS |
| N023 | 5831 | Recurrent and persistent hematuria with diffuse | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS |
| | | mesangial proliferative glomerulonephritis | ACUTE OR CHRONIC WITH LESION OF MEMBRANOUS |
| 1100.4 | 5000 | D | GLOMERULONEPHRITIS |
| N024 | 5832 | Recurrent and persistent hematuria with diffuse | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS |
| | | endocapillary proliferative glomerulonephritis | ACUTE OR CHRONIC WITH LESION OF |
| | | | MEMBRANOPROLIFERATIVE GLOMERULONEPHRITIS |
| N025 | 5834 | Recurrent and persistent hematuria with diffuse | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS |
| | | mesangiocapillary glomerulonephritis | ACUTE OR CHRONIC WITH LESION OF RAPIDLY |
| | | | PROGRESSIVE GLOMERULONEPHRITIS |
| N026 | 5836 | Recurrent and persistent hematuria with dense deposit | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS |
| | | disease | ACUTE OR CHRONIC WITH LESION OF RENAL CORTICAL |
| N027 | 5837 | Recurrent and persistent hematuria with diffuse | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS |
| | | crescentic glomerulonephritis | ACUTE OR CHRONIC WITH LESION OF RENAL |
| N028 | 5838 | Recurrent and persistent hematuria with other | NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS |
| | 5555 | | |
| | | morphologic changes | ACUTE OR CHRONIC WITH OTHER SPECIFIED |
| | 3333 | morphologic changes | ACUTE OR CHRONIC WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY |
| N029 | 5839 | morphologic changes Recurrent and persistent hematuria with unspecified | |
| | | | PATHOLOGICAL LESION IN KIDNEY |
| | | Recurrent and persistent hematuria with unspecified | PATHOLOGICAL LESION IN KIDNEY NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS |
| | | Recurrent and persistent hematuria with unspecified | PATHOLOGICAL LESION IN KIDNEY NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL |
| N029 | 5839 | Recurrent and persistent hematuria with unspecified morphologic changes | PATHOLOGICAL LESION IN KIDNEY NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS |
| N029 | 5839 | Recurrent and persistent hematuria with unspecified morphologic changes Chronic nephritic syndrome with minor glomerular | PATHOLOGICAL LESION IN KIDNEY NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL |
| N029<br>N030 | 5839<br>5846 | Recurrent and persistent hematuria with unspecified morphologic changes Chronic nephritic syndrome with minor glomerular abnormality | PATHOLOGICAL LESION IN KIDNEY NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS |
| N029<br>N030 | 5839<br>5846 | Recurrent and persistent hematuria with unspecified morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental | PATHOLOGICAL LESION IN KIDNEY NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL |
| N029<br>N030<br>N031 | 5839<br>5846<br>5847 | Recurrent and persistent hematuria with unspecified morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions | PATHOLOGICAL LESION IN KIDNEY NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLARY (PAPILLARY) NECROSIS |
| N029<br>N030<br>N031 | 5839<br>5846<br>5847 | Recurrent and persistent hematuria with unspecified morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous | PATHOLOGICAL LESION IN KIDNEY NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLARY (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED |
| N029<br>N030<br>N031<br>N032 | 5839<br>5846<br>5847<br>5848 | Recurrent and persistent hematuria with unspecified morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous glomerulonephritis | PATHOLOGICAL LESION IN KIDNEY NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLARY (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY |
| N029<br>N030<br>N031<br>N032 | 5839<br>5846<br>5847<br>5848 | Recurrent and persistent hematuria with unspecified morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous glomerulonephritis Chronic nephritic syndrome with diffuse mesangial | PATHOLOGICAL LESION IN KIDNEY NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLARY (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY |
| N029<br>N030<br>N031<br>N032 | 5839<br>5846<br>5847<br>5848<br>5849 | Recurrent and persistent hematuria with unspecified morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous glomerulonephritis Chronic nephritic syndrome with diffuse mesangial proliferative glomerulonephritis | PATHOLOGICAL LESION IN KIDNEY NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLARY (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE UNSPECIFIED |
| N029<br>N030<br>N031<br>N032 | 5839<br>5846<br>5847<br>5848<br>5849 | Recurrent and persistent hematuria with unspecified morphologic changes Chronic nephritic syndrome with minor glomerular abnormality Chronic nephritic syndrome with focal and segmental glomerular lesions Chronic nephritic syndrome with diffuse membranous glomerulonephritis Chronic nephritic syndrome with diffuse mesangial proliferative glomerulonephritis Chronic nephritic syndrome with diffuse endocapillary | PATHOLOGICAL LESION IN KIDNEY NEPHRITIS AND NEPHROPATHY NOT SPECIFIED AS ACUTE OR CHRONIC WITH UNSPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE WITH LESION OF RENAL CORTICAL NECROSIS ACUTE KIDNEY FAILURE WITH LESION OF RENAL MEDULLARY (PAPILLARY) NECROSIS ACUTE KIDNEY FAILURE WITH OTHER SPECIFIED PATHOLOGICAL LESION IN KIDNEY ACUTE KIDNEY FAILURE UNSPECIFIED |

| N037<br>N038 | 5854 | Chronic nephritic syndrome with diffuse crescentic | CURONIC VIDNEY DICEACE CTACE IV (CEVEDE) |
|---|---|---|---|
| | | | CHRONIC KIDNEY DISEASE STAGE IV (SEVERE) |
| | | glomerulonephritis | |
| *1000 | 5855 | Chronic nephritic syndrome with other morphologic changes | CHRONIC KIDNEY DISEASE STAGE V |
| N039 | 5856 | Chronic nephritic syndrome with unspecified morphologic changes | END STAGE RENAL DISEASE |
| N040 | 5859 | Nephrotic syndrome with minor glomerular abnormality | CHRONIC KIDNEY DISEASE UNSPECIFIED |
| N041 | 86600 | Nephrotic syndrome with focal and segmental glomerular lesions | UNSPECIFIED INJURY TO KIDNEY WITHOUT OPEN WOUND INTO CAVITY |
| N042 | 86601 | Nephrotic syndrome with diffuse membranous glomerulonephritis | HEMATOMA OF KIDNEY WITHOUT RUPTURE OF CAPSULE WITHOUT OPEN WOUND INTO CAVITY |
| N043 | 8661 | Nephrotic syndrome with diffuse mesangial proliferative glomerulonephritis | |
| N044 | | Nephrotic syndrome with diffuse endocapillary proliferative glomerulonephritis | |
| N045 | | Nephrotic syndrome with diffuse mesangiocapillary glomerulonephritis | |
| N046 | | Nephrotic syndrome with dense deposit disease | |
| N047 | | Nephrotic syndrome with diffuse crescentic | |
| | | glomerulonephritis | |
| N048 | | Nephrotic syndrome with other morphologic changes | |
| N049 | | Nephrotic syndrome with unspecified morphologic | |
| N050 | | Unspecified nephritic syndrome with minor glomerular | |
| | | abnormality | |
| N051 | | Unspecified nephritic syndrome with focal and | |
| | | segmental glomerular lesions | |
| N052 | | Unspecified nephritic syndrome with diffuse | |
| | | membranous glomerulonephritis | |
| N053 | | Unspecified nephritic syndrome with diffuse mesangial | |
| | | proliferative glomerulonephritis | |
| N054 | | Unspecified nephritic syndrome with diffuse | |
| | | endocapillary proliferative glomerulonephritis | |
| N055 | | Unspecified nephritic syndrome with diffuse | |
| | | mesangiocapillary glomerulonephritis | |
| N056 | | Unspecified nephritic syndrome with dense deposit | |
| N057 | | Unspecified nephritic syndrome with diffuse crescentic | |
| | | glomerulonephritis | |
| N058 | | Unspecified nephritic syndrome with other morphologic | |
| 11050 | | changes | |
| N059 | | Unspecified nephritic syndrome with unspecified | |
| NOSO | | morphologic changes Isolated proteinuria with minor glomerular abnormality | |
| N060<br>N061 | | Isolated proteinuria with minor glomerular abnormality Isolated proteinuria with focal and segmental | |
| MOOT | | glomerular lesions | |
| N062 | | Isolated proteinuria with diffuse membranous | |
| .1002 | | glomerulonephritis | |
| N063 | | Isolated proteinuria with diffuse mesangial proliferative | |
| | | glomerulonephritis | |
| N064 | | Isolated proteinuria with diffuse endocapillary | |
| | | proliferative glomerulonephritis | |
| N065 | | Isolated proteinuria with diffuse mesangiocapillary | |
| | | glomerulonephritis | |
| N066 | | Isolated proteinuria with dense deposit disease | |
| | | Isolated proteinuria with diffuse crescentic | |
| N067 | | glomerulonephritis | |
| N067 | | Isolated proteinuria with other morphologic lesion | |
| N067<br>N068 | | isolated proteinura with other morphologic lesion | |
| | | Isolated proteinuria with other morphologic lesion | |
| N068 | | | |
| N068<br>N069 | | Isolated proteinuria with unspecified morphologic lesion | |

| Comorbia conc | JILIO 15 | |
|---|---|---|
| N072 | Hereditary nephropathy, not elsewhere classified with diffuse membranous glomerulonephritis | |
| N073 | Hereditary nephropathy, not elsewhere classified with | |
| N074 | diffuse mesangial proliferative glomerulonephritis Hereditary nephropathy, not elsewhere classified with | |
| | diffuse endocapillary proliferative glomerulonephritis | |
| N075 | Hereditary nephropathy, not elsewhere classified with | |
| | diffuse mesangiocapillary glomerulonephritis | |
| N076 | Hereditary nephropathy, not elsewhere classified with dense deposit disease | |
| N077 | Hereditary nephropathy, not elsewhere classified with diffuse crescentic glomerulonephritis | |
| N078 | Hereditary nephropathy, not elsewhere classified with other morphologic lesions | |
| N079 | Hereditary nephropathy, not elsewhere classified with | |
| 1100 | unspecified morphologic lesions | |
| N08 | Glomerular disorders in diseases classified elsewhere | |
| N140 | Analgesic nephropathy | |
| N141 | Nephropathy induced by other drugs, medicaments and biological substances | |
| N142 | Nephropathy induced by unspecified drug, medicament or biological substance | |
| N143 | Nephropathy induced by heavy metals | |
| N144 | Toxic nephropathy, not elsewhere classified | |
| N150 | Balkan nephropathy | |
| N158 | Other specified renal tubulo-interstitial diseases | |
| N159 | Renal tubulo-interstitial disease, unspecified | |
| N16 | Renal tubulo-interstitial disorders in diseases classified elsewhere | |
| N171 | Acute kidney failure with acute cortical necrosis | |
| N172 | Acute kidney failure with medullary necrosis | |
| N178 | Other acute kidney failure | |
| N179 | Acute kidney failure, unspecified | |
| N181 | Chronic kidney disease, stage 1 | |
| N182 | Chronic kidney disease, stage 2 (mild) | |
| N183 | Chronic kidney disease, stage 3 (moderate) | |
| N184 | Chronic kidney disease, stage 4 (severe) | |
| N185 | Chronic kidney disease, stage 5 | |
| N186 | End stage renal disease | |
| N189 | Chronic kidney disease, unspecified | |
| N19 | Unspecified kidney failure | |
| N261 | Atrophy of kidney (terminal) | |
| N269 | Renal sclerosis, unspecified | |
| S31001A | Unspecified open wound of lower back and pelvis with | |
| C27004 A | penetration into retroperitoneum, initial encounter | |
| \$37001A | Unspecified injury of left kidney, initial encounter | |
| \$37002A | Unspecified injury of left kidney, initial encounter | |
| \$37009A | Unspecified injury of unspecified kidney, initial | |
| S37011A<br>S37012A | Minor contusion of right kidney, initial encounter | |
| S37012A<br>S37019A | Minor contusion of left kidney, initial encounter | |
| S37019A<br>S37021A | Minor contusion of unspecified kidney, initial encounter Major contusion of right kidney, initial encounter | |
| S37021A<br>S37022A | Major contusion of left kidney, initial encounter | |
| S37022A | Major contusion of unspecified kidney, initial encounter | |
| S37029A<br>S37039A | Laceration of unspecified kidney, unspecified degree, | |
| | initial encounter | |
| S37049A | Minor laceration of unspecified kidney, initial encounter | |
| S37059A | Moderate laceration of unspecified kidney, initial encounter | |
| S37069A | Major laceration of unspecified kidney, initial encounter | |
| Z4931 | Encounter for adequacy testing for hemodialysis | |
| Z4932 | Encounter for adequacy testing for peritoneal dialysis | |
| <u> </u> | | • |

#### Comorbid conditions

| ICD10 Px | ICD9 Px | LongDesICD10 | LongDeslCD9 |
|---|---|---|---|
| 3E1M39Z | 3995 | Irrigation of Peritoneal Cavity using Dialysate, | HEMODIALYSIS |
| | | Percutaneous Approach | |
| 5A1D00Z | 5498 | Performance of Urinary Filtration, Single | PERITONEAL DIALYSIS |
| 5A1D60Z | | Performance of Urinary Filtration, Multiple | |
| HCPCS | | | |
| 90935 | | | |
| 90937 | | | |
| 90939 | | | |
| 90940 | | | |
| 90945 | | | |
| 90947 | | | |
| 90951 | | | |
| 90952 | | | |
| 90953 | | | |
| 90954 | | | |
| 90955 | | | |
| 90956 | | | |
| 90957 | | | |
| 90958 | | | |
| 90959 | | | |
| 90960 | | | |
| 90961 | | | |
| 90962 | | | |
| 90963 | | | |
| 90964 | | | |
| 90965 | | | |
| 90966 | | | |
| 90967 | | | |
| 90968 | | | |
| 90969 | | | |
| 90970 | | | |
| 90989 | | | |
| 90993 | | | |
| 99512 | | | |

Chronic liver disease

99559


#### Comorbid conditions

| K7211 | 5732 | Chronic hepatic failure with coma | HEPATITIS IN OTHER INFECTIOUS DISEASES CLASSIFIED ELSEWHERE |
|---|---|---|---|
| K7290 | 5733 | Hepatic failure, unspecified without coma | HEPATITIS UNSPECIFIED |
| K7291 | 5734 | Hepatic failure, unspecified with coma | HEPATIC INFARCTION |
| K730 | 5735 | Chronic persistent hepatitis, not elsewhere classified | HEPATOPULMONARY SYNDROME |
| K731 | 5738 | Chronic lobular hepatitis, not elsewhere classified | OTHER SPECIFIED DISORDERS OF LIVER |
| K732 | 5739 | Chronic active hepatitis, not elsewhere classified | UNSPECIFIED DISORDER OF LIVER |
| K738 | | Other chronic hepatitis, not elsewhere classified | |
| K739 | | Chronic hepatitis, unspecified | |
| K740 | | Hepatic fibrosis | |
| K741 | | Hepatic sclerosis | |
| K742 | | Hepatic fibrosis with hepatic sclerosis | |
| K743 | | Primary biliary cirrhosis | |
| K744 | | Secondary biliary cirrhosis | |
| K745 | | Biliary cirrhosis, unspecified | |
| K7460 | | Unspecified cirrhosis of liver | |
| K7469 | | Other cirrhosis of liver | |
| K750 | | Abscess of liver | |
| K751 | | Phlebitis of portal vein | |
| K752 | | Nonspecific reactive hepatitis | |
| K753 | | Granulomatous hepatitis, not elsewhere classified | |
| K754 | | Autoimmune hepatitis | |
| K7581 | | Nonalcoholic steatohepatitis (NASH) | |
| K7589 | | Other specified inflammatory liver diseases | |
| K759 | | Inflammatory liver disease, unspecified | |
| K760 | | Fatty (change of) liver, not elsewhere classified | |
| K761 | | Chronic passive congestion of liver | |
| K763 | | Infarction of liver | |
| K764 | | Peliosis hepatis | |
| K765 | | Hepatic veno-occlusive disease | |
| K766 | | Portal hypertension | |
| K767 | | Hepatorenal syndrome | |
| K7681 | | Hepatopulmonary syndrome | |
| K7689 | | Other specified diseases of liver | |
| K769 | | Liver disease, unspecified | |
| K77 | | Liver disorders in diseases classified elsewhere | |

<u>Asthma</u>


#### Comorbid conditions

| J45991 | 49392 | Cough variant asthma | ASTHMA UNSPECIFIED WITH (ACUTE) EXACERBATION |
|---|---|---|---|
| J45998 | | Other asthma | |

Ischemic heart disease

## Comorbid conditions


### COPD

| ICD10 Dx | ICD9 Dx | LongDeslCD10 | LongDeslCD9 |
|---|---|---|---|
| J40 | 490 | Bronchitis, not specified as acute or chronic | BRONCHITIS NOT SPECIFIED AS ACUTE OR CHRONIC |
| J410 | 491 | Simple chronic bronchitis | CHRONIC BRONCHITIS |
| J411 | 4910 | Mucopurulent chronic bronchitis | SIMPLE CHRONIC BRONCHITIS |
| J418 | 4911 | Mixed simple and mucopurulent chronic bronchitis | MUCOPURULENT CHRONIC BRONCHITIS |
| J42 | 4912 | Unspecified chronic bronchitis | OBSTRUCTIVE CHRONIC BRONCHITIS |
| J430 | 49120 | Unilateral pulmonary emphysema [MacLeod's | OBSTRUCTIVE CHRONIC BRONCHITIS WITHOUT |
| | | syndrome] | EXACERBATION |
| J431 | 49121 | Panlobular emphysema | OBSTRUCTIVE CHRONIC BRONCHITIS WITH (ACUTE) |
| | | | EXACERBATION |
| J432 | 49122 | Centrilobular emphysema | OBSTRUCTIVE CHRONIC BRONCHITIS WITH ACUTE |
| | | | BRONCHITIS |
| J438 | 4918 | Other emphysema | OTHER CHRONIC BRONCHITIS |
| J439 | 4919 | Emphysema, unspecified | UNSPECIFIED CHRONIC BRONCHITIS |
| J440 | 492 | Chronic obstructive pulmonary disease with acute lower | EMPHYSEMA |
| | | respiratory infection | |
| J441 | 4920 | Chronic obstructive pulmonary disease with (acute) | EMPHYSEMATOUS BLEB |
| | | exacerbation | |
| J449 | 4928 | Chronic obstructive pulmonary disease, unspecified | OTHER EMPHYSEMA |
| J470 | 494 | Bronchiectasis with acute lower respiratory infection | BRONCHIECTASIS |
| J471 | 4940 | Bronchiectasis with (acute) exacerbation | BRONCHIECTASIS WITHOUT ACUTE EXACERBATION |
| J479 | 4941 | Bronchiectasis, uncomplicated | BRONCHIECTASIS WITH ACUTE EXACERBATION |

| Ī | 496 | CHRONIC AIRWAY OBSTRUCTION NOT ELSEWHERE |
|---|-----|------------------------------------------|
| | | CLASSIFIED |

Occurence of malignancy

| Occurence of r | malignancy | | |
|---|---|---|---|
| ICD10 Dx | ICD9 Dx | LongDeslCD10 | LongDesiCD9 |
| C000 | 140 | Malignant neoplasm of external upper lip | MALIGNANT NEOPLASM OF LIP |
| C001 | 1400 | Malignant neoplasm of external lower lip | MALIGNANT NEOPLASM OF UPPER LIP VERMILION |
| C002 | 1401 | Malignant neoplasm of external lip, unspecified | MALIGNANT NEOPLASM OF LOWER LIP VERMILION |
| C003 | 1403 | Malignant neoplasm of upper lip, inner aspect | MALIGNANT NEOPLASM OF UPPER LIP INNER ASPECT |
| C004 | 1404 | Malignant neoplasm of lower lip, inner aspect | MALIGNANT NEOPLASM OF LOWER LIP INNER ASPECT |
| C005 | 1405 | Malignant neoplasm of lip, unspecified, inner aspect | MALIGNANT NEOPLASM OF LIP UNSPECIFIED INNER |
| | | | ASPECT |
| C006 | 1406 | Malignant neoplasm of commissure of lip, unspecified | MALIGNANT NEOPLASM OF COMMISSURE OF LIP |
| C008 | 1408 | Malignant neoplasm of overlapping sites of lip | MALIGNANT NEOPLASM OF OTHER SITES OF LIP |
| C009 | 1409 | Malignant neoplasm of lip, unspecified | MALIGNANT NEOPLASM OF LIP UNSPECIFIED |
| 2003 | 1103 | Wangilane neoplasii of hp, anspeaned | VERMILION BORDER |
| C01 | 141 | Malignant neoplasm of base of tongue | MALIGNANT NEOPLASM OF TONGUE |
| C020 | 1410 | Malignant neoplasm of dorsal surface of tongue | MALIGNANT NEOPLASM OF BASE OF TONGUE |
| C020 | 1411 | Malignant neoplasm of border of tongue | MALIGNANT NEOFLASM OF DORSAL SURFACE OF |
| C021 | 1412 | Malignant neoplasm of ventral surface of tongue | MALIGNANT NEOFLASM OF TIP AND LATERAL BORDER |
| C022 | 1412 | Walighant heopiasin of ventral surface of torigue | OF TONGUE |
| CO22 | 1413 | Malignant noonlasm of antorior two thirds of tonguo | MALIGNANT NEOPLASM OF VENTRAL SURFACE OF |
| C023 | 1413 | Malignant neoplasm of anterior two-thirds of tongue, | |
| 602.4 | 4444 | part unspecified | TONGUE |
| C024 | 1414 | Malignant neoplasm of lingual tonsil | MALIGNANT NEOPLASM OF ANTERIOR TWO-THIRDS |
| 0000 | 4445 | | OF TONGUE PART UNSPECIFIED |
| C028 | 1415 | Malignant neoplasm of overlapping sites of tongue | MALIGNANT NEOPLASM OF JUNCTIONAL ZONE OF |
| | | | TONGUE |
| C029 | 1416 | Malignant neoplasm of tongue, unspecified | MALIGNANT NEOPLASM OF LINGUAL TONSIL |
| C030 | 1418 | Malignant neoplasm of upper gum | MALIGNANT NEOPLASM OF OTHER SITES OF TONGUE |
| C031 | 1419 | Malignant neoplasm of lower gum | MALIGNANT NEOPLASM OF TONGUE UNSPECIFIED |
| C039 | 142 | Malignant neoplasm of gum, unspecified | MALIGNANT NEOPLASM OF MAJOR SALIVARY |
| C040 | 1420 | Malignant neoplasm of anterior floor of mouth | MALIGNANT NEOPLASM OF PAROTID GLAND |
| C041 | 1421 | Malignant neoplasm of lateral floor of mouth | MALIGNANT NEOPLASM OF SUBMANDIBULAR GLAND |
| C048 | 1422 | Malignant neoplasm of overlapping sites of floor of | MALIGNANT NEOPLASM OF SUBLINGUAL GLAND |
| C049 | 1428 | Malignant neoplasm of floor of mouth, unspecified | MALIGNANT NEOPLASM OF OTHER MAJOR SALIVARY |
| | | | GLANDS |
| C050 | 1429 | Malignant neoplasm of hard palate | MALIGNANT NEOPLASM OF SALIVARY GLAND |
| | | | UNSPECIFIED |
| C051 | 143 | Malignant neoplasm of soft palate | MALIGNANT NEOPLASM OF GUM |
| C052 | 1430 | Malignant neoplasm of uvula | MALIGNANT NEOPLASM OF UPPER GUM |
| C058 | 1431 | Malignant neoplasm of overlapping sites of palate | MALIGNANT NEOPLASM OF LOWER GUM |
| C059 | 1438 | Malignant neoplasm of palate, unspecified | MALIGNANT NEOPLASM OF OTHER SITES OF GUM |
| C060 | 1439 | Malignant neoplasm of cheek mucosa | MALIGNANT NEOPLASM OF GUM UNSPECIFIED |
| C061 | 144 | Malignant neoplasm of vestibule of mouth | MALIGNANT NEOPLASM OF FLOOR OF MOUTH |
| C062 | 1440 | Malignant neoplasm of retromolar area | MALIGNANT NEOPLASM OF ANTERIOR PORTION OF |
| | | | FLOOR OF MOUTH |
| C0680 | 1441 | Malignant neoplasm of overlapping sites of unspecified | MALIGNANT NEOPLASM OF LATERAL PORTION OF |
| | | parts of mouth | FLOOR OF MOUTH |
| C0689 | 1448 | Malignant neoplasm of overlapping sites of other parts | MALIGNANT NEOPLASM OF OTHER SITES OF FLOOR |
| | | of mouth | OF MOUTH |
| C069 | 1449 | Malignant neoplasm of mouth, unspecified | MALIGNANT NEOPLASM OF FLOOR OF MOUTH PART |
| | | | UNSPECIFIED |
| C07 | 145 | Malignant neoplasm of parotid gland | MALIGNANT NEOPLASM OF OTHER AND UNSPECIFIED |
| | | | PARTS OF MOUTH |
| C080 | 1450 | Malignant neoplasm of submandibular gland | MALIGNANT NEOPLASM OF CHEEK MUCOSA |
| C081 | 1451 | Malignant neoplasm of sublingual gland | MALIGNANT NEOPLASM OF VESTIBULE OF MOUTH |
| C089 | 1452 | Malignant neoplasm of major salivary gland, unspecified | MALIGNANT NEOPLASM OF HARD PALATE |
| 0000 | 1453 | Malignant neoplasm of tonsillar fossa | MALIGNANT NEOPLASM OF SOFT PALATE |
| C090 | 1-00 | | |
| C090<br>C091 | 1454 | Malignant neoplasm of tonsillar pillar (anterior) | MALIGNANT NEOPLASM OF UVULA |
| | | Malignant neoplasm of tonsillar pillar (anterior) Malignant neoplasm of overlapping sites of tonsil | MALIGNANT NEOPLASM OF UVULA MALIGNANT NEOPLASM OF PALATE UNSPECIFIED |

| | | I | |
|---|---|---|---|
| C100 | 1458 | Malignant neoplasm of vallecula | MALIGNANT NEOPLASM OF OTHER SPECIFIED PARTS |
| | | | OF MOUTH |
| C101 | 1459 | Malignant neoplasm of anterior surface of epiglottis | MALIGNANT NEOPLASM OF MOUTH UNSPECIFIED |
| C102 | 146 | Malignant neoplasm of lateral wall of oropharynx | MALIGNANT NEOPLASM OF OROPHARYNX |
| C103 | 1460 | Malignant neoplasm of posterior wall of oropharynx | MALIGNANT NEOPLASM OF TONSIL |
| C104 | 1461 | Malignant neoplasm of branchial cleft | MALIGNANT NEOPLASM OF TONSILLAR FOSSA |
| C108 | 1462 | Malignant neoplasm of overlapping sites of oropharynx | MALIGNANT NEOPLASM OF TONSILLAR PILLARS |
| | | | (ANTERIOR) (POSTERIOR) |
| C109 | 1463 | Malignant neoplasm of oropharynx, unspecified | MALIGNANT NEOPLASM OF VALLECULA EPIGLOTTICA |
| C110 | 1464 | Malignant neoplasm of superior wall of nasopharynx | MALIGNANT NEOPLASM OF ANTERIOR ASPECT OF |
| | | | EPIGLOTTIS |
| C111 | 1465 | Malignant neoplasm of posterior wall of nasopharynx | MALIGNANT NEOPLASM OF JUNCTIONAL REGION OF |
| | | | OROPHARYNX |
| C112 | 1466 | Malignant neoplasm of lateral wall of nasopharynx | MALIGNANT NEOPLASM OF LATERAL WALL OF |
| | | | OROPHARYNX |
| C113 | 1467 | Malignant neoplasm of anterior wall of nasopharynx | MALIGNANT NEOPLASM OF POSTERIOR WALL OF |
| | | | OROPHARYNX |
| C118 | 1468 | Malignant neoplasm of overlapping sites of nasopharynx | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES |
| | | The state of the s | OF OROPHARYNX |
| C119 | 1469 | Malignant neoplasm of nasopharynx, unspecified | MALIGNANT NEOPLASM OF OROPHARYNX |
| 0113 | 1103 | Wanghant neoplasm of hasophary my anspeamed | UNSPECIFIED SITE |
| C12 | 147 | Malignant neoplasm of pyriform sinus | MALIGNANT NEOPLASM OF NASOPHARYNX |
| C120 | 1470 | Malignant neoplasm of postcricoid region | MALIGNANT NEOPLASM OF SUPERIOR WALL OF |
| C130 | 1470 | Manghant heopiasin of posturcold region | |
| 6424 | 4.474 | Malta and an allow of a control of the | NASOPHARYNX |
| C131 | 1471 | Malignant neoplasm of aryepiglottic fold, | MALIGNANT NEOPLASM OF POSTERIOR WALL OF |
| | | hypopharyngeal aspect | NASOPHARYNX |
| C132 | 1472 | Malignant neoplasm of posterior wall of hypopharynx | MALIGNANT NEOPLASM OF LATERAL WALL OF |
| | | | NASOPHARYNX |
| C138 | 1473 | Malignant neoplasm of overlapping sites of | MALIGNANT NEOPLASM OF ANTERIOR WALL OF |
| | | hypopharynx | NASOPHARYNX |
| C139 | 1478 | Malignant neoplasm of hypopharynx, unspecified | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES |
| | | | OF NASOPHARYNX |
| C140 | 1479 | Malignant neoplasm of pharynx, unspecified | MALIGNANT NEOPLASM OF NASOPHARYNX |
| | | | UNSPECIFIED SITE |
| C142 | 148 | Malignant neoplasm of Waldeyer's ring | MALIGNANT NEOPLASM OF HYPOPHARYNX |
| C148 | 1480 | Malignant neoplasm of overlapping sites of lip, oral | MALIGNANT NEOPLASM OF POSTCRICOID REGION O |
| | | cavity and pharynx | HYPOPHARYNX |
| C153 | 1481 | Malignant neoplasm of upper third of esophagus | MALIGNANT NEOPLASM OF PYRIFORM SINUS |
| C154 | 1482 | Malignant neoplasm of middle third of esophagus | MALIGNANT NEOPLASM OF ARYEPIGLOTTIC FOLD |
| | | | HYPOPHARYNGEAL ASPECT |
| C155 | 1483 | Malignant neoplasm of lower third of esophagus | MALIGNANT NEOPLASM OF POSTERIOR |
| | | | HYPOPHARYNGEAL WALL |
| C158 | 1488 | Malignant neoplasm of overlapping sites of esophagus | MALIGNANT NEOPLASM OF OTHER SPECIFIED SITES |
| | | | OF HYPOPHARYNX |
| C159 | 1489 | Malignant neoplasm of esophagus, unspecified | MALIGNANT NEOPLASM OF HYPOPHARYNX |
| | | | UNSPECIFIED SITE |
| C160 | 149 | Malignant neoplasm of cardia | MALIGNANT NEOPLASM OF OTHER AND ILL-DEFINED |
| 0200 | 2.5 | manghant neophasm or car ara | SITES WITHIN THE LIP ORAL CAVITY AND PHARYNX |
| C161 | 1490 | Malignant neoplasm of fundus of stomach | MALIGNANT NEOPLASM OF PHARYNX UNSPECIFIED |
| C162 | 1491 | Malignant neoplasm of body of stomach | MALIGNANT NEOPLASM OF PHARTIX ONSFECTIVE MALIGNANT NEOPLASM OF WALDEYER'S RING |
| C162 | 1491 | Malignant neoplasm of pyloric antrum | MALIGNANT NEOPLASM OF WALDETER'S KING MALIGNANT NEOPLASM OF OTHER SITES WITHIN TI |
| C102 | 1430 | ivianguant neopiasin of pyrotic and uni | LIP AND ORAL CAVITY |
| C164 | 1/100 | Malignant noonlasm of pulgrus | MALIGNANT NEOPLASM OF ILL-DEFINED SITES WITH |
| C104 | 1499 | Malignant neoplasm of pylorus | |
| 64.65 | 450 | Maliana da canda con effectiva | THE LIP AND ORAL CAVITY |
| C165 | 150 | Malignant neoplasm of lesser curvature of stomach, | MALIGNANT NEOPLASM OF ESOPHAGUS |
| | | unspecified | |
| C166 | 1500 | Malignant neoplasm of greater curvature of stomach, | MALIGNANT NEOPLASM OF CERVICAL ESOPHAGUS |
| | | unspecified | |
| C168 | 1501 | Malignant neoplasm of overlapping sites of stomach | MALIGNANT NEOPLASM OF THORACIC ESOPHAGUS |
| | i e | lastic contract to the contract of the contrac | • |
| C169 | 1502 | Malignant neoplasm of stomach, unspecified | MALIGNANT NEOPLASM OF ABDOMINAL ESOPHAGE |

| C171 |
|---|
| C172 1505 Malignant neoplasm of ielum MALIGNANT NEOPLASM OF LOWER THIBD |
| C173 1508 Meckel's diverticulum, malignant MALIGMANT NEOPLASM OF OTHER SPECIF OF ESOPHAGUS L intestine C179 151 Malignant neoplasm of overlapping sites of small MALIGMANT NEOPLASM OF ESOPHAGUS L Intestine C180 1510 Malignant neoplasm of small intestine, unspecified MALIGMANT NEOPLASM OF STOMACH C180 1511 Malignant neoplasm of scerum MALIGMANT NEOPLASM OF STOMACH C181 1511 Malignant neoplasm of ascending colon MALIGMANT NEOPLASM OF PYLORIC ANTR C182 1512 Malignant neoplasm of specific flexure MALIGMANT NEOPLASM OF PYLORIC ANTR C183 1513 Malignant neoplasm of specific flexure MALIGMANT NEOPLASM OF FUCORIC ANTR C184 1514 Malignant neoplasm of specific flexure MALIGMANT NEOPLASM OF FUCORIC ANTR C184 1515 Malignant neoplasm of specific flexure MALIGMANT NEOPLASM OF EUROSJO OF STOMACH UNSPECIFIED MALIGMANT NEOPLASM OF BOOLY OF STOMACH UNSPECIFIED MALIGMANT NEOPLASM OF GREATER CURVA STOMACH UNSPECIFIED MALIGMANT NEOPLASM OF GREATER CURVA STOMACH UNSPECIFIED MALIGMANT NEOPLASM OF GREATER CURVA STOMACH UNSPECIFIED MALIGMANT NEOPLASM OF GREATER CURVA STOMACH UNSPECIFIED MALIGMANT NEOPLASM OF GREATER CURVA STOMACH UNSPECIFIED MALIGMANT NEOPLASM OF STOMACH UNSPECIFIED OF STOMACH UNSPECIFIED MALIGMANT NEOPLASM OF STOMACH UNSPECIFIED OF STOMACH UNSPECIFIED MALIGMANT NEOPLASM OF STOMACH UNSPECIFIED OF STOMACH UNSPECIFIED MALIGMANT NEOPLASM OF STOMACH UNSPECIFIED OF STOMACH UNSPECIFIED MALIGMANT NEOPLASM OF STOMACH UNSPECIFIED OF STOMAC |
| C178 1509 Malignant neoplasm of overlapping sites of small MALIGNANT NEOPLASM OF ESOPHAGUS Unitestine STE C179 151 Malignant neoplasm of small intestine, unspecified MALIGNANT NEOPLASM OF STOMACH C180 1510 Malignant neoplasm of appendix MALIGNANT NEOPLASM OF STOMACH C181 1511 Malignant neoplasm of appendix MALIGNANT NEOPLASM OF PYLORUS C182 1512 Malignant neoplasm of appendix MALIGNANT NEOPLASM OF PYLORUS C183 1513 Malignant neoplasm of specific flexure MALIGNANT NEOPLASM OF PYLORUS C184 1514 Malignant neoplasm of frepatic flexure MALIGNANT NEOPLASM OF PURDIX OF STOMACH C185 1515 Malignant neoplasm of specific flexure MALIGNANT NEOPLASM OF BUNDUS OF STOM MALIGNANT NEOPLASM OF EURDUS OF STOMACH UNSPECIFIED STOMACH UNSPECIFIED STOMACH UNSPECIFIED STOMACH UNSPECIFIED OF STOMACH C185 1516 Malignant neoplasm of specific flexure STOMACH UNSPECIFIED OF STOMACH UNSPECIFIED OF STOMACH C185 1518 Malignant neoplasm of solverlapping sites of colon MALIGNANT NEOPLASM OF OTHER SPECIFICAL STOMACH UNSPECIFIED OF STOMACH C189 152 Malignant neoplasm of overlapping sites of colon MALIGNANT NEOPLASM OF STOMACH UNSPECIFIED OF STOMACH C189 152 Malignant neoplasm of rectosigmoid junction MALIGNANT NEOPLASM OF STOMACH UNSPECIFIED STOMACH C189 152 Malignant neoplasm of rectosigmoid junction MALIGNANT NEOPLASM OF EURUNUM C20 1521 Malignant neoplasm of anus, unspecified MALIGNANT NEOPLASM OF EURUNUM C210 1522 Malignant neoplasm of anus, unspecified MALIGNANT NEOPLASM OF EURUNUM C210 1522 Malignant neoplasm of anus can be supported to the MALIGNANT NEOPLASM OF FROM STOMACH C210 1522 Malignant neoplasm of of unspecified MALIGNANT NEOPLASM OF FROM STOMACH C210 1522 Malignant neoplasm of of unspecified MALIGNANT NEOPLASM OF FROM STOMACH C210 1522 Malignant neoplasm of inspecified MALIGNANT NEOPLASM OF FROM STOMACH C210 1522 Malignant neoplasm of of unspecified MALIGNANT NEOPLASM OF FROM STOMACH C210 1522 Malignant neoplasm of of unspecified MALIGNANT NEOPLASM OF STOMACH C221 1533 Unterell cardioma MALIGNANT NEOPLASM OF STOMACH C222 1533 Hepa |
| C178 1509 Malignant neoplasm of overlapping sites of small intestine. C179 151 Malignant neoplasm of small intestine, unspecified MALIGNANT NEOPLASM OF STOMACH C180 1510 Malignant neoplasm of cacum MALIGNANT NEOPLASM OF CARDIA C181 1511 Malignant neoplasm of ascending colon MALIGNANT NEOPLASM OF PYLORIC ANTR C182 1512 Malignant neoplasm of ascending colon MALIGNANT NEOPLASM OF PYLORIC ANTR C183 1513 Malignant neoplasm of hepatic flexure MALIGNANT NEOPLASM OF PYLORIC ANTR C184 1514 Malignant neoplasm of fransverse colon MALIGNANT NEOPLASM OF PULORIC ANTR C184 1515 Malignant neoplasm of splenic flexure MALIGNANT NEOPLASM OF BOYO OF STOM MALIGNANT NEOPLASM OF EDVOY OF STOM MALIGNANT NEOPLASM OF EDVOY OF STOM MALIGNANT NEOPLASM OF EDVOY OF STOMACH UNSPECIFIED MALIGNANT NEOPLASM OF GREATER CURVA STOMACH UNSPECIFIED MALIGNANT NEOPLASM OF GREATER CURVA STOMACH UNSPECIFIED MALIGNANT NEOPLASM OF GREATER CURVA STOMACH UNSPECIFIED MALIGNANT NEOPLASM OF GREATER CURVA STOMACH UNSPECIFIED MALIGNANT NEOPLASM OF OTHER SPECIFIC OF STOMACH UNSPECIFIED MALIGNANT NEOPLASM OF STOMACH UNSPECIFIED STOMACH UNSPECIFIED MALIGNANT NEOPLASM OF STOMACH UNSPECIFIED STOMACH |
| Intestine |
| C179 151 Malignant neoplasm of small intestine, unspecified MAUGNANT NEOPLASM OF STOMACH C180 1510 Malignant neoplasm of secum MAUGNANT NEOPLASM OF PYLORUS C182 1512 Malignant neoplasm of ascending colon MAUGNANT NEOPLASM OF PYLORUS C183 1513 Malignant neoplasm of hepatic flexure MAUGNANT NEOPLASM OF PYLORUS OF STOMACH C183 1513 Malignant neoplasm of transverse colon MAUGNANT NEOPLASM OF PYLORUS OF STOMACH UNSPECIFIED MALIGNANT NEOPLASM OF BYLORUS OF STOMACH UNSPECIFIED STEE C185 Malignant neoplasm of splenic flexure MAUGNANT NEOPLASM OF BODY OF STOM C185 1516 Malignant neoplasm of splenic flexure MAUGNANT NEOPLASM OF BODY OF STOM C186 TSOMACH UNSPECIFIED MALIGNANT NEOPLASM OF GREATER CURVA STOMACH UNSPECIFIED MALIGNANT NEOPLASM OF GREATER CURVA STOMACH UNSPECIFIED MALIGNANT NEOPLASM OF GREATER CURVA STOMACH UNSPECIFIED MALIGNANT NEOPLASM OF GREATER CURVA STOMACH UNSPECIFIED MALIGNANT NEOPLASM OF STOMACH UNSPECIFIED OF STOMACH UNSPECIFIED MALIGNANT NEOPLASM OF STOMACH UNSPECIFIED OF STOMACH UNSPECIFIED MALIGNANT NEOPLASM OF STOMACH UNSPECIFIED OF STOMACH UNSPECIFI |
| C180 1510 Malignant neoplasm of cecum MALIGNANT NEOPLASM OF CARDIA C181 1511 Malignant neoplasm of appendix MALIGNANT NEOPLASM OF PYLORIC ANTR C182 1512 Malignant neoplasm of aspending colon MALIGNANT NEOPLASM OF PYLORIC ANTR C183 1513 Malignant neoplasm of hepatic flexure MALIGNANT NEOPLASM OF PULDRUS OF STOM C184 1514 Malignant neoplasm of penatic flexure MALIGNANT NEOPLASM OF BODY OF STOM STOMACH UNSPECIFIED MALIGNANT NEOPLASM OF EDSY OF STOM MALIGNANT NEOPLASM OF LESSER CURVA STOMACH UNSPECIFIED C186 1516 Malignant neoplasm of descending colon MALIGNANT NEOPLASM OF LESSER CURVA STOMACH UNSPECIFIED C187 1518 Malignant neoplasm of sigmoid colon MALIGNANT NEOPLASM OF LESSER CURVA STOMACH UNSPECIFIED C187 1518 Malignant neoplasm of overlapping sites of colon MALIGNANT NEOPLASM OF OTHER SPECIFICATION OF STOMACH UNSPECIFIED C188 1519 Malignant neoplasm of overlapping sites of colon MALIGNANT NEOPLASM OF STOMACH UNSPECIFIED C188 1519 Malignant neoplasm of overlapping sites of colon MALIGNANT NEOPLASM OF STOMACH UNSPECIFICATION OF STOMACH UNSPECIFIED C189 152 Malignant neoplasm of rectosigmoid junction MALIGNANT NEOPLASM OF STOMACH UNSPECIFICATION OF STOMACH UNSPECIFIED C19 1520 Malignant neoplasm of rectom MALIGNANT NEOPLASM OF JELIUNUM C210 1521 Malignant neoplasm of rectum MALIGNANT NEOPLASM OF JELIUNUM C210 1522 Malignant neoplasm of overlapping sites of rectum, MALIGNANT NEOPLASM OF JELIUNUM C211 1523 Malignant neoplasm of doacogenic zone MALIGNANT NEOPLASM OF DILUDENCE C11 1523 Malignant neoplasm of overlapping sites of rectum, MALIGNANT NEOPLASM OF OTHER SPECIFICATION OF SMALL INTESTINE MALIGNANT NEOPLASM OF SMALL INTESTINE MALIGNANT N |
| C181 1511 Malignant neoplasm of appendix MALIGNANT NEOPLASM OF PYLORUS C182 1512 Malignant neoplasm of appendix MALIGNANT NEOPLASM OF PYLORUS OR TICLUS OF STORY C183 1513 Malignant neoplasm of hepatic flexure MALIGNANT NEOPLASM OF FUNDUS OF STORY C184 1514 Malignant neoplasm of transverse colon MALIGNANT NEOPLASM OF FUNDUS OF STORY C185 1515 Malignant neoplasm of splenic flexure MALIGNANT NEOPLASM OF BODY OF STORY C186 1516 Malignant neoplasm of descending colon MALIGNANT NEOPLASM OF GREATER CURVA STOMACH UNSPECIFIED C187 1518 Malignant neoplasm of sigmoid colon MALIGNANT NEOPLASM OF GREATER CURVA STOMACH UNSPECIFIED C188 1519 Malignant neoplasm of overlapping sites of colon MALIGNANT NEOPLASM OF OTHER SPECIFIC OF STOMACH C189 152 Malignant neoplasm of colon, unspecified MALIGNANT NEOPLASM OF STOMACH UNSPECIFIED C19 1520 Malignant neoplasm of rectosigmoid junction MALIGNANT NEOPLASM OF SMALL INTEST INCLUDING DUDDENUM C20 1521 Malignant neoplasm of rectosigmoid junction MALIGNANT NEOPLASM OF JEJUNUM C210 1522 Malignant neoplasm of rectosigmoid junction MALIGNANT NEOPLASM OF JEJUNUM C211 1523 Malignant neoplasm of anal canal MALIGNANT NEOPLASM OF JEJUNUM C212 1528 Malignant neoplasm of anal canal MALIGNANT NEOPLASM OF MECKEL'S DIV. C212 1528 Malignant neoplasm of doacogenic zone MALIGNANT NEOPLASM OF MECKEL'S DIV. C213 1529 Malignant neoplasm of overlapping sites of rectum, MALIGNANT NEOPLASM OF MECKEL'S DIV. C214 1529 Malignant neoplasm of overlapping sites of mectum. MALIGNANT NEOPLASM OF SMALL INTEST UNSPECIFIED SITE C220 153 Liver cell cardinoma MALIGNANT NEOPLASM OF SMALL INTEST UNSPECIFIED SITE C221 1530 Intrahepatic bile duct cardinoma MALIGNANT NEOPLASM OF SMALL INTEST UNSPECIFIED SITE C222 1531 Hepatoblastoma MALIGNANT NEOPLASM OF FOLION OF SMALL INTEST UNSPECIFIED SITE C224 1533 Other specified cardinomas of liver MALIGNANT NEOPLASM OF FOLION OF SPECIFIC PLEXI. C224 1533 Other specified arcinomas of liver MALIGNANT NEOPLASM OF FOLION OF SPECIFIC C224 1533 Other specified arcinomas of liver MALIGNANT NEO |
| C182 1512 Malignant neoplasm of ascending colon MALIGNANT NEOPLASM OF PYLORIC ANTR C183 1513 Malignant neoplasm of hepatic flexure MALIGNANT NEOPLASM OF POLOSAN OF STOM C185 1515 Malignant neoplasm of splenic flexure MALIGNANT NEOPLASM OF BODY OF STOM C185 1515 Malignant neoplasm of splenic flexure MALIGNANT NEOPLASM OF LESSER CURVA STOMACH UNSPECIFIED C186 1516 Malignant neoplasm of descending colon MALIGNANT NEOPLASM OF GREATER CURVA STOMACH UNSPECIFIED C187 1518 Malignant neoplasm of sigmoid colon MALIGNANT NEOPLASM OF OTHER SPECIFIC OF STOMACH UNSPECIFIED C188 1519 Malignant neoplasm of overlapping sites of colon MALIGNANT NEOPLASM OF STOMACH UNSPECIFIED C189 152 Malignant neoplasm of rectoming sites of colon MALIGNANT NEOPLASM OF STOMACH UNSPECIFIED C19 1520 Malignant neoplasm of rectosigmoid junction MALIGNANT NEOPLASM OF DUODENUM MALIGNANT NEOPLASM OF DUODENUM MALIGNANT NEOPLASM OF DUODENUM MALIGNANT NEOPLASM OF DUODENUM MALIGNANT NEOPLASM OF ILLIUM MALIGNANT NEOPLASM OF MECKEL'S DIVI 1522 Malignant neoplasm of anal canal MALIGNANT NEOPLASM OF MECKEL'S DIVI 1523 Malignant neoplasm of overlapping sites of rectum, MALIGNANT NEOPLASM OF MECKEL'S DIVI 1524 Malignant neoplasm of overlapping sites of rectum, MALIGNANT NEOPLASM OF MECKEL'S DIVI 1525 MALIGNANT NEOPLASM OF MECKEL'S DIVI 1526 Malignant neoplasm of illium MALIGNANT NEOPLASM OF SMALL INTEST INC. C210 1531 User cell carcinoma MALIGNANT NEOPLASM OF SMALL INTEST INC. C221 1530 Intrahepatic bile duct carcinoma MALIGNANT NEOPLASM OF SMALL INTEST INC. C222 1531 Hepatoblastoma MALIGNANT NEOPLASM OF SECRIONING OF SMALL INTEST INC. C223 1532 Analignant neoplasm of liver MALIGNANT NEOPLASM OF SIGMOID COLO 1524 Malignant neoplasm of liver, primary, unspecified as to MALIGNANT NEOPLASM OF SECRIONING OF SECONDARY OF SECRIONIN |
| C183 1513 Malignant neoplasm of hepatic flexure MAUGNANT NEOPLASM OF FUNDUS OF STORM C184 1514 Malignant neoplasm of transverse colon MAUGNANT NEOPLASM OF EBDY OF STORM C185 1515 Malignant neoplasm of splenic flexure MAUGNANT NEOPLASM OF LESSER CURVA STOMACH UNSPECIFIED C186 1516 Malignant neoplasm of splenic flexure MAUGNANT NEOPLASM OF GREATER CURVA STOMACH UNSPECIFIED C187 1518 Malignant neoplasm of sigmoid colon MAUGNANT NEOPLASM OF OTHER SPECIFICATION OF STOMACH UNSPECIFIED C188 1519 Malignant neoplasm of overlapping sites of colon MAUGNANT NEOPLASM OF STOMACH UNSPECIFIED C188 1519 Malignant neoplasm of rectosigmoid junction MAUGNANT NEOPLASM OF STOMACH UNSPECIFIED OF STO |
| C184 1514 Malignant neoplasm of transverse colon C185 1515 Malignant neoplasm of splenic flexure C186 1516 Malignant neoplasm of splenic flexure C186 1516 Malignant neoplasm of descending colon C187 1518 Malignant neoplasm of descending colon C187 1518 Malignant neoplasm of sigmoid colon C188 1519 Malignant neoplasm of sigmoid colon C188 1519 Malignant neoplasm of overlapping sites of colon C189 152 Malignant neoplasm of overlapping sites of colon C189 1520 Malignant neoplasm of rectosigmoid junction C19 1520 Malignant neoplasm of rectosigmoid junction C20 1521 Malignant neoplasm of rectosigmoid junction C210 1522 Malignant neoplasm of anus, unspecified MALIGNANT NEOPLASM OF DUDDENUM C210 1522 Malignant neoplasm of anus, unspecified MALIGNANT NEOPLASM OF JUDDENUM C210 1522 Malignant neoplasm of anal canal MALIGNANT NEOPLASM OF JUDDENUM C211 1523 Malignant neoplasm of anal canal MALIGNANT NEOPLASM OF MECKEL'S DIV. C212 1528 Malignant neoplasm of overlapping sites of rectum, MALIGNANT NEOPLASM OF MECKEL'S DIV. C213 1529 Malignant neoplasm of overlapping sites of rectum, MALIGNANT NEOPLASM OF OF HEEAST DIV. C214 1520 Malignant neoplasm of overlapping sites of rectum, MALIGNANT NEOPLASM OF OTHER SPECIF. OF SMALL INTESTINE C220 1531 Liver cell carcinoma MALIGNANT NEOPLASM OF OTHER SPECIF. C221 1530 Intrahepatic bile duct carcinoma MALIGNANT NEOPLASM OF SMALL INTEST. C222 1531 Hepatolastoma MALIGNANT NEOPLASM OF SMALL INTEST. C222 1531 Hepatolastoma MALIGNANT NEOPLASM OF SIGMOID COLC C221 1530 Other sarcomas of liver MALIGNANT NEOPLASM OF DESCENDING OF MALIGNANT NEOPLASM OF OTHER SPECIF. C221 1530 Other sarcomas of liver MALIGNANT NEOPLASM OF DESCENDING OF MALIGNANT NEOPLASM OF OTHER SPECIF. C222 1531 Malignant neoplasm of liver, primary, unspecified as to MALIGNANT NEOPLASM OF OTHER SPECIF. C224 1539 Mal |
| C184 1514 Malignant neoplasm of transverse colon C185 1515 Malignant neoplasm of splenic flexure MALIGNANT NEOPLASM OF BODY OF STON STOMACH UNSPECIFIED C186 1516 Malignant neoplasm of descending colon MALIGNANT NEOPLASM OF GREATER CURVA STOMACH UNSPECIFIED C187 1518 Malignant neoplasm of sigmoid colon MALIGNANT NEOPLASM OF GREATER CURVA STOMACH UNSPECIFIED C187 1518 Malignant neoplasm of sigmoid colon MALIGNANT NEOPLASM OF OTHER SPECIFICO OF STOMACH C188 1519 Malignant neoplasm of overlapping sites of colon MALIGNANT NEOPLASM OF STOMACH UNCLUDING DUODENUM C189 1520 Malignant neoplasm of rectosigmoid junction MALIGNANT NEOPLASM OF STOMACH UNCLUDING DUODENUM C20 1521 Malignant neoplasm of rectosigmoid junction MALIGNANT NEOPLASM OF JUDIODENUM C20 1521 Malignant neoplasm of anal canal MALIGNANT NEOPLASM OF JUDIODENUM C210 1522 Malignant neoplasm of anal canal MALIGNANT NEOPLASM OF JUDIODENUM C211 1523 Malignant neoplasm of anal canal MALIGNANT NEOPLASM OF MECKEL'S DIV. C212 1528 Malignant neoplasm of doacogenic zone MALIGNANT NEOPLASM OF OTHER SPECIFICO OF SMALL INTESTINE C218 1529 Malignant neoplasm of doacogenic zone MALIGNANT NEOPLASM OF OTHER SPECIFICO OF SMALL INTESTINE C220 1531 Liver cell carcinoma MALIGNANT NEOPLASM OF OTHER SPECIFICO C221 1530 Intrahepatic bile duct carcinoma MALIGNANT NEOPLASM OF OTHER SPECIFICO C222 1531 Hepatoblastoma MALIGNANT NEOPLASM OF BEATLIC FLEXI C222 1531 Hapatoblastoma MALIGNANT NEOPLASM OF DESCENDING CI C224 1533 Other sarcomas of liver MALIGNANT NEOPLASM OF DESCENDING CI C224 1533 Other sarcomas of liver MALIGNANT NEOPLASM OF DESCENDING CI C227 1534 Other sarcomas of liver MALIGNANT NEOPLASM OF SIGMOID COLC C227 1534 Other sarcomas of liver MALIGNANT NEOPLASM OF ASCENDING CI C228 1535 Malignant neoplasm of liver, primary, unspecified as to type C249 1536 Malignant neoplasm of serahepatic bile duct MALIGNANT NEOPLASM OF ASCENDING CI C240 1538 Malignant neoplasm of primary of secondary MALIGNANT NEOPLASM OF ASCENDING CI C240 1538 Malignant neoplasm of primary of secondary C240 |
| C185 1515 Malignant neoplasm of splenic flexure MALIGNANT NEOPLASM OF LESSER CURVA STOMACH UNSPECIFIED C186 1516 Malignant neoplasm of descending colon MALIGNANT NEOPLASM OF GREATER CURVA STOMACH UNSPECIFIED C187 1518 Malignant neoplasm of sigmoid colon MALIGNANT NEOPLASM OF OTHER SPECIFIC OF STOMACH C188 1519 Malignant neoplasm of overlapping sites of colon MALIGNANT NEOPLASM OF STOMACH UNSPECIFIED C189 152 Malignant neoplasm of colon, unspecified MALIGNANT NEOPLASM OF SMALL INTEST INCLUDING DUODENUM C189 1520 Malignant neoplasm of rectosigmoid junction MALIGNANT NEOPLASM OF SMALL INTEST INCLUDING DUODENUM DEOPLASM OF SMALL INTEST INCLUDING DUODENUM MALIGNANT NEOPLASM OF JEJUNUM C20 1521 Malignant neoplasm of anus, unspecified MALIGNANT NEOPLASM OF JEJUNUM C210 1522 Malignant neoplasm of anus and sanal MALIGNANT NEOPLASM OF DIEUM C211 1523 Malignant neoplasm of anus inspecified MALIGNANT NEOPLASM OF MECKEL'S DIV. C212 1528 Malignant neoplasm of overlapping sites of rectum, MALIGNANT NEOPLASM OF OTHER SPECIFICATION OF SMALL INTEST INCLUDING MALIGNANT NEOPLASM OF OTHER SPECIFICATION OF SMALL INTEST INCLUDING MALIGNANT NEOPLASM OF OTHER SPECIFICATION OF SMALL INTEST INCLUDING MALIGNANT NEOPLASM OF OTHER SPECIFICATION OF SMALL INTEST INCLUDING MALIGNANT NEOPLASM OF OTHER SPECIFICATION OF SMALL INTEST INCLUDING MALIGNANT NEOPLASM OF MERCELLY MALIGNANT NEOPLASM OF DESCENDING (MALIGNANT NEOPLASM OF SMALL INTEST INCLUDING MALIGNANT NEOPLASM OF ASCENDING (MALIGNANT NEOPLASM OF ASCENDING (MALIGNANT NEOPLASM OF ASCENDING (MALIGNANT NEOPLASM OF ASCENDING (MALIGNANT NEOPLASM OF ASCENDING OF SECONDAY OF ANALIGNANT NEOPLASM OF OTHER SPECIFICATION OF ANALIGNANT NE |
| C186 1516 Malignant neoplasm of descending colon MALIGNANT NEOPLASM OF GREATER CURY STOMACH UNSPECIFIED C187 1518 Malignant neoplasm of sigmoid colon MALIGNANT NEOPLASM OF OTHER SPECIFIC OF STOMACH UNSPECIFIED C188 1519 Malignant neoplasm of overlapping sites of colon MALIGNANT NEOPLASM OF STOMACH UNSPECIFIC OF STOMACH C189 152 Malignant neoplasm of colon, unspecified MALIGNANT NEOPLASM OF SMALL INTEST INCLUDING DUODENUM C19 1520 Malignant neoplasm of rectosigmoid junction MALIGNANT NEOPLASM OF DUODENUM C20 1521 Malignant neoplasm of rectum MALIGNANT NEOPLASM OF DIJUNUM C210 1522 Malignant neoplasm of anus, unspecified MALIGNANT NEOPLASM OF JEJUNUM C211 1523 Malignant neoplasm of ania canal MALIGNANT NEOPLASM OF OTHER SPECIFIC OF SMALL INTESTINE C212 1528 Malignant neoplasm of doacogenic zone MALIGNANT NEOPLASM OF OTHER SPECIFIC OF SMALL INTESTINE C218 1529 Malignant neoplasm of overlapping sites of rectum, MALIGNANT NEOPLASM OF OTHER SPECIFIC OF SMALL INTESTINE C220 1531 Liver cell carcinoma MALIGNANT NEOPLASM OF SMALL INTEST ON SMALL INTEST O |
| C186 1516 Malignant neoplasm of descending colon MALIGNANT NEOPLASM OF GREATER CURN STOMACH UNSPECIFIED OF STOMACH |
| C187 1518 Malignant neoplasm of sigmoid colon MALIGNANT NEOPLASM OF OTHER SPECIFIC OF STOMACH UNSPECIFIED C188 1519 Malignant neoplasm of overlapping sites of colon MALIGNANT NEOPLASM OF STOMACH UNSPECIFIC OTHER SPECIFIC OF STOMACH UNSPECIFIC OTHER SPECIFIC OTHER SPECIF |
| C187 1518 Malignant neoplasm of sigmoid colon C189 1519 Malignant neoplasm of overlapping sites of colon C189 152 Malignant neoplasm of colon, unspecified C189 152 Malignant neoplasm of rectosigmoid junction C19 1520 Malignant neoplasm of rectosigmoid junction C20 1521 Malignant neoplasm of rectosigmoid junction C210 1522 Malignant neoplasm of rectosigmoid junction C210 1521 Malignant neoplasm of rectom C210 1522 Malignant neoplasm of rectom C210 1523 Malignant neoplasm of anus, unspecified C211 1523 Malignant neoplasm of anus, unspecified C212 1528 Malignant neoplasm of colon C212 1528 Malignant neoplasm of color of overlapping sites of rectum, C218 1529 Malignant neoplasm of overlapping sites of rectum, C219 Malignant neoplasm of overlapping sites of rectum, C210 1531 Liver cell carcinoma C220 1531 Liver cell carcinoma C221 1530 Intrahepatic bile duct carcinoma C222 1531 Hepatoblastoma C223 1532 Angiosarcoma of liver C224 1533 Other sarcomas of liver C226 1534 Other sarcomas of liver C227 1534 Other sarcomas of liver C228 1535 Malignant neoplasm of liver, primary, unspecified as to type C229 1536 Malignant neoplasm of liver, primary, unspecified as to MALIGNANT NEOPLASM OF ASCENDING of Secondary C23 1537 Malignant neoplasm of servanhepatic bile duct C24 1538 Malignant neoplasm of servanhepatic bile duct MALIGNANT NEOPLASM OF SECENDING of Secondary C24 1539 Malignant neoplasm of liver, primary, unspecified as to MALIGNANT NEOPLASM OF ASCENDING of Secondary C24 1539 Malignant neoplasm of servanhepatic bile duct MALIGNANT NEOPLASM OF ASCENDING of Secondary C24 1539 Malignant neoplasm of overlapping sites of biliary tract MALIGNANT NEOPLASM OF ASCENDING of Secondary C24 Malignant neoplasm of overlapping sites of biliary tract MALIGNANT NEOPLASM OF ASCENDING of Secondary C24 Malignant neoplasm of overlapping sites of biliary tract MALIGNANT NEOPLASM OF ASCENDING of Secondary C25 1540 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL MALIGNANT NEOPLASM OF |
| C188 1519 Malignant neoplasm of overlapping sites of colon MALIGNANT NEOPLASM OF STOMACH UNITED TO STO |
| C188 1519 Malignant neoplasm of overlapping sites of colon MALIGNANT NEOPLASM OF STOMACH UNITED TO THE STOMACH UNITED THE STOMACH UNITED TO THE STOMACH UNITED TO THE STOMACH UNITED THE STOMACH UNITED TO THE STOMACH UNITED TO THE STOMACH UNITED TO THE STOMACH UNITED TO THE STOMACH UNITED TO THE STOMACH UNITED THE STOMACH UNITED TO THE STOMACH UNITED TO THE STOMACH UNITED THE STOMACH UNITED TO THE STOMACH UNITED TO THE STOMACH UNITED THE STOMACH UNITED TO THE STOMACH UNITED TO THE STOMACH UNITED TO THE STOMACH UNITED TO THE STOMACH UNITED TO THE STOMACH UNITED THE STOMACH UNITED TO THE STOMACH UNITED TO THE STOMACH UNITED THE STOMACH UNITED TO THE STOMAC |
| C189 152 Malignant neoplasm of colon, unspecified MALIGNANT NEOPLASM OF SMALL INTEST INCLUDING DUODENUM C19 1520 Malignant neoplasm of rectosigmoid junction MALIGNANT NEOPLASM OF DUODENUM C20 1521 Malignant neoplasm of rectum MALIGNANT NEOPLASM OF JEJUNUM C210 1522 Malignant neoplasm of anus, unspecified MALIGNANT NEOPLASM OF ILEUM C211 1523 Malignant neoplasm of anal canal MALIGNANT NEOPLASM OF MECKEL'S DIV. C212 1528 Malignant neoplasm of doacogenic zone MALIGNANT NEOPLASM OF OTHER SPECIFIC OF SMALL INTESTINE C218 1529 Malignant neoplasm of overlapping sites of rectum, anus and anal canal UNSPECIFIED SITE C220 153 Liver cell carcinoma MALIGNANT NEOPLASM OF SMALL INTEST C221 1530 Intrahepatic bile duct carcinoma MALIGNANT NEOPLASM OF HEPATIC FLEXI C222 1531 Hepatoblastoma MALIGNANT NEOPLASM OF TRANSVERSE (C223 1532 Angiosarcoma of liver MALIGNANT NEOPLASM OF DESCENDING (C224 1533) Other sarcomas of liver MALIGNANT NEOPLASM OF DESCENDING (C227 1534 Other specified carcinomas of liver MALIGNANT NEOPLASM OF CECUM MALIGNANT NEOPLASM OF APPENDIX VER (C228 1535 Malignant neoplasm of liver, primary, unspecified as to type C229 1536 Malignant neoplasm of liver, not specified as primary or secondary C23 1537 Malignant neoplasm of gallbladder MALIGNANT NEOPLASM OF ASCENDING (C229 1538 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF OTHER SPECIFIC PLEXIC MALIGNANT NEOPLASM OF OTHER SPECIFIC PLEXIC MALIGNANT NEOPLASM OF OTHER SPECIFIC PLEXIC MALIGNANT NEOPLASM OF OTHER SPECIFIC PLEXIC MALIGNANT NEOPLASM OF RECTUM RECTUDING AND ANUS C249 1540 Malignant neoplasm of biliary tract, unspecified MALIGNANT NEOPLASM OF RECTUM RECTUDING AND ANUS C249 1540 Malignant neoplasm of biliary tract, unspecified MALIGNANT NEOPLASM OF RECTUM RECTUDING AND ANUS C250 1541 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF RECTOSIGMOIC C250 1543 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANUS UNSPECED C250 1543 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANUS UNSPECE |
| C19 1520 Malignant neoplasm of rectosigmoid junction MALIGNANT NEOPLASM OF DUODENUM C20 1521 Malignant neoplasm of rectum MALIGNANT NEOPLASM OF JEJUNUM C210 1522 Malignant neoplasm of anus, unspecified MALIGNANT NEOPLASM OF JEJUNUM C211 1523 Malignant neoplasm of anal canal MALIGNANT NEOPLASM OF ILEUM C212 1528 Malignant neoplasm of cloacogenic zone MALIGNANT NEOPLASM OF OTHER SPECIFIOF OF SMALL INTESTINE C218 1529 Malignant neoplasm of overlapping sites of rectum, MALIGNANT NEOPLASM OF SMALL INTEST C220 153 Liver cell carcinoma MALIGNANT NEOPLASM OF SMALL INTEST C220 1530 Intrahepatic bile duct carcinoma MALIGNANT NEOPLASM OF COLON C221 1530 Intrahepatic bile duct carcinoma MALIGNANT NEOPLASM OF HEPATIC FLEXI C222 1531 Hepatoblastoma MALIGNANT NEOPLASM OF TRANSVERSE (C223 1532 Angiosarcoma of liver MALIGNANT NEOPLASM OF DESCENDING (C224 1533 Other sarcomas of liver MALIGNANT NEOPLASM OF DESCENDING (C227 1534 Other specified carcinomas of liver MALIGNANT NEOPLASM OF DESCENDING (C227 1534 Other specified carcinomas of liver MALIGNANT NEOPLASM OF ASCENDING (C228 1535 Malignant neoplasm of liver, primary, unspecified as to type C229 1536 Malignant neoplasm of liver, not specified as primary or secondary C23 1537 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF ASCENDING (C224 1538 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF OTHER SPECIFICAL MALIGNANT NEOPLASM OF RECTUM RELIGIORANT NEOPLASM OF RECTUM RECTUM RELIGIORANT NEOPLASM OF RECTUM RE |
| C19 1520 Malignant neoplasm of rectosigmoid junction MALIGNANT NEOPLASM OF DUODENUM C20 1521 Malignant neoplasm of rectum MALIGNANT NEOPLASM OF JEJUNUM C210 1522 Malignant neoplasm of anal, unspecified MALIGNANT NEOPLASM OF ILEUM C211 1523 Malignant neoplasm of anal canal MALIGNANT NEOPLASM OF MECKEL'S DIV. C212 1528 Malignant neoplasm of cloacogenic zone MALIGNANT NEOPLASM OF MECKEL'S DIV. C212 1528 Malignant neoplasm of overlapping sites of rectum, anus and anal canal C218 1529 Malignant neoplasm of overlapping sites of rectum, anus and anal canal MALIGNANT NEOPLASM OF SMALL INTEST C220 153 Liver cell carcinoma MALIGNANT NEOPLASM OF COLON C221 1530 Intrahepatic bile duct carcinoma MALIGNANT NEOPLASM OF HEPATIC FLEXI C222 1531 Hepatoblastoma MALIGNANT NEOPLASM OF TRANSVERSE ( C223 1532 Angiosarcoma of liver MALIGNANT NEOPLASM OF DESCENDING ( C224 1533 Other sarcomas of liver MALIGNANT NEOPLASM OF SIGMOID COLC C227 1534 Other sarcomas of liver MALIGNANT NEOPLASM OF CECUM C228 1535 Malignant neoplasm of liver, primary, unspecified as to type C229 1536 Malignant neoplasm of liver, not specified as primary or secondary C23 1537 Malignant neoplasm of gallbladder MALIGNANT NEOPLASM OF SPLENIC FLEXU MALIGNANT NEOPLASM OF APPENDIX VER C240 1538 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF SPLENIC FLEXU MALIGNANT NEOPLASM OF APPENDIX VER C241 1539 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF RECTUM RECT DIARGE INTESTINE C241 1539 Malignant neoplasm of overlapping sites of biliary tract MALIGNANT NEOPLASM OF RECTUM RECT JUNCTION AND ANUS C249 1540 Malignant neoplasm of head of pancreas MALIGNANT NEOPLASM OF RECTUM RECT JUNCTION AND ANUS C250 1541 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C251 1543 Malignant neoplasm of fooly of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of fooly of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of fooly of pancreas |
| C20 1521 Malignant neoplasm of rectum MALIGNANT NEOPLASM OF JEJUNUM C210 1522 Malignant neoplasm of anus, unspecified MALIGNANT NEOPLASM OF ILEUM C211 1523 Malignant neoplasm of anal canal MALIGNANT NEOPLASM OF MECKEL'S DIVI C212 1528 Malignant neoplasm of cloacogenic zone MALIGNANT NEOPLASM OF OTHER SPECIFI C218 1529 Malignant neoplasm of overlapping sites of rectum, |
| C210 1522 Malignant neoplasm of anus, unspecified MALIGNANT NEOPLASM OF ILEUM C211 1523 Malignant neoplasm of anal canal MALIGNANT NEOPLASM OF MECKEL'S DIVI C212 1528 Malignant neoplasm of cloacogenic zone MALIGNANT NEOPLASM OF OTHER SPECIF OF SMALL INTESTINE C218 1529 Malignant neoplasm of overlapping sites of rectum, MALIGNANT NEOPLASM OF SMALL INTEST anus and anal canal MALIGNANT NEOPLASM OF SMALL INTEST UNSPECIFIED SITE C220 1531 Liver cell carcinoma MALIGNANT NEOPLASM OF COLON C221 1530 Intrahepatic bile duct carcinoma MALIGNANT NEOPLASM OF HEPATIC FLEXI C222 1531 Hepatoblastoma MALIGNANT NEOPLASM OF TRANSVERSE C C223 1532 Angiosarcoma of liver MALIGNANT NEOPLASM OF DESCENDING C C224 1533 Other sarcomas of liver MALIGNANT NEOPLASM OF DESCENDING C C227 1534 Other specified carcinomas of liver MALIGNANT NEOPLASM OF CECUM C228 1535 Malignant neoplasm of liver, primary, unspecified as to type C229 1536 Malignant neoplasm of liver, not specified as primary or secondary C23 1537 Malignant neoplasm of gallbladder MALIGNANT NEOPLASM OF ASCENDING C C240 1538 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF OTHER SPECIF OF LARGE INTESTINE C241 1539 Malignant neoplasm of overlapping sites of biliary tract MALIGNANT NEOPLASM OF OTHER SPECIF OF LARGE INTESTINE C248 1540 Malignant neoplasm of overlapping sites of biliary tract JUNCTION AND ANUS C249 1540 Malignant neoplasm of head of pancreas MALIGNANT NEOPLASM OF RECTUM RECTUME C250 1541 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of body of pancreas |
| C211 1523 Malignant neoplasm of anal canal MALIGNANT NEOPLASM OF MECKEL'S DIVI C212 1528 Malignant neoplasm of cloacogenic zone MALIGNANT NEOPLASM OF OTHER SPECIFIOF SMALL INTESTINE C218 1529 Malignant neoplasm of overlapping sites of rectum, anus and anal canal UNSPECIFIED SITE C220 1531 Liver cell carcinoma MALIGNANT NEOPLASM OF SMALL INTEST UNSPECIFIED SITE C221 1530 Intrahepatic bile duct carcinoma MALIGNANT NEOPLASM OF COLON C221 1531 Hepatoblastoma MALIGNANT NEOPLASM OF HEPATIC FLEXI C222 1531 Hepatoblastoma MALIGNANT NEOPLASM OF DESCENDING OF C224 1533 Other sarcomas of liver MALIGNANT NEOPLASM OF DESCENDING OF C224 1534 Other specified carcinomas of liver MALIGNANT NEOPLASM OF SIGMOID COLO C227 1534 Other specified carcinomas of liver MALIGNANT NEOPLASM OF APPENDIX VER C229 1536 Malignant neoplasm of liver, not specified as to MALIGNANT NEOPLASM OF APPENDIX VER C229 1536 Malignant neoplasm of liver, not specified as primary or MALIGNANT NEOPLASM OF APPENDIX VER C229 1536 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF SPLENIC FLEXU C240 1538 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF OTHER SPECIFICAL C241 1539 Malignant neoplasm of overlapping sites of biliary tract MALIGNANT NEOPLASM OF COLON UNSPECTIVE C248 1540 Malignant neoplasm of overlapping sites of biliary tract MALIGNANT NEOPLASM OF RECTUM RECTUM C249 1541 Malignant neoplasm of head of pancreas MALIGNANT NEOPLASM OF RECTUM RECTUM C250 1541 Malignant neoplasm of head of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C251 1542 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of bad of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 |
| C212 1528 Malignant neoplasm of cloacogenic zone MALIGNANT NEOPLASM OF OTHER SPECIFIC OF SMALL INTESTINE C218 1529 Malignant neoplasm of overlapping sites of rectum, MALIGNANT NEOPLASM OF SMALL INTEST anus and anal canal UNSPECIFIED SITE C220 1531 Liver cell carcinoma MALIGNANT NEOPLASM OF COLON C221 1530 Intrahepatic bile duct carcinoma MALIGNANT NEOPLASM OF HEPATIC FLEXI C222 1531 Hepatoblastoma MALIGNANT NEOPLASM OF TRANSVERSE (C223 1532 Angiosarcoma of liver MALIGNANT NEOPLASM OF DESCENDING (C224 1533 Other sarcomas of liver MALIGNANT NEOPLASM OF SIGMOID COLO (C227 1534 Other specified carcinomas of liver MALIGNANT NEOPLASM OF APPENDIX VER (C228 1535 Malignant neoplasm of liver, primary, unspecified as to MALIGNANT NEOPLASM OF APPENDIX VER (C229 1536 Malignant neoplasm of liver, not specified as primary or Secondary MALIGNANT NEOPLASM OF ASCENDING (C230 1537 Malignant neoplasm of secondary MALIGNANT NEOPLASM OF ASCENDING (C230 1538 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF OTHER SPECIFIC FLEXU (C240 1538 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF COLON UNSPECIFICATION (C248 1540 Malignant neoplasm of overlapping sites of biliary tract (C249 1540 Malignant neoplasm of biliary tract, unspecified (C249 1540 Malignant neoplasm of biliary tract, unspecified (C250 1541 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL (C252 1543 Malignant neoplasm of tail of pancreas MALIGNANT NEOPLASM OF ANAL CANAL (C252 1543 Malignant neoplasm of tail of pancreas MALIGNANT NEOPLASM OF ANAL CANAL (C252 1543 Malignant neoplasm of tail of pancreas MALIGNANT NEOPLASM OF ANUS UNSPEC |
| C218 1529 Malignant neoplasm of overlapping sites of rectum, anus and anal canal UNSPECIFIED SITE C220 153 Liver cell carcinoma MALIGNANT NEOPLASM OF COLON C221 1530 Intrahepatic bile duct carcinoma MALIGNANT NEOPLASM OF HEPATIC FLEXI C222 1531 Hepatoblastoma MALIGNANT NEOPLASM OF TRANSVERSE C C223 1532 Angiosarcoma of liver MALIGNANT NEOPLASM OF FRANSVERSE C C224 1533 Other sarcomas of liver MALIGNANT NEOPLASM OF DESCENDING C C224 1534 Other specified carcinomas of liver MALIGNANT NEOPLASM OF SIGMOID COLC C227 1534 Other specified carcinomas of liver MALIGNANT NEOPLASM OF CECUM C228 1535 Malignant neoplasm of liver, primary, unspecified as to type C229 1536 Malignant neoplasm of liver, not specified as primary or MALIGNANT NEOPLASM OF APPENDIX VER type C229 1536 Malignant neoplasm of gallbladder MALIGNANT NEOPLASM OF SPLENIC FLEXU C240 1538 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF OTHER SPECIFIC OF LARGE INTESTINE C241 1539 Malignant neoplasm of ampulla of Vater MALIGNANT NEOPLASM OF COLON UNSPECIFICATION OF ADAMS C249 1540 Malignant neoplasm of overlapping sites of biliary tract MALIGNANT NEOPLASM OF RECTUM RECTUM C250 1541 Malignant neoplasm of head of pancreas MALIGNANT NEOPLASM OF RECTUM C251 1542 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of tail of pancreas MALIGNAN |
| C220 153 Liver cell carcinoma MALIGNANT NEOPLASM OF SMALL INTEST C220 153 Liver cell carcinoma MALIGNANT NEOPLASM OF COLON C221 1530 Intrahepatic bile duct carcinoma MALIGNANT NEOPLASM OF HEPATIC FLEXI C222 1531 Hepatoblastoma MALIGNANT NEOPLASM OF TRANSVERSE ( C223 1532 Angiosarcoma of liver MALIGNANT NEOPLASM OF DESCENDING ( C224 1533 Other sarcomas of liver MALIGNANT NEOPLASM OF SIGMOID COLO C227 1534 Other specified carcinomas of liver MALIGNANT NEOPLASM OF SIGMOID COLO C228 1535 Malignant neoplasm of liver, primary, unspecified as to type C229 1536 Malignant neoplasm of liver, not specified as primary or secondary C23 1537 Malignant neoplasm of gallbladder MALIGNANT NEOPLASM OF ASCENDING ( C240 1538 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF OTHER SPECIFIC FLEXU C241 1539 Malignant neoplasm of ampulla of Vater MALIGNANT NEOPLASM OF COLON UNSPECIFICATION OF ADJUST O |
| anus and anal canal C220 153 Liver cell carcinoma MALIGNANT NEOPLASM OF COLON C221 1530 Intrahepatic bile duct carcinoma MALIGNANT NEOPLASM OF HEPATIC FLEXU C222 1531 Hepatoblastoma MALIGNANT NEOPLASM OF TRANSVERSE OF C223 1532 Angiosarcoma of liver MALIGNANT NEOPLASM OF DESCENDING OF C224 1533 Other sarcomas of liver MALIGNANT NEOPLASM OF SIGMOID COLOR C224 1533 Other sarcomas of liver MALIGNANT NEOPLASM OF SIGMOID COLOR C227 1534 Other specified carcinomas of liver MALIGNANT NEOPLASM OF CECUM C228 1535 Malignant neoplasm of liver, primary, unspecified as to type C229 1536 Malignant neoplasm of liver, not specified as primary or secondary C23 1537 Malignant neoplasm of gallbladder MALIGNANT NEOPLASM OF ASCENDING OF SECONDARY C240 1538 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF OTHER SPECIFIC OF LARGE INTESTINE C241 1539 Malignant neoplasm of overlapping sites of biliary tract MALIGNANT NEOPLASM OF RECTUM RECTUM C248 154 Malignant neoplasm of biliary tract, unspecified MALIGNANT NEOPLASM OF RECTUM RECTUM C250 1541 Malignant neoplasm of head of pancreas MALIGNANT NEOPLASM OF RECTUM OF ANAL CANAL C252 1543 Malignant neoplasm of tail of pancreas MALIGNANT NEOPLASM OF ANAL CANA |
| C220 1530 Liver cell carcinoma MALIGNANT NEOPLASM OF COLON C221 1530 Intrahepatic bile duct carcinoma MALIGNANT NEOPLASM OF HEPATIC FLEXI C222 1531 Hepatoblastoma MALIGNANT NEOPLASM OF TRANSVERSE (C223 1532 Angiosarcoma of liver MALIGNANT NEOPLASM OF DESCENDING (C224 1533 Other sarcomas of liver MALIGNANT NEOPLASM OF SIGMOID COLO C227 1534 Other specified carcinomas of liver MALIGNANT NEOPLASM OF CECUM C228 1535 Malignant neoplasm of liver, primary, unspecified as to type C229 1536 Malignant neoplasm of liver, not specified as primary or secondary C23 1537 Malignant neoplasm of gallbladder MALIGNANT NEOPLASM OF ASCENDING CO240 1538 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF OTHER SPECIFIC OF LARGE INTESTINE C241 1539 Malignant neoplasm of ampulla of Vater MALIGNANT NEOPLASM OF COLON UNSPECIFICATION AND ANUS C249 1540 Malignant neoplasm of biliary tract, unspecified MALIGNANT NEOPLASM OF RECTUM RECTURN MALIGNANT NEOPLASM OF RECTURN OF RECTURN MALIGNANT NEOPLASM OF RECTURN OF RECTURN MALIGNANT NEOPLASM OF RECTURN OF RECTURN MALIGNANT NEOPLASM OF RECTURN OF RECTURN MALIGNANT NEOPLASM OF RECTURN OF RECTURN OF RECTURN MALIGNANT NEOPLASM OF RECTURN OF RECTURN OF RECTURN OF ANALIGNANT NEOPLASM OF ANALIGNANT NEOPL |
| C221 1530 Intrahepatic bile duct carcinoma MALIGNANT NEOPLASM OF HEPATIC FLEXI C222 1531 Hepatoblastoma MALIGNANT NEOPLASM OF TRANSVERSE ( C223 1532 Angiosarcoma of liver MALIGNANT NEOPLASM OF DESCENDING ( C224 1533 Other sarcomas of liver MALIGNANT NEOPLASM OF DESCENDING ( C227 1534 Other specified carcinomas of liver MALIGNANT NEOPLASM OF CECUM C228 1535 Malignant neoplasm of liver, primary, unspecified as to type C229 1536 Malignant neoplasm of liver, not specified as primary or secondary C23 1537 Malignant neoplasm of gallbladder MALIGNANT NEOPLASM OF ASCENDING CO secondary C240 1538 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF OTHER SPECIFICATION OF LARGE INTESTINE C241 1539 Malignant neoplasm of ampulla of Vater MALIGNANT NEOPLASM OF COLON UNSPECIFICATION AND ANUS C249 1540 Malignant neoplasm of biliary tract, unspecified MALIGNANT NEOPLASM OF RECTUM RECTUM C250 1541 Malignant neoplasm of head of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of tail of pancreas MALIGNANT NEOPLASM OF ANAL C |
| C222 1531 Hepatoblastoma MALIGNANT NEOPLASM OF TRANSVERSE (C223 1532 Angiosarcoma of liver MALIGNANT NEOPLASM OF DESCENDING (C224 1533 Other sarcomas of liver MALIGNANT NEOPLASM OF SIGMOID COLC (C227 1534 Other specified carcinomas of liver MALIGNANT NEOPLASM OF CECUM (C228 1535 Malignant neoplasm of liver, primary, unspecified as to type (C229 1536 Malignant neoplasm of liver, not specified as primary or secondary (C23 1537 Malignant neoplasm of gallbladder MALIGNANT NEOPLASM OF ASCENDING CO (C240 1538 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF OTHER SPECIFIC (C241 1539 Malignant neoplasm of ampulla of Vater MALIGNANT NEOPLASM OF COLON UNSPECIFIC (C248 1540 Malignant neoplasm of overlapping sites of biliary tract (MALIGNANT NEOPLASM OF RECTUM RECTUM (C250 1541 Malignant neoplasm of head of pancreas MALIGNANT NEOPLASM OF RECTUM (C251 1542 Malignant neoplasm of body of pancreas (MALIGNANT NEOPLASM OF ANAL CANAL (C252 1543 Malignant neoplasm of tail of pancreas (MALIGNANT NEOPLASM OF ANAL CANAL (C252 1543 MALIGNANT NEOPLASM OF ANAL (C252 1543 MALIGNANT NEOPLASM OF ANAL (C |
| C223 1532 Angiosarcoma of liver MALIGNANT NEOPLASM OF DESCENDING OF C224 1533 Other sarcomas of liver MALIGNANT NEOPLASM OF SIGMOID COLOR C227 1534 Other specified carcinomas of liver MALIGNANT NEOPLASM OF CECUM C228 1535 Malignant neoplasm of liver, primary, unspecified as to type MALIGNANT NEOPLASM OF APPENDIX VER C229 1536 Malignant neoplasm of liver, not specified as primary or secondary MALIGNANT NEOPLASM OF ASCENDING OF SECONDARY MALIGNANT NEOPLASM OF ASCENDING OF C23 1537 Malignant neoplasm of gallbladder MALIGNANT NEOPLASM OF SPLENIC FLEXU MALIGNANT NEOPLASM OF OTHER SPECIFIC OF LARGE INTESTINE C241 1539 Malignant neoplasm of ampulla of Vater MALIGNANT NEOPLASM OF COLON UNSPECIFIC C248 154 Malignant neoplasm of overlapping sites of biliary tract MALIGNANT NEOPLASM OF RECTUM RECTUM C250 1541 Malignant neoplasm of head of pancreas MALIGNANT NEOPLASM OF RECTUM MALIGNANT NEOPLASM OF ANAL CANAL MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of tail of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 MA |
| C224 1533 Other sarcomas of liver MALIGNANT NEOPLASM OF SIGMOID COLOR C227 1534 Other specified carcinomas of liver MALIGNANT NEOPLASM OF CECUM C228 1535 Malignant neoplasm of liver, primary, unspecified as to type C229 1536 Malignant neoplasm of liver, not specified as primary or secondary C23 1537 Malignant neoplasm of gallbladder MALIGNANT NEOPLASM OF ASCENDING CO C240 1538 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF OTHER SPECIFI OF LARGE INTESTINE C241 1539 Malignant neoplasm of ampulla of Vater MALIGNANT NEOPLASM OF COLON UNSPECIAL MALIGNANT NEOPLASM OF RECTUM RECTUMING COLOR MALIGNANT NEOPLASM OF RECTUM RECTUMING COLOR MALIGNANT NEOPLASM OF ANAL CANAL COLOR MALIGNANT NEOPLASM OF ANAL CANAL COLO |
| C227 1534 Other specified carcinomas of liver MALIGNANT NEOPLASM OF CECUM C228 1535 Malignant neoplasm of liver, primary, unspecified as to type C229 1536 Malignant neoplasm of liver, not specified as primary or secondary C23 1537 Malignant neoplasm of gallbladder MALIGNANT NEOPLASM OF ASCENDING CO secondary C240 1538 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF OTHER SPECIFIC OF LARGE INTESTINE C241 1539 Malignant neoplasm of ampulla of Vater MALIGNANT NEOPLASM OF COLON UNSPECIFICATION AND ANUS C249 1540 Malignant neoplasm of overlapping sites of biliary tract MALIGNANT NEOPLASM OF RECTUM RECTURED MALIGNANT NEOPLASM OF RECTUM RECTURED MALIGNANT NEOPLASM OF RECTUM RECTURED MALIGNANT NEOPLASM OF ANAL CANAL CANAL MALIGNANT NEOPLASM OF ANAL CANAL CANAL CASCER MALIGNANT NEOPLASM OF ANAL CASCER MALIGNANT NEOPLASM OF ANAL |
| C228 1535 Malignant neoplasm of liver, primary, unspecified as to type C229 1536 Malignant neoplasm of liver, not specified as primary or secondary C23 1537 Malignant neoplasm of gallbladder MALIGNANT NEOPLASM OF ASCENDING CCCCCCCCCCCCCCCCCCCCCCCCCCCCCCCCCCCC |
| type C229 1536 Malignant neoplasm of liver, not specified as primary or secondary C23 1537 Malignant neoplasm of gallbladder MALIGNANT NEOPLASM OF SPLENIC FLEXU C240 1538 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF OTHER SPECIFIC OF LARGE INTESTINE C241 1539 Malignant neoplasm of ampulla of Vater MALIGNANT NEOPLASM OF COLON UNSPECTABLE OF LARGE INTESTINE C248 154 Malignant neoplasm of overlapping sites of biliary tract MALIGNANT NEOPLASM OF RECTUM RECTUM SECTION AND ANUS C249 1540 Malignant neoplasm of biliary tract, unspecified MALIGNANT NEOPLASM OF RECTUM MALIGNANT NEOPLASM OF ANAL CANAL C251 1542 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of tail of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of tail of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of tail of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of tail of pancreas MALIGNANT NEOPLASM OF ANUS UNSPEC |
| secondary C23 1537 Malignant neoplasm of gallbladder MALIGNANT NEOPLASM OF SPLENIC FLEXU C240 1538 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF OTHER SPECIFION OF LARGE INTESTINE C241 1539 Malignant neoplasm of ampulla of Vater MALIGNANT NEOPLASM OF COLON UNSPECTABLE OF LARGE INTESTINE C248 154 Malignant neoplasm of overlapping sites of biliary tract MALIGNANT NEOPLASM OF RECTUM RECTUM SECTION OF COLON UNSPECTABLE OF LARGE INTESTINE C249 1540 Malignant neoplasm of biliary tract, unspecified MALIGNANT NEOPLASM OF RECTOSIGMON C250 1541 Malignant neoplasm of head of pancreas MALIGNANT NEOPLASM OF RECTUM C251 1542 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of tail of pancreas MALIGNANT NEOPLASM OF ANUS UNSPECTABLE O |
| C240 1538 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF OTHER SPECIFICATION OF LARGE INTESTINE C241 1539 Malignant neoplasm of ampulla of Vater MALIGNANT NEOPLASM OF COLON UNSPECT MALIGNANT NEOPLASM OF RECTUM RECTUM RECTUM NEOPLASM OF RECTUM RECTUM NEOPLASM OF RECTUM RECTUM NEOPLASM OF ANAL CANAL NEOPLASM OF ANAL NEOPLASM OF ANAL CANAL NEOPLASM OF ANAL CANAL NEOPLASM OF ANAL CANAL NEOPLASM OF ANAL CANAL NEOPLASM OF ANAL CANAL NEOPLASM OF ANAL NEOPLASM OF ANAL CANAL NEOPLASM OF ANAL CANAL NEOPLASM OF ANA |
| C240 1538 Malignant neoplasm of extrahepatic bile duct MALIGNANT NEOPLASM OF OTHER SPECIFICATION OF LARGE INTESTINE C241 1539 Malignant neoplasm of ampulla of Vater MALIGNANT NEOPLASM OF COLON UNSPECT MALIGNANT NEOPLASM OF RECTUM RECTUM RECTUM NEOPLASM OF RECTUM RECTUM NEOPLASM OF RECTUM RECTUM NEOPLASM OF ANAL CANAL NEOPLASM OF ANAL NEOPLASM OF ANAL CANAL NEOPLASM OF ANAL CANAL NEOPLASM OF ANAL CANAL NEOPLASM OF ANAL CANAL NEOPLASM OF ANAL CANAL NEOPLASM OF ANAL NEOPLASM OF ANAL CANAL NEOPLASM OF ANAL CANAL NEOPLASM OF ANA |
| C241 1539 Malignant neoplasm of ampulla of Vater MALIGNANT NEOPLASM OF COLON UNSPECTOR C248 154 Malignant neoplasm of overlapping sites of biliary tract MALIGNANT NEOPLASM OF RECTUM RECTURNATION AND ANUS MALIGNANT NEOPLASM OF RECTOSIGMOIN C250 1541 Malignant neoplasm of biliary tract, unspecified MALIGNANT NEOPLASM OF RECTOSIGMOIN C251 1542 Malignant neoplasm of head of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of tail of pancreas MALIGNANT NEOPLASM OF ANUS UNSPECTOR C252 1543 MALIGNANT NEOPLASM OF ANUS UNSPECTOR C252 1544 MA |
| C241 1539 Malignant neoplasm of ampulla of Vater MALIGNANT NEOPLASM OF COLON UNSPECTOR C248 154 Malignant neoplasm of overlapping sites of biliary tract MALIGNANT NEOPLASM OF RECTUM RECTURNATION AND ANUS MALIGNANT NEOPLASM OF RECTOSIGMOIN C250 1541 Malignant neoplasm of biliary tract, unspecified MALIGNANT NEOPLASM OF RECTOSIGMOIN C251 1542 Malignant neoplasm of head of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of tail of pancreas MALIGNANT NEOPLASM OF ANUS UNSPECTOR C252 1543 MALIGNANT NEOPLASM OF ANUS UNSPECTOR C252 1544 MA |
| C248 154 Malignant neoplasm of overlapping sites of biliary tract MALIGNANT NEOPLASM OF RECTUM RECTURENT JUNCTION AND ANUS C249 1540 Malignant neoplasm of biliary tract, unspecified MALIGNANT NEOPLASM OF RECTOSIGMON C250 1541 Malignant neoplasm of head of pancreas MALIGNANT NEOPLASM OF RECTUM C251 1542 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of tail of pancreas MALIGNANT NEOPLASM OF ANUS UNSPEC |
| JUNCTION AND ANUS C249 1540 Malignant neoplasm of biliary tract, unspecified MALIGNANT NEOPLASM OF RECTOSIGMON C250 1541 Malignant neoplasm of head of pancreas MALIGNANT NEOPLASM OF RECTUM C251 1542 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of tail of pancreas MALIGNANT NEOPLASM OF ANUS UNSPEC |
| C249 1540 Malignant neoplasm of biliary tract, unspecified MALIGNANT NEOPLASM OF RECTOSIGMON C250 1541 Malignant neoplasm of head of pancreas MALIGNANT NEOPLASM OF RECTUM C251 1542 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of tail of pancreas MALIGNANT NEOPLASM OF ANUS UNSPECTION |
| C250 1541 Malignant neoplasm of head of pancreas MALIGNANT NEOPLASM OF RECTUM C251 1542 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of tail of pancreas MALIGNANT NEOPLASM OF ANUS UNSPEC |
| C251 1542 Malignant neoplasm of body of pancreas MALIGNANT NEOPLASM OF ANAL CANAL C252 1543 Malignant neoplasm of tail of pancreas MALIGNANT NEOPLASM OF ANUS UNSPEC |
| C252 1543 Malignant neoplasm of tail of pancreas MALIGNANT NEOPLASM OF ANUS UNSPEC |
| 1 25 to Manghant neophasti of patient additional patients and the patients are patients and the patients are patients and the patients and the patients and the patients are patients and the patients are patients and the patients are patients and the patients and the patients are patients and the pat |
| RECTOSIGMOID JUNCTION AND ANUS |
| C254 155 Malignant neoplasm of endocrine pancreas MALIGNANT NEOPLASM OF LIVER AND INT |
| BILE DUCTS |
| C257 1550 Malignant neoplasm of other parts of pancreas MALIGNANT NEOPLASM OF LIVER PRIMAR |
| C258 1551 Malignant neoplasm of overlapping sites of pancreas MALIGNANT NEOPLASM OF INTRAHEPATIC |
| I (CIED I 1EE) I Malignant noonlosm of nangrood upgranifical I MALICNIANT NEODIACA OF UVERNOT OR |
| C259 1552 Malignant neoplasm of pancreas, unspecified MALIGNANT NEOPLASM OF LIVER NOT SPE |
| PRIMARY OR SECONDARY |
| C260 156 Malignant neoplasm of intestinal tract, part unspecified MALIGNANT NEOPLASM OF GALLBLADDER |
| PRIMARY OR SECONDARY |


| C9001 2398 Multiple myeloma in remission SPECIFIED SITES GLANDS AND OTHER PAR NEOPLASMS OF UNSPEC SPECIFIED SITES | |
|---|---|
| C9000 2397 Multiple myeloma not having achieved remission NEOPLASM OF UNSPECIF GLANDS AND OTHER PAR C9001 2398 Multiple myeloma in remission NEOPLASMS OF UNSPECIF SPECIFIED SITES C9002 23981 Multiple myeloma in relapse NEOPLASM OF UNSPECIF CHOROID C9010 23989 Plasma cell leukemia not having achieved remission NEOPLASM OF UNSPECIF SPECIFIED SITES | FIED NATURE OF ENDOCRINE<br>RTS OF NERVOUS SYSTEM |
| C9001 2398 Multiple myeloma in remission NEOPLASMS OF UNSPECT SPECIFIED SITES C9002 23981 Multiple myeloma in relapse NEOPLASM OF UNSPECT CHOROID C9010 23989 Plasma cell leukemia not having achieved remission NEOPLASM OF UNSPECT SPECIFIED SITES | |
| C9002 23981 Multiple myeloma in relapse NEOPLASM OF UNSPECIF CHOROID C9010 23989 Plasma cell leukemia not having achieved remission NEOPLASM OF UNSPECIF SPECIFIED SITES | IFIED NATURE OF OTHER |
| C9002 23981 Multiple myeloma in relapse NEOPLASM OF UNSPECIF CHOROID C9010 23989 Plasma cell leukemia not having achieved remission NEOPLASM OF UNSPECIF SPECIFIED SITES | |
| CHOROID C9010 23989 Plasma cell leukemia not having achieved remission NEOPLASM OF UNSPECIFIED SITES | |
| C9010 23989 Plasma cell leukemia not having achieved remission NEOPLASM OF UNSPECIFIED SITES | FIED NATURE OF RETINA AND |
| SPECIFIED SITES | |
| | FIED NATURE OF OTHER |
| C9011 2399 Plasma cell leukemia in remission NEOPLASM OF UNSPECIF | |
| | FIED NATURE SITE |
| C9012 Plasma cell leukemia in relapse | |
| C9020 Extramedullary plasmacytoma not having achieved | |
| remission | |
| C9021 Extramedullary plasmacytoma in remission | |
| C9022 Extramedullary plasmacytoma in relapse | |
| C9030 Solitary plasmacytoma not having achieved remission | |
| C9031 Solitary plasmacytoma in remission | |
| C9032 Solitary plasmacytoma in relapse | |
| C9100 Acute lymphoblastic leukemia not having achieved | |
| remission | |
| C9101 Acute lymphoblastic leukemia, in remission | |
| C9102 Acute lymphoblastic leukemia, in relapse | |
| C9110 Chronic lymphocytic leukemia of B-cell type not having | |
| achieved remission | |
| C9111 Chronic lymphocytic leukemia of B-cell type in remission | |
| C9112 Chronic lymphocytic leukemia of B-cell type in relapse | |
| C9130 Prolymphocytic leukemia of B-cell type not having | |
| achieved remission | |
| C9131 Prolymphocytic leukemia of B-cell type, in remission | |
| C9132 Prolymphocytic leukemia of B-cell type, in relapse | |
| C9140 Hairy cell leukemia not having achieved remission | |
| C9141 Hairy cell leukemia, in remission C9142 Hairy cell leukemia, in relapse | |
| C9142 Hairy cell leukemia, in relapse C9150 Adult T-cell lymphoma/leukemia (HTLV-1-associated) not | |
| having achieved remission | |
| C9151 Adult T-cell lymphoma/leukemia (HTLV-1-associated), in | |
| remission | |
| C9152 Adult T-cell lymphoma/leukemia (HTLV-1-associated), in | |
| relapse | |
| C9160 Prolymphocytic leukemia of T-cell type not having | |
| achieved remission | |
| C9161 Prolymphocytic leukemia of T-cell type, in remission | |
| C9162 Prolymphocytic leukemia of T-cell type, in relapse | |
| C9190 Lymphoid leukemia, unspecified not having achieved | |
| remission | |
| C9191 Lymphoid leukemia, unspecified, in remission | |
| C9192 Lymphoid leukemia, unspecified, in relapse | |
| C91A0 Mature B-cell leukemia Burkitt | |
| C91A1 Mature B-cell leukemia Burkitt | |
| C91A2 Mature B-cell leukemia Burkitt | |
| C91Z0 Other lymphoid leukemia not having achieved remission | |
| C91Z1 Other lymphoid leukemia, in remission | |
| C91Z2 Other lymphoid leukemia, in relapse | |
| C9200 Acute myeloblastic leukemia, not having achieved | |
| remission | |
| C9201 Acute myeloblastic leukemia, in remission | |
| C9202 Acute myeloblastic leukemia, in relapse | |
| C9210 Chronic myeloid leukemia, BCR/ABL-positive, not having | |
| achieved remission | |
| C9211 Chronic myeloid leukemia, BCR/ABL-positive, in | |


## Comorbid conditions


Drug abuse or dependence (includes alcohol)


#### Comorbid conditions


Venous thromboem bolism


#### Comorbid conditions


**Erectile Dysfunction** 


Rheumatoid Arthritis


#### Comorbid conditions


Ravnaud's syndrome


Raynaud's syndrome


Systemic lupus erythematosus
